# CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN FOR

DMID PROTOCOL: 21-0002 (COHORT 2)

## STUDY TITLE:

PHASE I, OPEN-LABEL, RANDOMIZED STUDY OF THE SAFETY AND IMMUNOGENICITY OF A SARS-CoV-2 VARIANT VACCINE (mRNA-1273.351) IN NAÏVE AND PREVIOUSLY VACCINATED ADULTS

NCT04785144

**VERSION 2.0** 

**DATE: 23 MAY 2023** 

RESTRICTED

## **STUDY TITLE**

| <b>Protocol Number Code:</b> | DMID Protocol:21-0002 Cohort 2 |
|---|---|
| <b>Development Phase:</b> | Phase 1 |
| Products: | mRNA-1273/mRNA-1273.351 |
| Form/Route: | Injection |
| Indication Studied: | COVID-19 |
| Sponsor: | Division of Microbiology and Infectious Diseases National Institute of Allergy and Infectious Diseases National Institutes of Health |
| <b>Clinical Trial Initiation Date:</b> | 30MAR2021 |
| <b>Clinical Trial Completion Date:</b> | Ongoing |
| Date of the Analysis Plan: | 23 May 2023 |
| Version Number: | 2.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# TABLE OF CONTENTS

| STUDY | TITLE | 1 |
|---|---|---|
| TABLE | OF CONTENTS | 2 |
| LIST OF | F ABBREVIATIONS | 5 |
| 1. | PREFACE | 7 |
| 2. | INTRODUCTION | 8 |
| 2.1. | Purpose of the Analyses. | 9 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 10 |
| 3.1. | Study Objectives and Endpoints | 10 |
| 3.2. | Study Definitions and Derived Variables | 11 |
| 4. | INVESTIGATIONAL PLAN | 12 |
| 4.1. | Overall Study Design and Plan | 12 |
| 4.2. | Discussion of Study Design, Including the Choice of Control Groups | 13 |
| 4.3. | Selection of Study Population | 14 |
| 4.4. | Treatments | 17 |
| 4.4.1. | Treatments Administered. | 17 |
| 4.4.2. | Identity of Investigational Product(s) | 18 |
| 4.4.3. | Method of Assigning Subjects to Treatment Groups (Randomization) | 18 |
| 4.4.4. | Selection of Dose in the Study | 18 |
| 4.4.5. | Prior and Concomitant Therapy | 18 |
| 4.4.6. | Treatment Compliance | 18 |
| 5. | SAMPLE SIZE CONSIDERATIONS | 19 |
| 6. | GENERAL STATISTICAL CONSIDERATIONS | 20 |
| 6.1. | General Principles | 20 |
| 6.2. | Analysis Populations | 20 |
| 6.2.1. | Safety Population | 20 |
| 6.2.2. | Modified Intent-to Treat Population | 20 |
| 6.2.3. | Per Protocol Population | 20 |
| 6.3. | Covariates and Subgroups | 20 |
| 6.4. | Missing Data | 20 |
| 6.5. | Interim Analyses and Data Monitoring | 21 |

| Table of | f Contents (continued) | |
|---|---|---|
| 6.6. | Multicenter Studies | 21 |
| 6.7. | Multiple Comparisons/Multiplicity | 21 |
| 7. | STUDY SUBJECTS | 22 |
| 7.1. | Disposition of Subjects | 22 |
| 7.2. | Protocol Deviations | 22 |
| 8. | IMMUNOGENICITY EVALUATION | 23 |
| 8.1. | Primary Immunogenicity Analysis | 23 |
| 8.2. | Secondary Immunogenicity Analyses | 23 |
| 8.3. | Exploratory Immunogenicity Analyses | 24 |
| 9. | SAFETY EVALUATION | 25 |
| 9.1. | Demographic and Other Baseline Characteristics | 25 |
| 9.1.1. | Prior and Concurrent Medical Conditions | 25 |
| 9.1.2. | Prior and Concomitant Medications | 25 |
| 9.2. | Measurements of Treatment Compliance | 26 |
| 9.3. | Adverse Events | 26 |
| 9.3.1. | Solicited Events and Symptoms | 26 |
| 9.3.2. | Unsolicited Adverse Events | 26 |
| 9.4. | Deaths, Serious Adverse Events and other Significant Adverse Events | 27 |
| 9.5. | Pregnancies | 27 |
| 9.6. | Clinical Laboratory Evaluations | 27 |
| 9.7. | Vital Signs and Physical Evaluations | 27 |
| 9.8. | Concomitant Medications | 28 |
| 9.9. | Other Safety Measures | 28 |
| 10. | PHARMACOKINETICS | 29 |
| 11. | IMMUNOGENICITY | 30 |
| 12. | OTHER ANALYSES | 31 |
| 13. | REPORTING CONVENTIONS | 32 |
| 14. | TECHNICAL DETAILS | 33 |
| 15. | SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES | 34 |
| 16. | REFERENCES | 35 |
| APPEN | DIX 1. TABLE MOCK-UPS | 37 |

| Statistical Anal | ysis Plan - | - DMID P | rotocol: 21 | -0002 Cohort 2 |
|------------------|-------------|----------|-------------|----------------|
|------------------|-------------|----------|-------------|----------------|

| V | <sup>7</sup> ersic | n | 2.0 |
|----|--------------------|---|-----|
| 23 | May | 2 | 023 |

| Table of Conte | its (continued) | |
|----------------|-----------------|-----|
| APPENDIX 2. | FIGURE MOCK-UPS | 246 |

# LIST OF ABBREVIATIONS

| AE | Adverse Event |
|--------|--------------------------------------------------|
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| AUC | Area Under the Curve |
| BP | Blood Pressure |
| С | Celsius |
| CI | Confidence Interval |
| CRF | Case Report Form |
| DMID | Division of Microbiology and Infectious Diseases |
| EDC | Electronic Data Capture |
| ECLIA | Electro-chemiluminescence |
| ELISA | Enzyme-linked Immunosorbent Assay |
| F | Fahrenheit |
| FRNT | Focus Reduction Neutralization Test |
| GMT | Geometric Mean Titer |
| GMFR | Geometric Mean Fold Rise |
| ICH | International Council on Harmonisation |
| IRB | Institutional Review Board |
| LLN | Lower Limit of Normal |
| μg | Microgram |
| MedDRA | Medical Dictionary for Regulatory Activities |
| N | Number (typically refers to subjects) |
| NIH | National Institutes of Health |
| PI | Principal Investigator |
| PP | Per Protocol |
| PT | Preferred Term |
| RBC | Red Blood Cell |
| S-2P | S Protein in its Prefusion Conformation |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SDCC | Statistical and Data Coordinating Center |

| SMC | Safety Monitoring Committee |
|-----|-------------------------------|
| SOC | System Organ Class |
| SOP | Standard Operating Procedures |
| ULN | Upper Limit of Normal |
| WBC | White Blood Cell |
| WHO | World Health Organization |

## 1. PREFACE

The Statistical Analysis Plan (SAP) for "Phase 1, Open-Label, Randomized Study of the Safety and Immunogenicity of a SARS-CoV-2 Variant Vaccine (mRNA-1273.351) in Naïve and Previously Vaccinated Adults" (DMID Protocol 21-0002) describes and expands upon the statistical information presented in the protocol for cohort 2 only. A separate SAP will be written for cohort 1. This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, listings, and figures planned for the final analyses. Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains a review of the study design, general statistical considerations, comprehensive statistical analysis methods for immunogenicity and safety outcomes, and a list of proposed tables, figures and listings. Within the table, figure, and listing mock-ups (Appendix 1, Appendix 2, and Appendix 3), references to CSR sections are included. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

## 2. INTRODUCTION

An outbreak of COVID-19 caused by a novel SARS-CoV-2 began in Wuhan, Hubei Province, China in December 2019, and the disease has since spread globally [10]. The World Health Organization (WHO) declared COVID-19 a pandemic on 11 Mar 2020; however, widespread community transmission was already occurring in many locations. As of 14 Jan 2021, more than 92 million cases and 1.9 million deaths worldwide have been attributed to the COVID-19 pandemic [2,10].

ModernaTX, Inc has developed a vaccine platform based on the principle and observations that cells *in vivo* can take up mRNA, translate it, and then express protein viral antigen(s) on the cell surface. mRNA is highly precise in its translation into proteins that match viral antigens. The delivered mRNA does not enter the cell nucleus or interact with the genome, is nonreplicating, and is expressed transiently. The estimated half-life for mRNA after injection is approximately 8 to 10 hours, before degradation by native RNases in the body, but the duration of effect also depends on the half-life of the expressed protein, which persists in the body for several days. mRNA vaccines have been used to induce immune responses against infectious viral pathogens such as cytomegalovirus, human metapneumovirus, parainfluenza virus type 3, Zika, and influenza.

The mRNA-1273 encodes for the full-length spike (S) protein of SARS-CoV-2, modified to introduce 2 proline residues to stabilize the S protein (S-2P) in a prefusion conformation, derived from the Wuhan-Hu-1 strain [5]. The mRNA-1273 vaccine is currently being evaluated for safety and immunogenicity in a dose-ranging Phase 1 study sponsored by DMID (NCT04283461), for safety and immunogenicity in a Moderna-sponsored Phase 2a study (NCT04405076), and for safety, efficacy, and immunogenicity in a Moderna-sponsored Phase 3 study (NCT04470427). All three of these studies are ongoing and conducted in the US.

The primary efficacy objective of the Phase 3 study was met, with the vaccine efficacy of mRNA-1273 to prevent symptomatic COVID-19 disease observed to be 94.1%. The vaccine was also observed to be efficacious in preventing severe COVID-19. In December 2020 the FDA issued Emergency Use Authorization of mRNA-1273 (Moderna COVID-19 Vaccine) for active immunization to prevent COVID-19 in individuals 18 years of age and older.

Recently, SARS-CoV-2 variants with mutations in the S protein have emerged. A variant first identified in South Africa (B.1.351) is associated with increased transmission, higher viral burden, and possibly increased mortality in infected persons [8]. To date, four vaccines, all based on the Wuhan-sequence of the S protein, have shown reduced activity against the B.1.351 variant. Sera from individuals vaccinated with mRNA-based vaccines had a 6-to-9-fold reduction in neutralizing activity against a B.1.351-matched pseudovirion relative to a Wuhan-matched pseudovirion [9,11]. More recently, pivotal studies testing both viral vector and adjuvanted protein technologies had lower efficacy in regions where B.1.351 was known to be circulating [2]. Hence, the development and testing of vaccines targeting this SARS-CoV-2 variant is urgently needed.

mRNA-1273.351, like mRNA-1273, encodes the prefusion stabilized S protein of SARS-CoV-2. However, the mRNA of mRNA-1273.351 incorporates the key mutations present in the B.1.351 strain of the virus. This phase 1 clinical trial will evaluate the immunological benefit of boosting subjects previously vaccinated with mRNA-1273 (DMID 20-0003) with the B.1.351

strain-specific S protein, as well as the breadth of response induced by vaccinating with mRNA-1273 and mRNA-1273.351 in naïve persons, who have not previously received a SARS-CoV-2 vaccine and are not known to have been previously infected with SARS-CoV-2.

## 2.1. Purpose of the Analyses

These analyses will assess the immunogenicity and safety of mRNA-1273.351, given in vaccination schedules alone, sequentially, or co-administered with mRNA-1273 in naïve adults.

## 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. Study Objectives and Endpoints

| OBJECTIVES | ENDPOINTS<br>(OUTCOME MEASURES) |
|---|---|
| Primary | (G G T G G T III T T III T G T III G T |
| To evaluate the safety and reactogenicity<br>of mRNA-1273 and mRNA-1273.351<br>vaccines, in naïve individuals. | Frequency and grade of each solicited local and systemic reactogenicity AE during a 7-day follow-up period post each vaccination. |
| | • Frequency and grade of any unsolicited AEs during the 28-day follow-up period post each vaccination. |
| | • Frequency of any SAEs, Protocol<br>Specified AESIs, NOCMCs, and MAAEs<br>from the first vaccination through 12<br>months after the last vaccination. |
| Secondary | |
| To assess humoral immunogenicity of<br>mRNA-1273 and mRNA-1273.351<br>vaccines, in naïve individuals. | • Response rate, and magnitude of SARS-CoV-2-specific antibody binding and neutralization titers in serum samples as assessed via a range of assays at all timepoints. |
| Exploratory | |
| To assess, in at least a subset of samples<br>the innate immune response and B cell<br>response following vaccination. | Magnitude, phenotype, and percentage of innate immune cells and SARS-CoV-2 specific B cells, as measured by flow cytometry, and targeted B cell repertoire analysis at different timepoints post vaccination relative to baseline. |
| • To assess, in at least a subset of samples, the SARS-CoV-2 S protein-specific T cell responses. | Magnitude, phenotype, and percentage of cytokine producing S protein-specific T cells, as measured by flow cytometry at different timepoints post vaccination relative to baseline. |

## 3.2. Study Definitions and Derived Variables

For calculations using the baseline value, the value obtained pre-first vaccination (Day 1) will be used. For samples with an AUC of zero at baseline, fold-rise will be calculated by dividing the post-vaccination result by the lowest reported value. AUC is calculated using the trapezoidal method applied to a serial dilution curve.

The Williams mean is a variation of the geometric mean using log(1+x) transformation of the data, where x is each data point. The Williams mean is used in cases where 0 is a possible and/or reported value of the data.

## 4. INVESTIGATIONAL PLAN

## 4.1. Overall Study Design and Plan

This is a phase 1, open-label, randomized clinical trial in males and non-pregnant females, 18 years of age and older, who are in good health, have no known history of COVID-19 or SARS-CoV-2 infection, and meet all other eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of mRNA-1273.351 manufactured by ModernaTX, Inc, given in vaccination schedules alone, sequentially, or co-administered with mRNA-1273. mRNA-1273.351 is a novel LNP-encapsulated mRNA-based vaccine that encodes for a full-length, prefusion stabilized S protein of the SARS-CoV-2 B.1.351 variant. Enrollment will occur at approximately five domestic clinical research sites.

This study includes two cohorts. Cohort 1 will provide rapid information about the immunogenicity of mRNA-1273.351 in a previously vaccinated group. This cohort can inform near term public health decisions if the variant virus becomes more widespread. Cohort 2 will evaluate different strategies for generation of cross protective immune responses in a naïve population. This cohort will take longer to provide information on the immunogenicity of mRNA-1273.351, but is important to inform future public health strategies. As Cohorts 1 and 2 are in different populations, they can be enrolled in parallel as determined by each site.

Cohort 1 will include subjects 18 years of age and older who received two vaccinations of mRNA-1273 at dosages of 50 mcg, 100 mcg, or 250 mcg in the Phase 1 clinical trial (DMID 20-0003). Those subjects will be offered enrollment into this study approximately 9 to 12 months after they received the second vaccination in DMID 20-0003. At enrollment in this study, their long-term follow-up in DMID 20-0003 will be terminated. Subjects will be randomized, within each of the DMID 20-0003 cohorts (age and dosage groups – 50 mcg, 100 mcg, and 250 mcg), 1:1 to either:

- Arm 1A, vaccination with a 50-mcg dose of the mRNA-1273.351 variant, or
- Arm 1B, vaccination with a combination vaccination that includes 25 mcg of mRNA-1273 and 25 mcg of mRNA-1273.351.

The anticipated sample size to be drawn from the DMID 20-0003 study population is approximately 45 subjects 18 through 55 years of age and approximately 20 subjects 56 years of age and older.

Subjects in Cohort 1 will receive a single intramuscular (IM) injection of the designated vaccine and will be followed through 12 months after vaccination. Follow-up visits will occur on Days 8, 15, and 29, as well as 3, 6, and 12 months after the vaccination.

Cohort 2 will include approximately 150 participants 18 through 55 years of age who have not received a COVID-19 vaccine, have no known history of COVID-19 or SARS-CoV-2 infection, and do not have underlying conditions that are associated with an increased risk of severe illness from SARS-CoV-2 infection. Enrollment may close before the full 150 participants based on estimates on the timing of immunogenicity results and the need to inform public health decisions. They will be randomly assigned to one of 8 treatment arms and will receive 2 or 3 IM injections of the vaccine and followed through 12 months after the last vaccination (Table 1).

Follow-up visits will occur 7, 14, and 28 days after each vaccination, as well as 3, 6, and 12 months post the last vaccination.

For both Cohorts 1 and 2, reactogenicity will be assessed and blood will be drawn for immunogenicity assays.

After the IND is in effect, IRB review and approval, and site activation, the participating sites will begin recruitment outreach efforts, which can include fliers, letters, telephone calls, etc. Information regarding this trial may be provided to potential subjects who have previously participated in other vaccine trials conducted at the participating site. Other forms and/or mechanisms of recruitment may also be used. The IRB will approve the recruitment process and all materials prior to use. Screening can occur up to 42 days prior to the first dose.

## 4.2. Discussion of Study Design, Including the Choice of Control Groups

This phase 1 clinical trial is designed as an open-label study, without administration of a placebo formulation. An open-label study will facilitate the need for rapid review and dissemination of study data for public health reasons.

In the Phase 1 clinical trial, DMID 20-0003, mRNA-1273, administered as two injections 28 days apart, was investigated at dosages of 25, 50, 100 and 250 mcg in subjects 18 through 55 years of age, and at dosages of 25, 50, and 100 mcg in older cohorts (56-70 years of age and >71 years of age) [1,7]. The 100-mcg dose induced higher antibody titers than the 25-mcg dose, whereas the 250-mcg dose did not lead to significant increases, which supported evaluation of the 100-mcg dose in Phase 2 and Phase 3 trials. Subsequent to the start of the Phase 3 trial, an interim analysis of immunogenicity data from the Phase 2 demonstrated that the 50 and 100-mcg doses in a two-dose series are similarly immunogenic [4] and warrants further evaluation. The primary efficacy analysis from the Phase 3 trial evaluating a two-dose schedule of a 100-mcg mRNA-1273 vaccine led to the issuance of the EUA and initiation of a vaccination campaign in the United States.

The Phase 2 trial of mRNA-1273 evaluated doses of 50 mcg and 100 mcg, administered as a two-vaccination series, in 600 adults ≥18 years of age. The safety profile of both formulations was acceptable [4]. Anti-SARS-CoV-2 S binding and neutralizing antibodies were induced by both dose levels of mRNA-1273 within 28 days after the first vaccination, and rose substantially to peak titers by 14 days after the second vaccination, exceeding levels of convalescent sera from COVID-19 patients. The antibodies remained elevated through the last timepoint assessed at 57 days. Neutralizing responses met criteria for seroconversion within 28 days after the first vaccination in the majority of participants, with rates of 100% observed at 14 and 28 days after the second vaccination. Binding and neutralizing antibody responses were generally comparable in participants who received the 100 mcg mRNA-1273 and the 50 mcg dose at all time points and across the age groups of ≥18 to <55 years and ≥55 years. These findings support the evaluation of mRNA-1273 and mRNA-1273.351 at total dosages of 50 or 100 mcg per vaccination.

## 4.3. Selection of Study Population

Two cohorts will be enrolled. For Cohort 1, approximately 60 males and non-pregnant female subjects 18 years of age and older, who are in good health and received two vaccinations of mRNA-1273 at dosages of 50 mcg, 100 mcg or 250 mcg in DMID 20-0003 will be invited to participate in this study.

For Cohort 2, approximately 150 males and non-pregnant females, 18 through 55 years of age, who have never been vaccinated against SARS-CoV-2 or are not known to have been infected with SARS-CoV-2, and are at low risk for severe disease, in good health, and meet all eligibility criteria will be enrolled. The target population should reflect the community at large.

The estimated time from initiation of enrollment to complete enrollment in this clinical trial is approximately 4 weeks (though could take up to 8 weeks). Information regarding this trial may be provided to potential subjects who have previously participated in other vaccine trials conducted at the participating site. Other forms and/or mechanisms of recruitment may also be used. The IRB will approve the recruitment process and all materials prior to use. Screening can occur up to 42 days prior to the first vaccination.

Subject Inclusion and Exclusion Criteria must be confirmed by a study clinician, licensed to make medical diagnoses and listed on the Form FDA 1572 as the participating site principal investigator (PI) or appropriate sub-investigator. No exemptions are granted on Subject Inclusion or Exclusion Criteria in DMID-sponsored studies.

#### **Inclusion Criteria**

A subject must meet all the following criteria to be eligible to participate in this study:

- 1. Provides written informed consent prior to initiation of any study procedures.
- 2. Be able to understand and agrees to comply with planned study procedures and be available for all study visits.
- 3. Agrees to the collection of venous blood per protocol.
- 4. Cohort 1: previously received 2 doses of mRNA-1273 IM as part of DMID 20-0003.
- 5. Cohort 1: Male or non-pregnant female, ≥18 years of age at time of enrollment.Cohort 2: Male or non-pregnant female, 18 through 55 years of age at time of enrollment.
- 6. Women of childbearing potential<sup>1</sup> must agree to practice abstinence or use at least one acceptable primary form of contraception.<sup>2,3</sup>
- Note: These criteria are applicable to females in a heterosexual relationship and childbearing potential (i.e., the criteria do not apply to subjects in a same sex relationship).
- <sup>1</sup>Not of childbearing potential post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure® placement).
- <sup>2</sup>Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the

subject's first vaccination, intrauterine devices, birth control pills, and injectable/implantable/insertable hormonal birth control products.

<sup>3</sup>Must use at least one acceptable primary form of contraception for at least 30 days prior to the first vaccination and at least one acceptable primary form of contraception for 60 days after the last vaccination.

## 7. In good health.<sup>4</sup>

- <sup>4</sup>As determined by medical history and physical examination to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the assessment of safety of subjects. Chronic medical diagnoses/conditions should be stable for the last 60 days (no hospitalizations, ER, or urgent care for condition or need for supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis/condition in the 60 days before enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or done for financial reasons, and in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to **improvement** of a disease outcome or for dose optimization, as determined by the participating site PI or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the participating site PI or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity, and do not indicate a worsening of medical diagnosis/condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided the change was not precipitated by deterioration in the chronic medical condition, and there is no anticipated additional risk to the subject or interference with the evaluation of responses to study vaccination.
- 8. Oral temperature is less than 100.0°F (37.8°C).
- 9. Must agree to have samples stored for secondary research.
- 10. Agrees to adhere to Lifestyle Considerations (defined in Section 5.4 of the Protocol) throughout study duration.
- 11. Must agree to refrain from donating blood or plasma during the study (outside of this study).

#### **Exclusion Criteria**

A subject who meets any of the following criteria will be excluded from participation in this study:

- 1. Positive pregnancy test prior to each vaccine administration.
- 2. BMI  $>40.0 \text{ kg/m}^2$ .
- 3. Female subject who is breastfeeding.
- 4. Has any medical disease or condition that, in the opinion of the participating site PI or appropriate sub-investigator, precludes study participation.<sup>5</sup>

- <sup>5</sup>Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
- 5. Presence of self-reported or medically documented significant medical or psychiatric condition(s).<sup>6</sup>
- <sup>6</sup>Significant medical or psychiatric conditions include but are not limited to:
  - Respiratory disease (e.g., chronic obstructive pulmonary disease [COPD], asthma) requiring daily medications currently or any treatment of respiratory disease exacerbations (e.g., asthma exacerbation) in the last 5 years. Asthma medications: inhaled, oral, or intravenous (IV) corticosteroids, leukotriene modifiers, long and short acting beta agonists, theophylline, ipratropium, biologics.
  - Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease), history of myocarditis or pericarditis as an adult, myocardial infarction (MI) within past 6 months, coronary artery bypass surgery or stent placement, or uncontrolled cardiac arrhythmia.
  - Neurological or neurodevelopmental conditions (e.g., history of migraines in the past 5 years, epilepsy, stroke, seizures in the last 3 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis, transverse myelitis, stroke or transient ischemic attack, multiple sclerosis, Parkinson's disease, amyotrophic lateral sclerosis, Creutzfeldt-Jakob disease, or Alzheimer's disease).
  - Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding basal cell and squamous cell carcinoma of the skin, which are allowed.
  - An autoimmune disease, including hypothyroidism without a defined non-autoimmune cause, localized or history of psoriasis.
  - An immunodeficiency of any cause.
  - Chronic kidney disease, estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m<sup>2</sup>. Type 2 diabetes mellitus, not including prediabetes.
- 6. Has an acute illness<sup>7</sup>, as determined by the participating site PI or appropriate sub-investigator, with or without fever [oral temperature ≥38.0°C (100.4°F)] within 72 hours prior to each vaccination.
- <sup>7</sup>An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the participating site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
- 7. Has participated in another investigational study involving any investigational product<sup>8</sup> within 5 half-lives before the first vaccine administration.
- <sup>8</sup>Study drug, biologic or device

8. Currently enrolled in or plans to participate in another clinical trial with an investigational agent<sup>9</sup> that will be received during the study-reporting period.<sup>10</sup>

- 9. Has a history of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to drugs or any previous licensed or unlicensed vaccines or to polyethylene glycol (PEG) or a PEG-containing product.
- 10. Chronic use (more than 14 continuous days) of any medications that may be associated with impaired immune responsiveness.<sup>11</sup>
- <sup>11</sup>Including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other similar or toxic drugs during the preceding 6-month period prior to vaccine administration (Day 1). The use of low dose topical, ophthalmic, inhaled and intranasal steroid preparations will be permitted.
- 11. Anticipating the need for immunosuppressive treatment within the next 6 months.
- 12. Received immunoglobulins and/or any blood or blood products within the 4 months before the first vaccine administration or at any time during the study.
- 13. Has any blood dyscrasias or significant disorder of coagulation.
- 14. Received or plans to receive a licensed, live vaccine within 4 weeks before or after each vaccination.
- 15. Received or plans to receive a licensed, inactivated vaccine within 2 weeks before or after each vaccination.
- 16. Receipt of any other SARS-CoV-2 vaccine or any experimental coronavirus vaccine at any time prior to or during the study, except Cohort 1 subjects who received mRNA-1273 in DMID 20-0003.
- 17. Close contact of anyone known to have SARS-CoV-2 infection within 14 days prior to vaccine administration.
- 18. History of COVID-19 diagnosis, positive SARS-CoV-2 PCR test, or, for Cohort 2 only, a known positive SARS-CoV-2 serologic test.
- 19. On current treatment with investigational agents for prophylaxis of COVID-19.

#### 4.4. Treatments

#### 4.4.1. Treatments Administered

Eight treatment arms administering various combinations of mRNA-1273 and mRNA-1273.351 (Table 1).

<sup>&</sup>lt;sup>9</sup>Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.

<sup>&</sup>lt;sup>10</sup>Up to 15 months after the first vaccination.

#### **Summary of Treatment Arms:**

- 2A: Evaluates the mRNA-1273 EUA vaccination series, plus a variant vaccine as a third dose.
- 2B: Evaluates a 50-mcg mRNA-1273 vaccination series, plus a variant vaccine as a third dose.
- 2C: Evaluate 2 doses of the homologous variant vaccine at 100mcg.
- 2D: Evaluate 2 doses of the homologous variant vaccine at 50mcg.
- 2E: Evaluate heterologous prime-boost strategies at 100mcg.
- 2F: Evaluate heterologous prime-boost strategies at 50mcg.
- 2G: Evaluate a 1:1 mix of vaccine (2 doses), with the total dose for <u>both vaccines</u> equal to 100 mcg.
- 2H: Evaluate a 1:1 mix of vaccine (2 doses), with the total dose for <u>both vaccines</u> equal to 50 mcg.

#### 4.4.2. Identity of Investigational Product(s)

# <u>Product: There are two clinical presentations of mRNA-1273 — mRNA-1273 and mRNA-1273.351</u>

mRNA-1273 (0.2 mg/mL) is an LNP dispersion containing an mRNA that encodes for the pre fusion stabilized S protein of the Wuhan-Hu-1 strain of SARS-CoV-2. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.

mRNA-1273.351 (0.5 mg/mL) is formulated in the same way but contains mRNA that encodes for the prefusion stabilized S protein of the B.1.351 variant SARS-CoV-2 strain.

#### 4.4.3. Method of Assigning Subjects to Treatment Groups (Randomization)

Subjects in Cohort 2 will be randomized in a ratio of 3:3:4:4:4:4:4 to Arms 2A-H. Randomization will be done in the SDCC's Advantage eClinical<sup>SM</sup> (Electronic Data Capture System).

#### 4.4.4. Selection of Dose in the Study

See Section 4.2 for a discussion of dose selection for this study.

## 4.4.5. Prior and Concomitant Therapy

Concomitant medications include only prescription medications and vaccines received outside of the study taken by the subject at the time of enrollment through 28 days after the last vaccination. At each study visit, if there are new SAEs, Protocol Specified AESIs, MAAEs, or NOCMCs, concomitant medications should be recorded on the appropriate DCF.

#### 4.4.6. Treatment Compliance

All subjects are to receive 2 (Arms 2C-H) or 3 (Arms 2A-B) doses of study product administered in the clinic. The number of doses received will be reported in Table 7 (Arms 2A-B) and Table 8 (Arms 2C-H).

## 5. SAMPLE SIZE CONSIDERATIONS

Rare AEs are not demonstrable in a clinical study of this size; however, the probabilities of observing one or more AEs given various true event rates are presented in Table 4. With the assumption that all enrolled subjects will likely complete immunizations and safety visits in this relatively short duration study, the following statistical considerations apply. With 15 subjects in Arms 2A and 2B, the chance of observing at least one AE of probability 20% or more is approximately 97%. Therefore, if no AEs of a given type occur in Arms 2A or 2B, we can be relatively confident that they will occur in fewer than 20% of people once the vaccine is implemented. With 20 subjects in each arm (Arms 2C-2H), the chance of observing at least one AE of probability 20% or more is approximately 99%. Therefore, if no AEs of a given type occur in Arms 2C-2H, we can be relatively confident that they will occur in fewer than 20% of people once the vaccine is implemented. With approximately 150 subjects across these eight Arms (2A-2H), the chance of observing at least one AE of probability 3% or more is at least 99%. Therefore, if no AEs of a given type occur across Cohort 2, we can be very confident that any dosage/combination independent event will occur in fewer than 3% of people once the vaccine is implemented.

#### 6. GENERAL STATISTICAL CONSIDERATIONS

## **6.1.** General Principles

In general, continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum, and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. In general, all data will be listed, sorted by site, treatment, and subject, and when appropriate by visit number within subject. All summary tables will be structured with a column for each treatment and will be annotated with the total population size relevant to that table/cohort, including any missing observations.

## **6.2.** Analysis Populations

#### **6.2.1.** Safety Population

The Safety Analysis population includes all subjects who received one dose of the vaccine.

#### **6.2.2.** Modified Intent-to Treat Population

The modified intent-to-treat (mITT) population includes all subjects who received at least one dose of the vaccine and contributed both pre- and at least one post-vaccination venous blood samples for immunogenicity testing for which valid results were reported.

## **6.2.3.** Per Protocol Population

In the final analysis, protocol deviations will be reviewed to determine which protocol deviations may affect the analysis. The per protocol (PP) population will then be defined – and this includes all subjects in the mITT subset with the following exclusions:

- Data from all available visits for subjects found to be ineligible at baseline.
- Data from all visits subsequent for the protocol deviations that are considered to affect the science.
- Data from any visit that occurs substantially out of window.

## 6.3. Covariates and Subgroups

The protocol does not define any formal subgroup analyses, and the study is not adequately powered to perform subgroup analyses.

# 6.4. Missing Data

There are no imputations planned for missing data.

For immunogenicity assays, any values below the lower limit of detection will be imputed as one-half the lower limit of detection for analysis purposes. Any such imputations will be noted in the corresponding analysis.

## 6.5. Interim Analyses and Data Monitoring

Cumulative safety information, study status, and primary endpoint results may be published, presented at a public forum, or presented as summaries aggregated by study arm at the discretion of the sponsor while the study is ongoing. Any ad-hoc analyses, jointly developed by the SDCC and/or the Vaccine Research Center (VRC), other participating laboratories and ModernaTX, Inc., will be executed by the SDCC as needed. None of the interim analyses will include any formal statistical hypothesis testing; therefore, p-value adjustment will not be made to any analyses.

The SMC will not need to meet (unless halting rules are met), and materials will be provided electronically. Documentation of review and any concerns noted will be solicited electronically. The SMC will review cumulative AE data after all subjects in Cohort 1 have been dosed and completed Day 8.

Interim data review of immunogenicity may be performed to inform public health decisions.

Statistical analyses of secondary immunogenicity endpoints, by vaccine schedule group, may be performed when subjects have completed key immunogenicity visits. Immunogenicity reviews may be shared with the SMC, as determined by DMID.

Data may be disseminated to public health officials and partners as needed and included in publications and presentations to inform the global scientific community.

Interim analyses of safety, reactogenicity, and immunologic response data may be done, as needed.

## 6.6. Multicenter Studies

Data will be pooled across all clinical sites. Center effects are not anticipated because the sites are using standardized procedures for vaccination and assessment of solicited and unsolicited adverse events, and the study relies on central laboratories for the assessment of immunogenicity endpoints.

# 6.7. Multiple Comparisons/Multiplicity

There are no adjustments planned for multiple comparisons.

#### 7. STUDY SUBJECTS

## 7.1. Disposition of Subjects

Table 11 will present a summary of the reasons that subjects were screened but not enrolled.

The composition of analysis populations, including reasons for subject exclusion, by treatment arm, is presented in Table 9 and Table 10.

The disposition of subjects in the study will be tabulated by treatment group (Table 7 and Table 8). The tables show the total number of subjects screened, enrolled, receiving the first vaccination, receiving second vaccination, receiving third vaccination (Arms 2A-B), terminated from study follow-up, and the number completing the study.

A flowchart showing the disposition of study subjects, adapted from the Consort Statement [5] will be included (Figure 1). This figure will present the number of subjects screened, enrolled, lost to follow-up, and analyzed, by treatment group.

A listing of subjects who discontinued dosing or terminated from study follow-up and the reason will be included in Listing 2.

## 7.2. Protocol Deviations

A summary of subject-specific protocol deviations will be presented by the reason for the deviation, the deviation category, and treatment group for all subjects (Table 5) as well as similar summaries for major subject-specific protocol deviations (Table 6). All subject-specific protocol deviations and non-subject specific protocol deviations will be included in Appendix 3 as data listings (Listing 3 and Listing 4, respectively).

## 8. IMMUNOGENICITY EVALUATION

## 8.1. Primary Immunogenicity Analysis

See Section 9 for safety analyses which are the primary endpoints of this study.

## 8.2. Secondary Immunogenicity Analyses

Summaries and analysis of immunogenicity data will be presented for the mITT population. If there are protocol deviations which may affect the analysis, a per-protocol (PP) analysis may also be performed.

Seropositive is defined as above LLOD (if available).

Binding will be measured by three types of ECLIA assays. The first is a single-plex (ECLIA) that produces arbitrary units/mL that is a validated assay and can be converted to binding antibody units for Wa-1 S-2P binding. The second is a 4-plex (ECLIAv2) assay that is also validated and produces arbitrary units/mL to measure variant specific binding. The final assay is a 10-plex (ECLIAv2) that is a fit for purpose assay that produces area under the curve and is used to assess binding for variants of concern.

Seropositive rates, geometric mean fold rise (GMFR) and geometric mean (GM) or Williams mean of arbitrary units per mL (AU/mL), binding antibody unit/mL (BAU, only for Wa-1 [S2-P] variant), and AUC for SARS-CoV-2 will be calculated at Study Days 1 (GM only), 15, 29, 43, 57, 71, 85, 147, 237, and 422 (Arms 2A-B) and Days 1, 15, 29, 43, 57, 119, 209, 394 (Arms 2C-H) by treatment group and will include both tabular and graphical summaries. Seropositive rates, GMFR, and GM will be presented with their corresponding 95% confidence interval (CI) estimates (using Student's t-distribution for GM and GMFR and the Clopper-Pearson binomial method for seropositive) at each post vaccination timepoint and overall peak GM. Summaries of GM are included starting with Table 15 and ending with Table 62; and summaries of GMFR and seroconversion are included starting with Table 191 and ending with Table 238. Graphical displays will include reverse cumulative distribution plots (starting with Figure 2, ending with Figure 25; and starting with Figure 86, ending with Figure 109), individual values over time (starting with Figure 170, ending with Figure 193; and starting with Figure 254, ending with Figure 277), geometric mean over time (starting with Figure 338, ending with Figure 361; and starting with Figure 422, ending with Figure 445), and distribution of responses over time (starting with Figure 506, ending with Figure 529; and starting with Figure 590, ending with Figure 613).

Neutralization assays using SARS-CoV-2 pseudovirus neutralization assay (PsVNA) and focus reduction neutralization test (FRNT) will be run using serial dilutions against available variants (e.g., Beta, Delta, Omicron). ID<sub>50</sub> and ID<sub>80</sub> will be calculated using methodology such as a 5-parameter logistic regression model by the laboratory. ID<sub>50</sub> and ID<sub>80</sub> will be summarized by group using the geometric mean and 95% CI (using Student's t-distribution) at each post vaccination timepoint and overall peak GM (starting with Table 63 and ending with Table 182). Summaries of GMFR and seropositive are included starting with Table 239 and ending with Table 358. The ratio of the result for each variant divided by the result of the D614G variant will be calculated and summarized as the geometric mean ratio (GMR) (starting with Table 359 and ending with Table 382). Graphical displays for PsVNA and FRNT will include reverse

cumulative distribution plots (starting with Figure 26, ending with Figure 85; and starting with Figure 110, ending with Figure 169), individual values over time (staring with Figure 194, ending with Figure 253; and starting with Figure 278, ending with Figure 337), geometric mean over time (starting with Figure 362, ending with Figure 421; and starting with Figure 446, ending with Figure 505) and distributions of responses over time (starting with Figure 530, ending with Figure 589; and starting with Figure 614, ending with Figure 673).

Correlations between all assays will be displayed in a heatmap (staring with Figure 674 and ending with Figure 697).

Summaries of N-antibody expression status and self-reported infection status will be reported in Table 383, Table 384, Table 385, and Table 386.

Individual immunogenicity responses are shown in Listing 8.

Any additional variants of concern not listed in the appendices that are of scientific interest may be analyzed in an analogous manner in the final report.

## 8.3. Exploratory Immunogenicity Analyses

The magnitude, phenotype and percentage of cytokine expressing S protein specific T cells will be summarized at each timepoint by Treatment Group. Mean percentages of CD4 and CD8 T cells expressing cytokines and proportions of responders with 95% CI along with median, minimum, and maximum will be presented by peptide pool stimulation (Table 183, Table 184, Table 185, Table 186, Table 187, Table 188, Table 189, and Table 190). Distributions of T cell percentages will be graphically displayed (starting with Figure 698 and ending with Figure 1249).

Individual T-cell responses are shown in Listing 9.

## 9. SAFETY EVALUATION

Summaries and analysis of safety data will be presented for the Safety Analysis Population.

Solicited AEs will be summarized by severity for each day post vaccination (Days 1-8) for each dose and as the maximum severity over all 8 days. Additionally, solicited AEs will be analyzed by taking the most severe response over the follow-up period and using standard techniques, such as exact confidence intervals (CI), to summarize the proportion of subjects reporting each symptom, any local symptom, and any systemic symptom.

Unsolicited non-serious AEs will be collected from the time of the first vaccination through 28 days after the final vaccination. Unsolicited AEs will be coded by MedDRA for preferred term and system organ class (SOC). SAEs, Protocol Specified AESIs, MAAEs, and NOCMCs will be collected from the time of first vaccination through 12 months after the final vaccination. The numbers of SAEs and MAAEs will be reported by detailed listings showing the event description, MedDRA preferred term and SOC, relevant dates (vaccinations and AEs), severity, relatedness, and outcome for each event. Non-serious unsolicited AEs will be summarized as number and percentage of subjects reporting at least one event in each MedDRA preferred term and SOC, cross tabulated by severity and relationship to study product. Additionally, the proportion of subjects and exact 95% CIs of AEs in aggregate and by MedDRA categories will be computed.

## 9.1. Demographic and Other Baseline Characteristics

Summaries of age, sex, ethnicity, and race will be presented by Treatment Group (Table 12 and Table 13). Ethnicity is categorized as Hispanic or Latino, or not Hispanic and not Latino. In accordance with NIH reporting policy, subjects may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the CRF as "No" to each racial option. Prior infection status by N-antibody will also be included.

Individual subject listings will be presented for all demographics (Listing 6).

#### 9.1.1. Prior and Concurrent Medical Conditions

All current illnesses and past pre-existing medical conditions will be MedDRA® coded using MedDRA dictionary version 23.0r higher.

Summaries of subjects' pre-existing medical conditions will be presented by Treatment Group (Table 14).

Individual subject listings will be presented for all medical conditions (Listing 7).

#### 9.1.2. Prior and Concomitant Medications

Summaries of medications that were started prior to dosing and continuing at the time of dosing will be presented by WHO Drug Terms 2 and 3 and Treatment Group (Table 425).

Individual subject listings will be presented for all concomitant medications (Listing 15).

## 9.2. Measurements of Treatment Compliance

All subjects are to receive 2 (Arms 2C-H) or 3 (Arms 2A-B) doses of study product administered in the clinic. The number of subjects receiving each dose will be summarized as part of the subject disposition table (Table 7 and Table 8).

#### 9.3. Adverse Events

When calculating the incidence of adverse events (i.e., on a per subject basis), each subject will only be counted once and any repetitions of adverse events within a subject will be ignored; the denominator will be the total population size. All adverse events reported will be included in the summaries and analyses.

## 9.3.1. Solicited Events and Symptoms

Systemic solicited adverse events were collected pre-vaccination, and systemic and local solicited adverse events were collected 30 minutes post-vaccination and then daily for 7 days after the vaccination and graded on a scale of 0 (absent), 1 (mild), 2 (moderate) and 3 (severe). Systemic events include: fatigue, headache, myalgia, arthralgia, nausea, chills and fever. Local events include: pain at injection site, erythema, and induration.

For each systemic and local event, any systemic event, any local event, and any solicited event, the maximum severity over 7 days after the third vaccination will be summarized for the Safety population. The number and percentage of subjects reporting each event will be summarized by the maximum severity and treatment group (Table 389). For each event the denominator is the number of subjects with non-missing data for the specific event.

The number of subjects reporting a solicited adverse event will be summarized for each day post-vaccination both in a summary table (staring with Table 390 and ending with Table 407) and graphically in a bar chart (Figure 1250, Figure 1251, Figure 1252, Figure 1253, Figure 1254, and Figure 1255).

The mean, standard deviation, median, minimum and maximum duration of solicited events will be summarized (Table 408).

Day of solicited symptom onset will be summarized graphically (Figure 1256, Figure 1257, Figure 1258, Figure 1259, Figure 1260, and Figure 1261).

Solicited adverse events by subject will be presented in listings (Listing 10 and Listing 11) and graphically (starting with Figure 1262 and ending with Figure 1275).

#### 9.3.2. Unsolicited Adverse Events

The proportion of subjects reporting at least one unsolicited adverse event will be summarized by MedDRA system organ class and preferred term. Denominators for percentages are the number of subjects who received the vaccination.

Adverse events by subject will be presented in Listing 12.

The following summaries for unsolicited adverse events will be presented by MedDRA system organ class, preferred term, and Treatment Group:

- Subject incidence and total frequency of adverse events (Table 409);
- Summary of severity and relationship to study product (Table 410 and Table 411);
- Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events (Table 412);
- Bar chart of frequency of adverse events by severity and MedDRA system organ class (Figure 1274);
- Bar chart of incidence of adverse events by severity and MedDRA system organ class (Figure 1275).

# 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

The following listings will be presented including Subject ID, Age (years) Adverse Event Description, Adverse Event Onset Date/End Date, Last Dose Received/Days Post Dose, Reason Reported as an SAE, Relationship to Treatment, Alternate Etiology if not Related, Outcome, and Duration of Event (days):

- Deaths and Serious Adverse Events (Table 412);
- Adverse Events of Special Interest, New Onset Chronic Medical Conditions and Medically Attended Adverse Events (Table 414).

## 9.5. Pregnancies

For any subjects in the Safety population who became pregnant during the study, every attempt will be made to follow these subjects to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery. A listing of pregnancies and outcomes will be presented (Listing 16, Listing 17, Listing 18, Listing 19, and Listing 20).

# 9.6. Clinical Laboratory Evaluations

Not applicable.

# 9.7. Vital Signs and Physical Evaluations

Vital sign measurements included systolic blood pressure, diastolic blood pressure, pulse, and oral temperature. Vital signs were assessed at Study Days 1, 15, 29, 43, 57, 71, 85, 147, 237, and 422 (Arms 2A-B) and Study Days 1, 15, 29, 43, 57, 119, 209, and 394 (Arms 2C-H). Vital signs will be tabulated by visit and Treatment Group starting with Table 415 and ending with Table 424 (Listing 13).

Physical Examinations were only to be performed if clinically indicated at Study Days 1, 15, 29, 43, 57, 71, 85, 147, 237, and 422 (Arms 2A-B) and Study Days 1, 15, 29, 43, 57, 119, 209, and 394 (Arms 2C-H). The following body systems will be assessed: Abdomen, Cardiovascular/heart, Extremities, General Appearance, Hepatobiliary/spleen, HEENT, Lymph nodes, Musculoskeletal, Neck, Neurological, Pulmonary/Chest, and Skin (Listing 14).

## 9.8. Concomitant Medications

Concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study will be recorded on the CRFs. A by-subject listing of concomitant medication use will be presented (Listing 15). The use of concomitant medications during the study will be summarized by ATC1, ATC2 code and Treatment Group for the Safety population (Table 425).

## 9.9. Other Safety Measures

Not applicable.

# 10. PHARMACOKINETICS

Not applicable.

## 11. IMMUNOGENICITY

See Section 8.

# 12. OTHER ANALYSES

Not Applicable.

## 13. REPORTING CONVENTIONS

The mean, standard deviation, and other statistics will be reported to 1 decimal place greater than the original data. The minimum and maximum will use the same number of decimal places as the original data. Proportions will be presented as 2 decimal places; values greater than zero but <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; values greater than zero but < 1% will be presented as "<1"; values greater than 99% but less than 100% will be reported as >99%. Estimated parameters, not on the same scale as raw observations (e.g., regression coefficients) will be reported to 3 significant figures.

# 14. TECHNICAL DETAILS

SAS version 9.4 and R 3.6.2 or above will be used to generate all tables, figures and listings.

# 15. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

Not Applicable.

## 16. REFERENCES

- Anderson, E. J., Rouphael, N. G., Widge, A. T., Jackson, L. A., Roberts, P. C., Makhene, M., Chappell, J. D., Denison, M. R., Stevens, L. J., Pruijssers, A. J., McDermott, A. B., Flach, B., Lin, B. C., Doria-Rose, N. A., O'Dell, S., Schmidt, S. D., Corbett, K. S., Swanson, P. A., 2nd, Padilla, M., Neuzil, K. M., ... mRNA-1273 Study Group (2020). Safety and Immunogenicity of SARS-CoV-2 mRNA-1273 Vaccine in Older Adults. The New England Journal of Medicine, 383(25), 2427–2438. https://doi.org/10.1056/NEJMoa2028436.
- 2. Callaway, E. & Mallapaty, S. (2021). Novavax offers first evidence that COVID vaccines protect people against variants. Nature, 10.1038/d41586-021-00268-9. Advance online publication. https://doi.org/10.1038/d41586-021-00268-9.
- 3. Center for Systems Science and Engineering (CCSE) at Johns Hopkins University (JHU). COVID-19 Dashboard. 2020. https://coronavirus.jhu.edu/map.html. Accessed 04 Feb 2021.
- 4. Chu L., McPhee R., Huang W., Bennett H., Pajon R., Nestorova B., Leav B., ... mRNA-1273 Study Group (2021). A Preliminary Report of a Randomized Controlled Phase 2 Trial of the Safety and Immunogenicity of mRNA-1273 SARS-CoV-2 Vaccine. Vaccine. Advance online publication. https://doi.org/10.1016/j.vaccine.2021.02.007.
- 5. Corbett, K. S., Edwards, D. K., Leist, S. R., Abiona, O. M., Boyoglu-Barnum, S., Gillespie, R. A., Himansu, S., Schäfer, A., Ziwawo, C. T., DiPiazza, A. T., Dinnon, K. H., Elbashir, S. M., Shaw, C. A., Woods, A., Fritch, E. J., Martinez, D. R., Bock, K. W., Minai, M., Nagata, B. M., Hutchinson, G. B., ... Graham, B. S. (2020). SARS-CoV-2 mRNA vaccine design enabled by prototype pathogen preparedness. Nature, 586(7830), 567–571. https://doi.org/10.1038/s41586-020-2622-0
- 6. Drummond R. CONSORT Revised: Improving the Reporting of Randomized Clinical Trials. JAMA. 2001; 285(15): 2006-2007.
- 7. Jackson, L. A., Anderson, E. J., Rouphael, N. G., Roberts, P. C., Makhene, M., Coler, R. N., McCullough, M. P., Chappell, J. D., Denison, M. R., Stevens, L. J., Pruijssers, A. J., McDermott, A., Flach, B., Doria-Rose, N. A., Corbett, K. S., Morabito, K. M., O'Dell, S., Schmidt, S. D., Swanson, P. A., 2nd, Padilla, M., ... mRNA-1273 Study Group (2020). An mRNA Vaccine against SARS-CoV-2 Preliminary Report. The New England Journal of Medicine, 383(20), 1920–1931. https://doi.org/10.1056/NEJMoa2022483.
- 8. Tegally H, Wilkinson E, Giovanetti M, Iranzadeh A, Fonseca V, Giandhari J, Doolabh D, Pillay S, San EJ, Msomi N, et al. Emergence and rapid spread of a new severe acute respiratory syndrome-related coronavus 2 (SARS-CoV-2) lineage with multiple spike mutations in South Africa. MedRxiv 2020.12.21.20248640.
- 9. Wang P, Liu L, Iketani S, et al. Increased resistance of SARS-CoV-2 variants B.1.351 and B.1.1.7 to antibody neutralization. bioRxiv: the preprint server for biology, 2021.01.428137. https://doi.org/10.1101/2021.01.25.428137.
- 10. World Health Organization (WHO). (Data reported as of 13 Nov 2020). Weekly Operational Update on COVID-19. 2020a.
- https://www.who.int/publications/m/item/weekly-operational-update-on-covid-19---13-november-2020. Accessed 04 Feb 2021.
- 11. Wu, K., Werner, A. P., Moliva, J. I., Koch, M., Choi, A., Stewart-Jones, G., Bennett, H., Boyoglu-Barnum, S., Shi, W., Graham, B. S., Carfi, A., Corbett, K. S., Seder, R. A., & Edwards, D. K. (2021). mRNA-1273 vaccine induces neutralizing antibodies against spike mutants from global SARS-CoV-2 variants. bioRxiv: the preprint server for biology, 2021.01.25.427948. https://doi.org/10.1101/2021.01.25.427948.

## APPENDIX 1. TABLE MOCK-UPS

## LIST OF TABLES

| Table 1: | Study Design. | 75 |
|---|---|---|
| Table 2: | Schedule of Study Procedures for Treatment Arms 2A-B (Three Vaccinations) | 76 |
| Table 3: | Schedule of Study Procedures for Treatment Arms 2C-H (Two Vaccinations) | 77 |
| Table 4: | Sample Size/Probability Estimates | 78 |
| Table 5: | Distribution of Protocol Deviations by Category, Type, and Treatment Group | 79 |
| Table 6: | Distribution of Major Protocol Deviations by Category, Type, and Treatment Group | 80 |
| Table 7: | Subject Disposition by Treatment Group for Arms 2A-B (Three Vaccinations) | 81 |
| Table 8: | Subject Disposition by Treatment Group for Arms 2C-H (Two Vaccinations) | 82 |
| Table 9: | Analysis Populations by Treatment Group - Treatment Arms 2A-B (Three Vaccinations) | 83 |
| Table 10: | Analysis Populations by Treatment Group - Treatment Arms 2C-H (Two Vaccinations) | 85 |
| Table 11: | Ineligibility Summary of Screen Failures | 87 |
| Table 12: | Summary of Categorical Demographic and Baseline Characteristics by Treatment Group | 88 |
| Table 13: | Summary of Continuous Demographic and Baseline Characteristics by Treatment Group | 89 |
| Table 14: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group | 91 |
| Table 15: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 92 |
| Table 16: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Results with 95% Confidence Intervals by Time Point and<br>Treatment Group, S-2P–Wa-1 – Per Protocol Population, Treatment Arms<br>2A-B (Three Vaccinations) | 94 |
| Table 17: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Results with 95% Confidence Intervals by Time Point and | |

| | Treatment Group, RBD–Wa-1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 94 |
|---|---|---|
| Table 18: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Results with 95% Confidence Intervals by Time Point and<br>Treatment Group, RBD–Wa-1 – Per Protocol Population, Treatment Arms<br>2A-B (Three Vaccinations) | 94 |
| Table 19: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 94 |
| Table 20: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 94 |
| Table 21: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 94 |
| Table 22: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 94 |
| Table 23: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 94 |
| Table 24: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 94 |
| Table 25: | Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 94 |
| Table 26: | Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 94 |
| Table 27: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time | |

| | Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 95 |
|---|---|---|
| Table 28: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 95 |
| Table 29: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 95 |
| Table 30: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 95 |
| Table 31: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.617.2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 95 |
| Table 32: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.617.2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 95 |
| Table 33: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 95 |
| Table 34: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 95 |
| Table 35: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.7 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 95 |
| Table 36: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.7 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 95 |
| Table 37: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time | |

| | Point and Treatment Group, S-2P–B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 96 |
|---|---|---|
| Table 38: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 96 |
| Table 39: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 97 |
| Table 40: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Results with 95% Confidence Intervals by Time Point and<br>Treatment Group, S-2P-Wa-1 – Per Protocol Population, Treatment Arms<br>2C-H (Two Vaccinations) | 99 |
| Table 41: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Results with 95% Confidence Intervals by Time Point and<br>Treatment Group, RBD–Wa-1 – mITT Population, Treatment Arms 2C-H<br>(Two Vaccinations) | 99 |
| Table 42: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Results with 95% Confidence Intervals by Time Point and<br>Treatment Group, RBD–Wa-1 – Per Protocol Population, Treatment Arms<br>2C-H (Two Vaccinations) | 99 |
| Table 43: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 99 |
| Table 44: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 99 |
| Table 45: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 99 |
| Table 46: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 99 |
| Table 47: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time | |

| | Point and Treatment Group, RBD–B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 99 |
|---|---|---|
| Table 48: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 99 |
| Table 49: | Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 99 |
| Table 50: | Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 100 |
| Table 51: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 100 |
| Table 52: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 100 |
| Table 53: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 100 |
| Table 54: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 100 |
| Table 55: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.617.2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 100 |
| Table 56: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.617.2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 100 |
| Table 57: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time | |

| | Point and Treatment Group, S-2P–P.1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations). | 100 |
|---|---|---|
| Table 58: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 100 |
| Table 59: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.7 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 100 |
| Table 60: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.7 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 101 |
| Table 61: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 101 |
| Table 62: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 101 |
| Table 63: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 102 |
| Table 64: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 103 |
| Table 65: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 103 |
| Table 66: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 103 |
| Table 67: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 103 |
| Table 68: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 104 |

| Table 69: Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Result Confidence Intervals by Time Point and Treatment Group, B.1 Population, Treatment Arms 2A-B (Three Vaccinations) | .351 - mITT |
|---|---|
| Table 70: Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Result Confidence Intervals by Time Point and Treatment Group, B.1 Protocol Population, Treatment Arms 2A-B (Three Vaccination | .351 – Per |
| Table 71: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Result Confidence Intervals by Time Point and Treatment Group, B.1 mITT Population, Treatment Arms 2A-B (Three Vaccinations) | .617.2 – |
| Table 72: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Result Confidence Intervals by Time Point and Treatment Group, B.1 Protocol Population, Treatment Arms 2A-B (Three Vaccination | .617.2 – Per |
| Table 73: Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Result Confidence Intervals by Time Point and Treatment Group, B.1 mITT Population, Treatment Arms 2A-B (Three Vaccinations) | .617.2 – |
| Table 74: Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Result Confidence Intervals by Time Point and Treatment Group, B.1 Protocol Population, Treatment Arms 2A-B (Three Vaccination | .617.2 – Per |
| Table 75: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Result Confidence Intervals by Time Point and Treatment Group, P.1 Population, Treatment Arms 2A-B (Three Vaccinations) | – mITT |
| Table 76: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Result Confidence Intervals by Time Point and Treatment Group, P.1 Protocol Population, Treatment Arms 2A-B (Three Vaccination | – Per |
| Table 77: Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Result Confidence Intervals by Time Point and Treatment Group, P.1 Population, Treatment Arms 2A-B (Three Vaccinations) | – mITT |
| Table 78: Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Result Confidence Intervals by Time Point and Treatment Group, P.1 Protocol Population, Treatment Arms 2A-B (Three Vaccination | – Per |
| Table 79: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Result Confidence Intervals by Time Point and Treatment Group, B.1 Population, Treatment Arms 2A-B (Three Vaccinations) | .1.7 - mITT |
| Table 80: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Result Confidence Intervals by Time Point and Treatment Group, B.1 Protocol Population, Treatment Arms 2A-B (Three Vaccination | ts with 95%<br>.1.7 – Per |
| Table 81: Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Result Confidence Intervals by Time Point and Treatment Group, B.1 Population, Treatment Arms 2A-B (Three Vaccinations) | ts with 95%<br>.1.7 – mITT |

| Table 82: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 105 |
|---|---|---|
| Table 83: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 105 |
| Table 84: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 105 |
| Table 85: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 105 |
| Table 86: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 105 |
| Table 87: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 106 |
| Table 88: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 108 |
| Table 89: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 108 |
| Table 90: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 108 |
| Table 91: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 108 |
| Table 92: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 108 |
| Table 93: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 108 |
| Table 94: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Table 95: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 108 |
|---|---|---|
| Table 96: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 108 |
| Table 97: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 108 |
| Table 98: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 108 |
| Table 99: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 108 |
| Table 100: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 108 |
| Table 101: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 109 |
| Table 102: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 109 |
| Table 103: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 109 |
| Table 104: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 109 |
| Table 105: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 109 |
| Table 106: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Table 107: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Table 108: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 19 |
|---|---|---|
| Table 109: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 19 |
| Table 110: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 19 |
| Table 111: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations)11 | 0 |
| Table 112: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)11 | 2 |
| Table 113: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 2 |
| Table 114: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 2 |
| Table 115: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)11 | 2 |
| Table 116: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)11 | 2 |
| Table 117: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 2 |
| Table 118: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 2 |
| Table 119: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Table 120: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Table 121: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 112 |
|---|---|---|
| Table 122: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 112 |
| Table 123: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 112 |
| Table 124: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 113 |
| Table 125: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 113 |
| Table 126: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 113 |
| Table 127: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 113 |
| Table 128: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 113 |
| Table 129: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 113 |
| Table 130: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 113 |
| Table 131: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 113 |
| Table 132: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 113 |
| Table 133: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Table 134: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
|---|---|
| Table 135: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations)113 |
| Table 136: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 137: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations)113 |
| Table 138: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 139: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)114 |
| Table 140: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 141: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)114 |
| Table 142: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 143: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)114 |
| Table 144: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 145: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)114 |

| Table 146: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three | |
|---|---|---|
| | Vaccinations) | 114 |
| Table 147: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 115 |
| Table 148: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 117 |
| Table 149: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 117 |
| Table 150: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 117 |
| Table 151: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 117 |
| Table 152: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 117 |
| Table 153: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 117 |
| Table 154: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Table 155: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 117 |
| Table 156: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 117 |
| Table 157: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 117 |
| Table 158: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Table 159: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations)117 |
|---|---|
| Table 160: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 161: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 162: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 163: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 164: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)118 |
| Table 165: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 166: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 167: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 168: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 169: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 170: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 171: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations)118 |

| Table 172: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
|---|---|
| Table 173: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations)118 |
| Table 174: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 175: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations)119 |
| Table 176: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 177: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations)119 |
| Table 178: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 179: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean |
| | Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations)119 |
| Table 180: | Results with 95% Confidence Intervals by Time Point and Treatment Group, |
| | Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations)119 Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two |
| Table 181: | Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations)119 Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |

| Table 184: | Percentages of CD4 T Cells Expressing Cytokines with 95% CI – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 126 |
|---|---|---|
| Table 185: | Percentages of CD4 T Cells Expressing Cytokines with 95% CI – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 127 |
| Table 186: | Percentages of CD4 T Cells Expressing Cytokines with 95% CI – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 133 |
| Table 187: | Percentages of CD8 T Cells Expressing Cytokines with 95% CI – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 134 |
| Table 188: | Percentages of CD8 T Cells Expressing Cytokines with 95% CI – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 136 |
| Table 189: | Percentages of CD8 T Cells Expressing Cytokines with 95% CI – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 137 |
| Table 190: | Percentages of CD8 T Cells Expressing Cytokines with 95% CI – Per<br>Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 139 |
| Table 191: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 140 |
| Table 192: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence<br>Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol<br>Population, Treatment Arms 2A-B (Three Vaccinations) | 142 |
| Table 193: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence<br>Intervals by Time Point and Treatment Group, RBD–Wa-1 – mITT<br>Population, Treatment Arms 2A-B (Three Vaccinations) | 142 |
| Table 194: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence<br>Intervals by Time Point and Treatment Group, RBD–Wa-1 – Per Protocol<br>Population, Treatment Arms 2A-B (Three Vaccinations) | 142 |
| Table 195: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 142 |
| Table 196: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 142 |
| Table 197: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% | |

| | Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
|---|---|
| Table 198: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 199: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 200: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 201: | Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P—Wa-1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)143 |
| Table 202: | Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 203: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 204: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 205: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 206: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 207: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% |

| | Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.617.2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
|---|---|
| Table 208: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.617.2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)143 |
| Table 209: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 210: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 211: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.7 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 212: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.7 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 213: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 214: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)144 |
| Table 215: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 216: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 217: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence |

| | Intervals by Time Point and Treatment Group, RBD–Wa-1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
|---|---|
| Table 218: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–Wa-1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 219: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 220: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 221: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 222: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 223: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 224: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 225: | Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 226: | Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 227: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% |

| | Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
|---|---|
| Table 228: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 229: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 230: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 231: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.617.2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 232: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.617.2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 233: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 234: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 235: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.7 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 236: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.7 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 237: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% |

| | Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
|---|---|
| Table 238: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 239: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 240: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 241: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 242: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 243: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 244: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 245: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 246: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Table 247: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and |

| | Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 152 |
|---|---|---|
| Table 248: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 152 |
| Table 249: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 152 |
| Table 250: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 152 |
| Table 251: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 152 |
| Table 252: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 152 |
| Table 253: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 152 |
| Table 254: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 152 |
| Table 255: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 152 |
| Table 256: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 152 |
| Table 257: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and | |

| | Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 152 |
|---|---|---|
| Table 258: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 152 |
| Table 259: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 152 |
| Table 260: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 153 |
| Table 261: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 153 |
| Table 262: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 153 |
| Table 263: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 154 |
| Table 264: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 155 |
| Table 265: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 155 |
| Table 266: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 155 |
| Table 267: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and | |

| | Treatment Group, B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 155 |
|---|---|---|
| Table 268: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 155 |
| Table 269: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 156 |
| Table 270: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 156 |
| Table 271: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 156 |
| Table 272: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 156 |
| Table 273: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 156 |
| Table 274: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 156 |
| Table 275: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 156 |
| Table 276: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 156 |
| Table 277: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and | |

| | Treatment Group, P.1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
|---|---|
| Table 278: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 279: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 280: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 281: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 282: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 283: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 284: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 285: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 286: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Table 287: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and |

| | Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 158 |
|---|---|---|
| Table 288: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 159 |
| Table 289: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 159 |
| Table 290: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 159 |
| Table 291: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 159 |
| Table 292: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 159 |
| Table 293: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 159 |
| Table 294: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 159 |
| Table 295: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 160 |
| Table 296: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 160 |
| Table 297: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and | |

| | Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 160 |
|---|---|---|
| Table 298: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 160 |
| Table 299: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 160 |
| Table 300: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 160 |
| Table 301: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 160 |
| Table 302: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 160 |
| Table 303: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 160 |
| Table 304: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 160 |
| Table 305: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 160 |
| Table 306: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 160 |
| Table 307: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and | |

| | Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 51 |
|---|---|---|
| Table 308: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 51 |
| Table 309: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 61 |
| Table 310: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 61 |
| Table 311: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 61 |
| Table 312: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 61 |
| Table 313: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 61 |
| Table 314: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 61 |
| Table 315: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 61 |
| Table 316: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 61 |
| Table 317: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by | |

| | Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 162 |
|---|---|---|
| Table 318: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 162 |
| Table 319: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 162 |
| Table 320: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 162 |
| Table 321: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 162 |
| Table 322: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 162 |
| Table 323: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 163 |
| Table 324: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 164 |
| Table 325: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 164 |
| Table 326: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 164 |
| Table 327: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and | |

| | Treatment Group, B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 164 |
|---|---|---|
| Table 328: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 164 |
| Table 329: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 164 |
| Table 330: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 164 |
| Table 331: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 165 |
| Table 332: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 165 |
| Table 333: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 165 |
| Table 334: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 165 |
| Table 335: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 165 |
| Table 336: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 165 |
| Table 337: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and | |

| | Treatment Group, P.1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 165 |
|---|---|---|
| Table 338: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 165 |
| Table 339: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 165 |
| Table 340: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 165 |
| Table 341: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 165 |
| Table 342: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 166 |
| Table 343: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 166 |
| Table 344: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 166 |
| Table 345: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 166 |
| Table 346: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 166 |
| Table 347: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by | |

| | Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 166 |
|---|---|---|
| Table 348: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 166 |
| Table 349: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 166 |
| Table 350: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 166 |
| Table 351: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 166 |
| Table 352: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 166 |
| Table 353: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 166 |
| Table 354: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 167 |
| Table 355: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 167 |
| Table 356: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 167 |
| Table 357: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by | |

| | Time Point and Treatment Group, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 167 |
|---|---|---|
| Table 358: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 167 |
| Table 359: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 168 |
| Table 360: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 175 |
| Table 361: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 175 |
| Table 362: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 175 |
| Table 363: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 176 |
| Table 364: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 182 |
| Table 365: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 182 |
| Table 366: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Table 367: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and | |

| | Treatment Group – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 183 |
|---|---|---|
| Table 368: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 190 |
| Table 369: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 190 |
| Table 370: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 190 |
| Table 371: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 191 |
| Table 372: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 194 |
| Table 373: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 194 |
| Table 374: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 194 |
| Table 375: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 195 |
| Table 376: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 200 |
| Table 377: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and | |

| | Treatment Group – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 200 |
|---|---|---|
| Table 378: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 200 |
| Table 379: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 201 |
| Table 380: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 203 |
| Table 381: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 203 |
| Table 382: | Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 203 |
| Table 383: | Summary of N-Antibody Expression and Self-Reported Infection Status by Time Point and Treatment Group – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 204 |
| Table 384: | Summary of N-Antibody Expression and Self-Reported Infection Status by Time Point and Treatment Group – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 206 |
| Table 385: | Summary of N-Antibody Expression and Self-Reported Infection Status by Time Point and Treatment Group – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 207 |
| Table 386: | Summary of N-Antibody Expression and Self-Reported Infection Status by Time Point and Treatment Group – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 209 |
| Table 387: | Overall Summary of Adverse Events by Treatment Group - All Subjects | 210 |
| Table 388: | Serious Adverse Events and Non-Serious Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - All Subjects | 212 |
| Table 389: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group | 213 |
| Table 390: | Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2A (Three Vaccinations) | 216 |
|---|---|---|
| Table 391: | Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2A (Three Vaccinations) | 219 |
| <b>Table 392:</b> | Summary of Solicited Events by Days Post Dose 3, Symptom, and Treatment Group – Treatment Arm 2A (Three Vaccinations) | 219 |
| Table 393: | Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2B (Three Vaccinations) | 219 |
| Table 394: | Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2B (Three Vaccinations) | 219 |
| Table 395: | Summary of Solicited Events by Days Post Dose 3, Symptom, and Treatment Group – Treatment Arm 2B (Three Vaccinations) | 219 |
| Table 396: | Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2C (Two Vaccinations) | 219 |
| Table 397: | Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2C (Two Vaccinations) | 219 |
| Table 398: | Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2D (Two Vaccinations) | 219 |
| Table 399: | Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2D (Two Vaccinations) | 219 |
| Table 400: | Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2E (Two Vaccinations) | 219 |
| Table 401: | Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2E (Two Vaccinations) | 219 |
| Table 402: | Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2F (Two Vaccinations) | 219 |
| Table 403: | Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2F (Two Vaccinations) | 219 |
| Table 404: | Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2G (Two Vaccinations) | 219 |
| Table 405: | Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2G (Two Vaccinations) | 219 |
| Table 406: | Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2H (Two Vaccinations) | 219 |
| Table 407: | Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2H (Two Vaccinations) | 219 |
| Table 408: | Summary of Number of Days of Solicited Symptoms by Treatment Group - All Subjects. | 220 |

| Table 409: | All Adverse Events Cross-Classified by MedDRA System Organ Class,<br>Severity, Relationship to Study Treatment, and Treatment Group | 224 |
|---|---|---|
| Table 410: | Summary of All Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship, and Treatment Group | 227 |
| Table 411: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Severity, Relationship, and Treatment Group | 228 |
| Table 412: | Listing of Serious Adverse Events | 230 |
| Table 413: | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events | 231 |
| Table 414: | Listing of AESIs, MAAEs, and NOCMCs | 232 |
| Table 415: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Any Assessment – All Subjects, Treatment Arms 2A-B (Three Vaccinations) | 234 |
| Table 416: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Systolic Blood Pressure – All Subjects, Treatment Arms 2A-B (Three Vaccinations) | 236 |
| Table 417: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Diastolic Blood Pressure – All Subjects, Treatment Arms 2A-B (Three Vaccinations) | 236 |
| Table 418: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Pulse Rate – All Subjects, Treatment Arms 2A-B (Three Vaccinations) | 236 |
| Table 419: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Temperature – All Subjects, Treatment Arms 2A-B (Three Vaccinations) | 236 |
| Table 420: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Any Assessment – All Subjects, Treatment Arms 2C-H (Two Vaccinations) | 237 |
| Table 421: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Systolic Blood Pressure – All Subjects, Treatment Arms 2C-H (Two Vaccinations) | 239 |
| Table 422: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Diastolic Blood Pressure – All Subjects, Treatment Arms 2C-H (Two Vaccinations) | 239 |
| Table 423: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Pulse Rate – All Subjects, Treatment Arms 2C-H (Two Vaccinations) | 239 |

| Table 424: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Temperature – All Subjects, Treatment Arms 2C-H (Two | |
|---|---|---|
| | Vaccinations) | 239 |
| Table 425: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group – All Subjects | 240 |

# 9.1 Overall Study Design and Plan Description

**Table 1:** Study Design

| A | Sample | First Vaccination | | Second Vaccination | Third Vaccination | |
|---|---|---|---|---|---|---|
| Arm | Size | <b>Product and Dose</b> | Interval | <b>Product and Dose</b> | Interval | <b>Product and Dose</b> |
| 2A | 15 | 100 mcg mRNA-1273 | 28 days | 100 mcg mRNA-1273 | 28 days | 50 mcg mRNA-<br>1273.351 |
| 2B | 15 | 50 mcg mRNA-1273 | 28 days | 50 mcg mRNA-1273 | 28 days | 50 mcg mRNA-<br>1273.351 |
| 2C | 20 | 100 mcg mRNA-1273.351 | 28 days | 100 mcg mRNA-1273.351 | | None |
| 2D | 20 | 50 mcg mRNA-1273.351 | 28 days | 50 mcg mRNA-1273.351 | | None |
| 2E | 20 | 100 mcg mRNA-1273 | 28 days | 100 mcg mRNA-1273.351 | | None |
| 2F | 20 | 50 mcg mRNA-1273 | 28 days | 50 mcg mRNA-1273.351 | | None |
| 2G | 20 | 50 mcg mRNA-1273<br>+ 50 mcg mRNA-1273.351 | 28 days | 50 mcg mRNA-1273<br>+ 50 mcg mRNA-1273.351 | | None |
| 2Н | 20 | 25 mcg mRNA-1273<br>+ 25 mcg mRNA-1273.351 | 28 days | 25 mcg mRNA-1273<br>+ 25 mcg mRNA-1273.351 | | None |

### 9.5.1 Efficacy/Immunogenicity and Safety Measurements Assessed and Flow Chart

**Table 2:** Schedule of Study Procedures for Treatment Arms 2A-B (Three Vaccinations)

| Study Day | -42 to -1 | 1 | 8* | 15 | 29 | 36* | 43 | 57 | 64* | 71 | 85 | 147 | 237 | 422 | Unsc<br>Visit | Early<br>Term<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Window (±number of days) | | 0 | 1 | 2 | 2 | 1 | 2 | 2 | 1 | 2 | 2 | 7 | 7 | 14 | | |
| Study Visit | Screening<br>(optional)<br>00 | 01 | 02 | 03 | 04 | 05° | 06e | 07e | 08 <sup>f</sup> | 09 <sup>f</sup> | 10 <sup>f</sup> | 11 <sup>f</sup> | 12 <sup>f</sup> | 13 <sup>f</sup> | | |
| Informed Consent | X | Xa | | | | | | | | | | | | | | |
| Review Eligibility Criteria | X | X | | | | | | | | | | | | | | |
| Medical History | X | Xa | | | | | | | | | | | | | | |
| Vaccination | | X | | | X | | | X | | | | | | | | |
| Concomitant Medications | | X | X | X | X | X | X | X | X | X | X | | | | | |
| Interim History | | $X^{b}$ | | X | X | | X | X | | X | X | X | X | X | X | X |
| Symptom-Directed Physical Examination | X | X | | X | X | | X | X | | X | X | X | X | X | X | X |
| Vital Signs <sup>c</sup> | | X | | X | X | | X | X | | X | X | X | X | X | X | X |
| Height and Weight (for BMI) | X | Xa | | | | | | | | | | | | | | |
| Pregnancy Test <sup>d</sup> | | X | | | X | | | X | | | | | | | | |
| Memory Aid: Solicited AEs | | X | X | Xg | X | X | $X^g$ | X | X | $X^g$ | | | | | | |
| Unsolicited AEs | | X | X | X | X | X | X | X | X | X | X | | | | | |
| SAEs, Protocol Specified AESIs,<br>MAAEs, and NOCMCs | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Serum for Serological Immunogenicity<br>Assays | | X | | X | X | | X | X | | X | X | X | X | X | | X |
| Peripheral Blood Mononuclear Cells<br>(PBMCs) for Cellular Immunology<br>Assays (and Plasma) | | X | | X | X | | X | X | | X | | | X | X | | X |

<sup>\*</sup> Telephone call.

- a) If not performed at Visit 00.
- b) If medical history performed at Visit 00, then interim history at Visit 01.
- c) Vital signs to be obtained pre and post vaccination. Otherwise, only as clinically indicated.
- d) For women of childbearing potential, a negative urine pregnancy test on Day 1 with results confirmed prior to enrollment.
- e) Visits 05-07 windows should be based off the actual Visit 04 date.
- f) Visits 08-13 windows should be based off the actual Visit 07 date.
- g) Collect Memory Aid and assess for delayed onset local reactions.

Table 3: Schedule of Study Procedures for Treatment Arms 2C-H (Two Vaccinations)

| Study Day | -42 to -1 | 1 | 8* | 15 | 29 | 36* | 43 | 57 | 119 | 209 | 394 | Unsc<br>Visit | Early<br>Term<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Window (±number of days) | | 0 | 1 | 2 | 2 | 1 | 2 | 2 | 7 | 7 | 14 | | |
| Study Visit | Screening<br>(optional)<br>00 | 01 | 02 | 03 | 04 | 05° | 06e | 07e | 08e | 09e | 10e | | |
| Informed Consent | X | Xa | | | | | | | | | | | |
| Review Eligibility Criteria | X | X | | | | | | | | | | | |
| Medical History | X | Xa | | | | | | | | | | | |
| Vaccination | | X | | | X | | | | | | | | |
| Concomitant Medications | | X | X | X | X | X | X | X | | | | | |
| Interim History | | $X^{b}$ | | X | X | | X | X | X | X | X | X | X |
| Symptom-Directed Physical Examination | X | X | | X | X | | X | X | X | X | X | X | X |
| Vital Signs <sup>c</sup> | | X | | X | X | | X | X | X | X | X | X | X |
| Height and Weight (for BMI) | X | Xa | | | | | | | | | | | |
| Pregnancy Test <sup>d</sup> | | X | | | X | | | | | | | | |
| Memory Aid: Solicited AEs | | X | X | $X^f$ | X | X | Xf | | | | | | |
| Unsolicited AEs | | X | X | X | X | X | X | X | | | | | |
| SAEs, Protocol Specified AESIs, MAAEs, and NOCMCs | | X | X | X | X | X | X | X | X | X | X | X | X |
| Serum for Serological Immunogenicity Assays | | X | | X | X | | X | X | X | X | X | | X |
| Peripheral Blood Mononuclear Cells (PBMCs) for<br>Cellular Immunology Assays (and Plasma) | | X | | X | X | | X | | | X | X | | X |

<sup>\*</sup> Telephone call.

- a) If not performed at Visit 00.
- b) If medical history performed at Visit 00, then interim history at Visit 01.
- c) Vital signs to be obtained pre and post vaccination. Otherwise, only as clinically indicated.
- d) For women of childbearing potential, a negative urine pregnancy test on Day 1 with results confirmed prior to enrollment.
- e) Visits 05-10 windows should be based off the actual Visit 04 date.
- f) Collect Memory Aid and assess for delayed onset local reactions.

# 9.7.1 Sample Size

 Table 4:
 Sample Size/Probability Estimates

| | | | | | Coh | ort 2 | | |
|---|---|---|---|---|---|---|---|---|
| N | "True"<br>Event<br>Rate | Probability of<br>Observation (%) | N | "True"<br>Event<br>Rate | Probability of<br>Observation (%) | N | "True"<br>Event<br>Rate | Probability of Observation (%) |
| | 0.1% | 1.5 | | 0.1% | 2.0 | | 0.1% | 13.9 |
| | 0.5% | 7.2 | | 0.5% | 9.5 | | 0.5% | 52.9 |
| | 1.0% | 14.0 | | 1.0% | 18.2 | | 1.0% | 77.9 |
| | 2.0% | 26.1 | | 2.0% | 33.2 | | 2.0% | 95.2 |
| 15 | 3.0% | 36.7 | 20 | 3.0% | 45.6 | 150 | 3.0% | 99.0 |
| 13 | 4.0% | 45.8 | 20 | 4.0% | 55.8 | 150 | 4.0% | 99.8 |
| | 5.0% | 53.7 | | 5.0% | 64.2 | | 5.0% | >99.9 |
| | 10.0% | 79.4 | | 10.0% | 87.8 | | 10.0% | >99.9 |
| | 15.0% | 91.3 | | 15.0% | 96.1 | | 15.0% | >99.9 |
| | 20.0% | 96.5 | | 20.0% | 98.8 | | 20.0% | >99.9 |

## **10.2** Protocol Deviations

Table 5: Distribution of Protocol Deviations by Category, Type, and Treatment Group

[Implementation Note: Below are example categories and deviation types. All reported categories and deviations types will be presented.]

| | | Arm<br>(N= | | | n 2B<br>=X) | | 1 2C<br>=X) | Arn<br>(N= | 1 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | n 2G<br>=X) | | 1 2H<br>=X) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation<br>Type | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. |
| Follow-up visit schedule | Missed<br>visit/visit not<br>conducted | | | | | | | | | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | | | | | | | | | |
| Protocol<br>procedure/assessmen<br>t | Other: breach of confidentiality | | | | | | | | | | | | | | | | | | |
| | Other: non-<br>required lab<br>tests<br>performed | | | | | | | | | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | | | | | | | | | |
| | Required procedure not conducted | | | | | | | | | | | | | | | | | | |
| | Specimen<br>result not<br>obtained | | | | | | | | | | | | | | | | | | |
| | Too few aliquots obtained | | | | | | | | | | | | | | | | | | |

| Category Deviation | | Arm<br>(N= | | Arm 2B Arm 2C (N=X) (N=X) | | Arn<br>(N= | n 2D<br>=X) | Arm 2E<br>(N=X) | | Arm 2F<br>(N=X) | | Arm 2G<br>(N=X) | | Arm 2H<br>(N=X) | | All Subjects<br>(N=X) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation<br>Type | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. |
| Freatment<br>administration<br>schedule | Required procedure done incorrectly | | | | | | | | | | | | | | | | | | |
| Note: N=Number of sub | v | Populatio | on . | | | | | | | | | | | | | | | | |

Table with Similar Format:

Table 6: Distribution of Major Protocol Deviations by Category, Type, and Treatment Group

## 14.1 Description of Study Subjects

## 14.1.1 Disposition of Subjects

**Table 7:** Subject Disposition by Treatment Group for Arms 2A-B (Three Vaccinations)

| | | rm 2A<br>N=X) | | Arm 2B<br>(N=X) | | Subjects<br>N=X) |
|---|---|---|---|---|---|---|
| Subject Disposition | n | % | n | % | n | % |
| Screened | | | | | | |
| Enrolled | | | | | | |
| Received dose 1 | | | | | | |
| Received dose 2 | | | | | | |
| Received dose 3 | | | | | | |
| Early termination <sup>a</sup> | | | | | | |
| Completed study | | | | | | |

<sup>a</sup>Refer to Listing 2 for reasons subjects discontinued or terminated early.

Note: N=Number of subjects in the Safety Population

Table 8: Subject Disposition by Treatment Group for Arms 2C-H (Two Vaccinations)

| | | n 2C<br>=X) | | n 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | 1 2G<br>=X) | Arn<br>(N= | 1 2H<br>=X) | Sub | All<br>jects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject Disposition | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Screened | | | | | | | | | | | | | | |
| Enrolled | | | | | | | | | | | | | | |
| Received dose 1 | | | | | | | | | | | | | | |
| Received dose 2 | | | | | | | | | | | | | | |
| Early termination <sup>a</sup> | | | | | | | | | | | | | | |
| Completed study | | | | | | | | | | | | | | |

<sup>a</sup>Refer to Listing 2 for reasons subjects discontinued or terminated early.

Note: N=Number of subjects in the Safety Population

Table 9: Analysis Populations by Treatment Group - Treatment Arms 2A-B (Three Vaccinations)

| Analysis<br>Populations | Reason Subjects Excluded | Arm<br>(N= | | Arm<br>(N= | | All Sub<br>(N= | = |
|---|---|---|---|---|---|---|---|
| | | % | n | % | n | 0/0 | n |
| Safety | Did not receive one dose of the vaccine | х | XX | Х | XX | X | XX |
| Modified<br>Intent-To-<br>Treat | Any Reason | | | | | | |
| | Did not contribute a pre-<br>vaccination blood sample for<br>which valid immunogenicity<br>results were reported | | | | | | |
| | Did not contribute at least one post-vaccination blood sample for which valid immunogenicity results were reported | | | | | | |
| Per Protocol | Any Timepoint | | | | | | |
| | Found to be ineligible at baseline <sup>a</sup> | | | | | | |
| | Protocol deviation considered to affect the science <sup>b</sup> | | | | | | |
| | Visit occurred substantially out of window <sup>c</sup> | | | | | | |
| | Prior to or at Day 1 visit (visit 01): | | | | | | |
| | Found to be ineligible at baseline <sup>a</sup> | | | | | | |
| | Protocol deviation considered to affect the science <sup>b</sup> | | | | | | |
| | Visit occurred substantially out of window <sup>c</sup> | | | | | | |
| | Repeat Day 1 for: | | | | | | |

| Analysis<br>Populations | Reason Subjects Excluded | Arm<br>(N= | | Arm<br>(N= | | All Subj<br>(N=X | |
|---|---|---|---|---|---|---|---|
| | | % | n | % | n | % | n |
| | Prior to or at Day 15 visit (visit 03): | | | | | | |
| | Prior to or at Day 29 visit (visit 04): | | | | | | |
| | Prior to or at Day 43 visit (visit 06): | | | | | | |
| | Prior to or at Day 57 visit (visit 07): | | | | | | |
| | Prior to or at Day 71 visit (visit 09): | | | | | | |
| | Prior to or at Day 85 visit (visit 10): | | | | | | |
| | Prior to or at Day 147 visit (visit 11): | | | | | | |
| | Prior to or at Day 237 visit (visit 12): | | | | | | |
| | Prior to or at Day 422 visit (visit 13): | | | | | | |

Notes: N=Number of subjects enrolled. n=Number of subjects meeting the criteria.

Subjects may be excluded from an analysis population for multiple reasons.

<sup>&</sup>lt;sup>a</sup> Subject data from all visits are excluded from the per protocol analyses. All instances of exclusion are summarized in this table.

<sup>&</sup>lt;sup>b</sup> Subject data are excluded from the per protocol analyses at all timepoints subsequent to the occurrence of this protocol deviation. All instances of exclusion are summarized in this table. Subject data collected up to the time the exclusionary criterion is met is eligible for analysis.

<sup>c</sup> Only data from the out of window visit are excluded from the per protocol analyses.

 Table 10:
 Analysis Populations by Treatment Group - Treatment Arms 2C-H (Two Vaccinations)

| Analysis<br>Populations | Reason Subjects Excluded | | n 2C<br>=X) | | n 2D<br>=X) | | m 2E<br>=X) | | n 2F<br>=X) | | n 2G<br>=X) | | n 2H<br>=X) | | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | % | n | % | n | % | n | % | n | % | n | % | n | % | n |
| Safety | Did not receive one dose of the vaccine | х | XX | Х | XX | х | XX | Х | xx | Х | XX | х | XX | X | xx |
| Modified Intent-<br>To-Treat | Any Reason | | | | | | | | | | | | | | |
| | Did not contribute a pre-vaccination<br>blood sample for which valid<br>immunogenicity results were reported | | | | | | | | | | | | | | |
| | Did not contribute at least one post-<br>vaccination blood sample for which<br>valid immunogenicity results were<br>reported | | | | | | | | | | | | | | |
| Per Protocol | Any Timepoint | | | | | | | | | | | | | | |
| | Found to be ineligible at baseline <sup>a</sup> | | | | | | | | | | | | | | |
| | Protocol deviation considered to affect<br>the science <sup>b</sup> | | | | | | | | | | | | | | |
| | Visit occurred substantially out of window <sup>c</sup> | | | | | | | | | | | | | | |
| | Prior to or at Day 1 visit (visit 01): | | | | | | | | | | | | | | |
| | Found to be ineligible at baseline <sup>a</sup> | | | | | | | | | | | | | | |
| | Protocol deviation considered to affect<br>the science <sup>b</sup> | | | | | | | | | | | | | | |
| | Visit occurred substantially out of window <sup>c</sup> | | | | | | | | | | | | | | |
| | Repeat Day 1 for: | | | | | | | | | | | | | | |
| | Prior to or at Day 15 visit (visit 03): | | | | | | | | | | | | | | |
| | Prior to or at Day 29 visit (visit 04): | | | | | | | | | | | | | | |
| | Prior to or at Day 43 visit (visit 06): | | | | | | | | | | | | | | |

| Analysis<br>Populations | Reason Subjects Excluded | | n 2C<br>=X) | | n 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | 1 2G<br>=X) | | 1 2H<br>=X) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | % | n | % | n | % | n | % | n | % | n | % | n | % | n |
| | Prior to or at Day 57 visit (visit 07): | | | | | | | | | | | | | | |
| | Prior to or at Day 91 visit (visit 09): | | | | | | | | | | | | | | |
| | Prior to or at Day 209 visit (visit 10): | | | | | | | | | | | | | | |
| | Prior to or at Day 394 visit (visit 11): | | | | | | | | | | | | | | |

Notes: N=Number of subjects enrolled.

n=Number of subjects meeting the criteria.

Subjects may be excluded from an analysis population for multiple reasons.

<sup>&</sup>lt;sup>a</sup> Subject data from all visits are excluded from the per protocol analyses. All instances of exclusion are summarized in this table.

<sup>&</sup>lt;sup>b</sup> Subject data are excluded from the per protocol analyses at all timepoints subsequent to the occurrence of this protocol deviation. All instances of exclusion are summarized in this table. Subject data collected up to the time the exclusionary criterion is met is eligible for analysis.

<sup>°</sup> Only data from the out of window visit are excluded from the per protocol analyses.

**Table 11:** Ineligibility Summary of Screen Failures

| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | n <sup>a</sup> | % b |
|---|---|---|---|
| Inclusion and Exclusion | Number of subjects failing any eligibility criterion | X | 100 |
| Inclusion | Any inclusion criterion | X | XX |
| | [inclusion criterion 1] | X | XX |
| | [inclusion criterion 2] | X | XX |
| | [inclusion criterion 3] | X | XX |
| Exclusion | Any exclusion criterion | X | XX |
| | [exclusion criterion 1] | X | XX |
| | [exclusion criterion 2] | X | XX |
| | [exclusion criterion 3] | X | XX |

<sup>&</sup>lt;sup>a</sup> More than one criterion may be marked per subject.

<sup>&</sup>lt;sup>b</sup> Denominator for percentages is the total number of screen failures.

## 14.1.2 Demographic Data by Treatment Group

Table 12: Summary of Categorical Demographic and Baseline Characteristics by Treatment Group

| | | | m 2A<br>=X) | | n 2B<br>=X) | | n 2C<br>=X) | | n 2D<br>=X) | | m 2E<br>=X) | | n 2F<br>=X) | | n 2G<br>=X) | | n 2H<br>=X) | Sub | all<br>jects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Demographic<br>Category | Characteristic | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Sex | Male | | | | | | | | | | | | | | | | | | |
| | Female | | | | | | | | | | | | | | | | | | |
| Ethnicity | Not Hispanic or<br>Latino | | | | | | | | | | | | | | | | | | |
| | Hispanic or Latino | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | | | | | |
| Race | American Indian or<br>Alaska Native | | | | | | | | | | | | | | | | | | |
| | Asian | | | | | | | | | | | | | | | | | | |
| | Native Hawaiian or other Pacific Islander | | | | | | | | | | | | | | | | | | |
| | Black | | | | | | | | | | | | | | | | | | |
| | White | | | | | | | | | | | | | | | | | | |
| | Multi Racial | | | | | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | | | | | |
| Baseline N- | Negative | | | | | | | | | | | | | | | | | | |
| antibody status | Positive | | | | | | | | | | | | | | | | | | |

Table 13: Summary of Continuous Demographic and Baseline Characteristics by Treatment Group

| Variable | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| Age (Years) | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| Height (cm) | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| Weight (kg) | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| BMI (kg/m²) | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |

| Variable | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| | Maximum | | | | | | | | | |
| Note: N=Number of subjects | in the Safety Populat | ion | | | | | | | | |

### 14.1.3 Prior and Concurrent Medical Conditions

Table 14: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group

| MedDRA System Organ<br>Class | Arm<br>(N= | | | m 2B<br>=X) | | n 2C<br>=X) | | 1 2D<br>=X) | | 1 2E<br>=X) | Arn<br>(N= | n 2F<br>=X) | | n 2G<br>=X) | | 1 2H<br>=X) | | ibjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any SOC | X | XX | х | XX | X | XX | X | xx | X | XX | X | XX | X | XX | X | XX | Х | XX |
| [SOC 1] | | | | | | | | | | | | | | | | | | |
| [SOC 2] | | | | | | | | | | | | | | | | | | |

Note: N = Number of subjects in the Safety Population; n = Number of subjects reporting medical history within the specified SOC. A subject is only counted once per SOC.

### 14.2 Immunogenicity Data

Table 15: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)

| Planned Time Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects |
|---|---|---|---|---|
| Day 1, Pre-Dose | n | (11, 11) | (11.11) | |
| | GM | | | |
| | 95% CI | | | |
| Day 15 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 29 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 43 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 57 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 71 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 85 | n | | | |
| | GM | | | |

| Planned Time Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects |
|---|---|---|---|---|
| | 95% CI | , , | | |
| Day 147 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 237 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 422 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Peak GM | n | | | |
| | GM | | | |
| | 95% CI | | | |

Notes: N=Number of subjects in the mITT population.

n=Number of subjects with results available at time point.

GM=Geometric Mean, NE=Not Estimable.

Confidence intervals of the geometric means were calculated with the Student's t distribution on log-transformed data.

#### Tables with Similar Format:

Implementation notes:

For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

For all AUC tables, add footnote reading: "Geometric Mean is calculated as the Williams mean using log(1+x)."

- Table 16: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 17: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-Wa-1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 18: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-Wa-1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 19: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 20: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 21: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 22: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 23: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 24: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 25: Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 26: Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Table 27: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 28: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 29: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 30: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 31: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.617.2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 32: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.617.2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 33: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-P.1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 34: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 35: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.7 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 36: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.7 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Table 37: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 38: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Table 39: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations)

| Planned Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Day 1, Pre-Dose | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 15 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 29 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 43 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 57 | n | | | | | | | |
| - | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 119 | n | | | | | | | |
| · | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 209 | n | | | | | | | |
| · | GM | | | | 1 | 1 | | |

| Planned Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| | 95% CI | | | | | | | |
| Day 394 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Peak GM | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |

Notes: N=Number of subjects in the mITT population. n=Number of subjects with results available at time point. GM=Geometric Mean, NE=Not Estimable.

Confidence intervals of the geometric means were calculated with the Student's t distribution on log-transformed data.

#### Tables with Similar Format:

[Implementation notes: For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population." For all AUC tables, add footnote reading: "Geometric Mean is calculated as the Williams mean using log(1+x)."]

- Table 40: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 41: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-Wa-1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 42: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-Wa-1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 43: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 44: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 45: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 46: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 47: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 48: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD– B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 49: Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Table 50: Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 51: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 52: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 53: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 54: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 55: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.617.2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 56: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.617.2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 57: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-P.1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 58: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 59: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.7 mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Table 60: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.7 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 61: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 62: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Table 63: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations)

| Planned Time Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects |
|---|---|---|---|---|
| Day 1, Pre-Dose | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 15 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 29 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 43 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 57 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 71 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 85 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 147 | n | | | |

| Planned Time Point | Statistic | Arm 2A | Arm 2B | All Subjects |
|--------------------|-----------|--------|--------|--------------|
| | GM | (N=X) | (N=X) | |
| | 95% CI | | | |
| Day 237 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 422 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Peak GM | n | | | |
| | GM | | | |
| | 95% CI | | | |

Notes: N=Number of subjects in the mITT population.

n=Number of subjects with results available at time point.

GM=Geometric Mean, NE=Not Estimable.

Confidence intervals of the geometric means were calculated with the Student's t distribution on log-transformed data.

#### Tables with Similar Format:

[Implementation note: For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."]

- Table 64: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 65: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 66: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 67: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Table 68: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 69: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 70: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 71: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 72: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 73: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 74: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 75: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 76: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 77: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 78: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 79: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 80: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 81: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Table 82: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 83: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 84: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 85: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 86: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Table 87: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations)

| Planned Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Day 1, Pre-Dose | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 15 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 29 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 43 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 57 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 119 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 209 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |

| Planned Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Day 394 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Peak GM | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |

Notes: N=Number of subjects in the mITT population.
n=Number of subjects with results available at time point.
GM=Geometric Mean, NE=Not Estimable.
Confidence intervals of the geometric means were calculated with the Student's t distribution on log-transformed data.
[Implementation note: For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."]

- Table 88: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 89: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 90: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 91: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 92: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 93: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 94: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 95: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 96: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 97: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 98: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 99: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 100: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Table 101: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 102: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 103: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 104: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 105: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 106: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 107: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 108: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 109: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 110: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Table 111: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations)

| Planned Time Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|
| Day 1, Pre-Dose | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 15 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 29 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 43 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 57 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 71 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 85 | n | | | |
| | GM | | | |
| | 95% CI | | | |

| Planned Time Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Day 147 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 237 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 422 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Peak GM | n | | | |
| | GM | | | |
| | 95% CI | | | |

Notes: N=Number of subjects in the mITT population. n=Number of subjects with results available at time point.

GM=Geometric Mean, NE=Not Estimable.

Confidence intervals of the geometric means were calculated with the Student's t distribution on log-transformed data.

[Implementation note: For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."]

- Table 112: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 113: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 114: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 115: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 116: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 117: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 118: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 119: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 120: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 121: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 122: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 123: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Table 124: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 125: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 126: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 127: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 128: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 129: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 130: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 131: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 132: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 133: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 134: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 135: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 136: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 137: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Table 138: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 139: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 140: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 141: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 142: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 143: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 144: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 145: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 146: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Table 147: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations)

| Planned Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Day 1, Pre-Dose | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 15 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 29 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 43 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 57 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 119 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Day 209 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |

| Planned Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Day 395 | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |
| Peak GM | n | | | | | | | |
| | GM | | | | | | | |
| | 95% CI | | | | | | | |

Notes: N=Number of subjects in the mITT population.
n=Number of subjects with results available at time point.
GM=Geometric Mean, NE=Not Estimable.
Confidence intervals of the geometric means were calculated with the Student's t distribution on log-transformed data.

[Implementation note: For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."]

- Table 148: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 149: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 150: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 151: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 152: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 153: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 154: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 155: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 156: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 157: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 158: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 159: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 160: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Table 161: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 162: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 163: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 164: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 165: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 166: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 167: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 168: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 169: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 170: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 171: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 172: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 173: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 174: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Table 175: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 176: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 177: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 178: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 179: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 180: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 181: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 182: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Table 183: Percentages of CD4 T Cells Expressing Cytokines with 95% CI – mITT Population, Treatment Arms 2A-B (Three Vaccinations)

| Time Point | Peptide Pool | Cytokine | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| Day 1, Pre- Dose | Beta Mutations | 154 | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | ΙΕΝγ | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/CM | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/EM | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/N | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|
| | | IFNγ or IL-2/TD | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 and 154 | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 or 154 | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 or 154/C | n | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 or 154/E | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 or 154/N | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 or 154/T | n | | | |
| | | | Minimum | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IL-17a | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IL-2 | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IL-4 and 154 | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IL-4 IL-5 IL-13 and 154 | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IL-5 or IL-13 and 154 | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | TNFα | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | Repeat for all peptide pools | s: Beta S, Conserved S1, Conserv | ed S2, Original Match | ed, Original S | | • |

Repeat for all study days

Note: N=Number of Subjects.

n=Number of subjects with results available at time point.

NE=Not Estimable

# Table with Similar Format:

Table 184: Percentages of CD4 T Cells Expressing Cytokines with 95% CI – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

<sup>&</sup>lt;sup>a</sup> Confidence interval calculated based on the Student's t-distribution

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

Table 185: Percentages of CD4 T Cells Expressing Cytokines with 95% CI – mITT Population, Treatment Arms 2C-H (Two Vaccinations)

| Time<br>Point | Peptide Pool | Cytokine | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| Day 1, | Beta Mutations | 154 | n | | | | | | | |
| Pre-<br>Dose | | | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ | n | | | | | | | |
| | | | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ or IL-2 | n | | | | | | | |
| | | | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |

| Time<br>Point | Peptide Pool | Cytokine | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ or IL-<br>2/CM | n | | | | | | | |
| | | 2/CM | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ or IL-<br>2/EM | n | | | | | | | |
| | | 2/EM | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ or IL-<br>2/N | n | | | | | | | |
| | | 2/11 | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |

| Time<br>Point | Peptide Pool | Cytokine | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| | | IFNγ or IL-<br>2/TD | n | | | | | | | |
| | | 2/TD | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ or IL-2<br>and 154 | n | | | | | | | |
| | | and 154 | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ or IL-2 | n | | | | | | | |
| | | or 154 | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | | n | | | | | | | |

| Time<br>Point | Peptide Pool | Cytokine | Statistic | Arm 2C<br>(N=X) | Arm 2D | Arm 2E | Arm 2F | Arm 2G | Arm 2H<br>(N=X) | 23 May 202 All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | (N=A) | (N=X) | (N=X) | (N=X) | (N=X) | (N=A) | |
| | | IFNγ or IL-2<br>or 154/CM | Minimum | | | | | | | |
| | | or 154/CM | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ or IL-2 | n | | | | | | | |
| | | or 154/EM | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ or IL-2<br>or 154/N | n | | | | | | | |
| | | 01 134/11 | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ or IL-2<br>or 154/TD | n | | | | | | | |
| | | 01 157/11 | Minimum | | | | | | | |

| Time<br>Point | Peptide Pool | Cytokine | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IL-17a | n | | | | | | | |
| | | | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IL-2 | n | | | | | | | |
| | | | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IL-4 and 154 | n | | | | | | | |
| | | | Minimum | | | | | | | |
| | | | Median | | | | | | | |

| Time<br>Point | Peptide Pool | Cytokine | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IL-4 IL-5 IL-<br>13 and 154 | n | | | | | | | |
| | | 13 and 134 | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IL-5 or IL-13<br>and 154 | n | | | | | | | |
| | | anu 154 | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | TNFα | n | | | | | | | |
| | | | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |

| Time<br>Point | Peptide Pool | Cytokine | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | Repeat for all peptide pools: Beta S, Conserved S1, Conserved S2, Original Matched, Original S | | | | | | | | | |

Repeat for all Study Days

Note: N=Number of Subjects.

n=Number of subjects with results available at time point.

NE=Not Estimable

<sup>a</sup> Confidence interval calculated based on the Student's t-distribution

# Table with Similar Format:

Table 186: Percentages of CD4 T Cells Expressing Cytokines with 95% CI – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

Table 187: Percentages of CD8 T Cells Expressing Cytokines with 95% CI – mITT Population, Treatment Arms 2A-B (Three Vaccinations)

| Time Point | Peptide Pool | Cytokine | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| Day 1, Pre- Dose | Beta Mutations | IFNγ or IL-2 | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2CM | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2EM | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | IFNγ or IL-2/N | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/TD | n | | | |
| | | | Minimum | | | |
| | | | Median | | | |
| | | | Maximum | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | Repeat for all peptide pools | s: Beta S, Conserved S1, Cons | erved S2, Original Matchea | l, Original S | • | • |

Repeat for all study days

Note: N=Number of Subjects. n=Number of subjects with results available at time point.

NE=Not Estimable

<sup>a</sup> Confidence interval calculated based on the Student's t-distribution

<sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

Table 188: Percentages of CD8 T Cells Expressing Cytokines with 95% CI – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Table 189: Percentages of CD8 T Cells Expressing Cytokines with 95% CI – mITT Population, Treatment Arms 2C-H (Two Vaccinations)

| Time Point | Peptide Pool | Cytokine | Statistic | Arm 2C | Arm 2D | Arm 2E | Arm 2F | Arm 2G | Arm 2H | All Subjects |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Tom | repelue 1 oor | Cytomic | Sucisie | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| Day 1, Pre- Dose | Beta Mutations | IFNγ or IL-2 | n | | | | | | | |
| | | | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response<br>Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ or IL-2CM | n | | | | | | | |
| | | | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response<br>Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ or IL-2EM | n | | | | | | | |
| | | | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Response<br>Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ or IL-2/N | n | | | | | | | |
| | | | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response<br>Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | | IFNγ or IL-2/TD | n | | | | | | | |
| | | | Minimum | | | | | | | |
| | | | Median | | | | | | | |
| | | | Maximum | | | | | | | |
| | | | Mean | | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | | |
| | | | Response<br>Rate | | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | | |
| | Repeat for all pep | otide pools: Beta S, Cor | iserved S1, Cons | erved S2, Original | Matched, Origina | al S | | 1 | | • |

Repeat for all study days

Note: N=Number of Subjects. n=Number of subjects with results available at time point.

NE=Not Estimable

<sup>a</sup> Confidence interval calculated based on the Student's t-distribution

<sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

Table 190: Percentages of CD8 T Cells Expressing Cytokines with 95% CI – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Table 191: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)

| Planned Time Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Day 15 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 29 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 43 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 57 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 71 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 85 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 147 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |

| Planned Time Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Day 237 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 422 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |

Notes: N=Number of subjects in the mITT population. n=Number of subjects with results available at time point. GMFR=Geometric Mean Fold Rise, NE=Not Estimable.

<sup>&</sup>lt;sup>a</sup> Confidence interval calculated based on the Student's t-distribution

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

- [Implementation notes: For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population." For all AUC tables, add footnote reading: "AUC results reported as 0 were imputed to the lowest non-zero reported value for the purposes of fold-rise calculations."]
- Table 192: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 193: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–Wa-1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 194: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–Wa-1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 195: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 196: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 197: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 198: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 199: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Table 200: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 201: Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 202: Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 203: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 204: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 205: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 206: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 207: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.617.2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 208: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.617.2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 209: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-P.1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 210: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 211: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.7 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 212: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.7 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 213: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 214: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Table 215: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations)

| Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Day 15 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 29 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 43 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 57 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 119 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 209 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |

| Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 394 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |

Notes: N=Number of subjects in the mITT population. n=Number of subjects with results available at time point. GMFR=Geometric Mean Fold Rise, NE=Not Estimable.

<sup>&</sup>lt;sup>a</sup> Confidence interval calculated based on the Student's t-distribution

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

### Tables with Similar Format:

- [Implementation notes: For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population." For all AUC tables, add footnote reading: "AUC results reported as 0 were imputed to the lowest non-zero reported value for the purposes of fold-rise calculations."]
- Table 216: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 217: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-Wa-1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 218: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-Wa-1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 219: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 220: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 221: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 222: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 223: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Table 224: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 225: Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 226: Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 227: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 228: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 229: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 230: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 231: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.617.2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 232: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.617.2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 233: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-P.1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Table 234: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 235: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.7 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 236: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.7 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 237: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 238: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Table 239: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

| Planned Time Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Day 15 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 29 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 43 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 57 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 71 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 85 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 147 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 237 | n | | | |

| Planned Time Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 422 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |

n=Number of subjects with results available at time point.

GMFR=Geometric Mean Fold Rise, NE=Not Estimable.

#### Tables with Similar Format:

## Implementation notes:

For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

- Table 240: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 241: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 242: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 243: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 244: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 245: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)

<sup>&</sup>lt;sup>a</sup> Confidence interval calculated based on the Student's t-distribution

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

- Table 246: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 247: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 248: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 249: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 250: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 251: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 252: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 253: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 254: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 255: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 256: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 257: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 258: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 259: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Table 260: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 261: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 262: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Table 263: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

| Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Day 15 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 29 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 43 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 57 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 119 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 209 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |

| Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Day 394 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |

n=Number of subjects with results available at time point.

GMFR=Geometric Mean Fold Rise, NE=Not Estimable.

### Tables with Similar Format:

# Implementation notes:

For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

- Table 264: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 265: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 266: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 267: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 268: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

<sup>&</sup>lt;sup>a</sup> Confidence interval calculated based on the Student's t-distribution

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

- Table 269: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 270: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 271: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 272: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 273: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 274: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 275: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 276: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 277: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 278: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 279: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 280: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 281: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Table 282: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 283: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 284: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 285: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 286: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Table 287: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations)

| Planned Time Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Day 15 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 29 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 43 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 57 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 71 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 85 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 147 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 237 | n | | | |

| Planned Time Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |
| Day 422 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | |

n=Number of subjects with results available at time point.

GMFR=Geometric Mean Fold Rise, NE=Not Estimable.

#### Tables with Similar Format:

[Implementation notes: For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."]

- Table 288: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 289: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 290: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 291: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 292: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 293: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 294: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

<sup>&</sup>lt;sup>a</sup> Confidence interval calculated based on the Student's t-distribution

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

- Table 295: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 296: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 297: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 298: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 299: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 300: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 301: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 302: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 303: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 304: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 305: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 306: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Table 307: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 308: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 309: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 310: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 311: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 312: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 313: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 314: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 315: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 316: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Table 317: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 318: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 319: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 320: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 321: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 322: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Table 323: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations)

| Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Day 15 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 29 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 43 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 57 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 119 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |
| Day 209 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |

| Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Day 394 | n | | | | | | | |
| | GMFR (95% CI) <sup>a</sup> | | | | | | | |
| | Seropositive - % (95% CI) <sup>b</sup> | | | | | | | |

n=Number of subjects with results available at time point.

GMFR=Geometric Mean Fold Rise, NE=Not Estimable.

#### Tables with Similar Format:

## Implementation notes:

For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

- Table 324: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 325: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 326: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 327: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 328: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 329: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 330: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals

<sup>&</sup>lt;sup>a</sup> Confidence interval calculated based on the Student's t-distribution

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

- by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 331: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 332: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 333: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 334: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 335: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 336: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 337: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 338: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 339: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 340: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 341: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Table 342: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 343: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 344: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 345: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 346: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 347: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 348: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 349: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 350: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 351: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 352: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 353: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95%

- Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 354: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 355: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 356: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 357: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 358: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Fold Rise and Seropositivity Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Table 359: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2A-B (Three Vaccinations)

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| B.1.351 | Day 1, Pre-Dose | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 43 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 57 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 71 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 85 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 147 | n | | | |

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 237 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 422 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| B.1.617.2 | Day 1, Pre-Dose | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 43 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 57 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 71 | n | | | |

| Variant | Planned Time | Statistic | Arm 2A | Arm 2B | 23 May 20 All Subjects |
|---|---|---|---|---|---|
| | Point | | (N=X) | (N=X) | (N=X) |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 85 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 147 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 237 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 422 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| P.1 | Day 1, Pre- Dose | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 43 | n | | | |

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 57 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 71 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 85 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 147 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 237 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 422 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| B.1.1.7 | Day 1, Pre-Dose | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 43 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 57 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 71 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 85 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 147 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 237 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 422 | n | | | |

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| B.1.1.529 | Day 1, Pre-Dose | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 43 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 57 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 71 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 85 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 147 | n | | | |

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 237 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 422 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |

Notes: N=Number of subjects in the mITT population. n=Number of subjects with results available at time point.

GMR=Geometric Mean Ratio, NE=Not Estimable.

Geometric Mean Ratio was calculated by taking the ratio of the result for each variant divided by the result of the D614G variant for each subject and calculating the geometric mean.

Confidence interval calculated based on the Student's t-distribution

## Tables with Similar Format:

- Table 360: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 361: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 362: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Table 363: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2C-H (Two Vaccinations)

| Variant | Planned<br>Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| B.1.351 | Day 1, | n | | | | | | | |
| | Pre-Dose | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 15 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 29 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 43 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 57 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 119 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 209 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |

| Variant | Planned<br>Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Day 394 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| B.1.617.2 | Day 1, | n | | | | | | | |
| | Pre-Dose | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 15 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 29 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 43 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 57 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 119 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 209 | n | | | | | | | |
| | | GMR | | | | | | | |

| Variant | Planned<br>Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | 95% CI | | | | | | | |
| | Day 394 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| P.1 | Day 1,<br>Pre- Dose | n | | | | | | | |
| | Pre- Dose | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 15 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 29 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 43 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 57 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 119 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 209 | n | | | | | | | |

| Variant | Planned<br>Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 394 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| B.1.1.7 | Day 1, | n | | | | | | | |
| | Pre-Dose | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 15 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 29 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 43 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 57 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day119 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| Variant | Planned<br>Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Day 209 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 394 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| B.1.1.529 | Day 1, | n | | | | | | | |
| | Pre-Dose | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 15 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 29 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 43 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 57 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 119 | n | | | | | | | |
| | | GMR | | | | | | | |

| Variant | Planned<br>Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | 95% CI | | | | | | | |
| | Day 209 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 394 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |

Notes: N=Number of subjects in the mITT population. n=Number of subjects with results available at time point.

GMR=Geometric Mean Ratio, NE=Not Estimable.

Geometric Mean Ratio was calculated by taking the ratio of the result for each variant divided by the result of the D614G variant for each subject and calculating the geometric mean.

Confidence interval calculated based on the Student's t-distribution

- Table 364: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 365: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 366: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Table 367: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2A-B (Three Vaccinations)

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| B.1.351 | Day 1, Pre-Dose | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 43 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 57 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 71 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 85 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 147 | n | | | |

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 237 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 422 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| B.1.617.2 | Day 1, Pre-Dose | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 43 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 57 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 71 | n | | | |

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 85 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 147 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 237 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 422 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| P.1 | Day 1, Pre-Dose | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 43 | n | | | |

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 57 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 71 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 85 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 147 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 237 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 422 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| B.1.1.7 | Day 1, Pre-Dose | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 43 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 57 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 71 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 85 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 147 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 237 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 422 | n | | | |

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| B.1.1.529 | Day 1, Pre-Dose | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 43 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 57 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 71 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 85 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 147 | n | | | |

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 237 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 422 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |

Notes: N=Number of subjects in the mITT population. n=Number of subjects with results available at time point.

GMR=Geometric Mean Ratio, NE=Not Estimable.

Geometric Mean Ratio was calculated by taking the ratio of the result for each variant divided by the result of the D614G variant for each subject and calculating the geometric mean.

Confidence interval calculated based on the Student's t-distribution

- Table 368: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 369: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 370: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Table 371: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2A-B (Three Vaccinations)

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| B.1.351 | Day 1, Pre-Dose | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 43 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 57 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 71 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 85 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 147 | n | | | |

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 237 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 422 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| B.1.617.2 | Day 1, Pre-Dose | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 43 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 57 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 71 | n | | | |

| Variant | Planned Time<br>Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 85 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 147 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 237 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 422 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |

Notes: N=Number of subjects in the mITT population. n=Number of subjects with results available at time point. GMR=Geometric Mean Ratio, NE=Not Estimable.

Geometric Mean Ratio was calculated by taking the ratio of the result for each variant divided by the result of the D614G variant for each subject and calculating the geometric mean.

Confidence interval calculated based on the Student's t-distribution

- Table 372: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 373: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Table 374: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Table 375: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2C-H (Two Vaccinations)

| Variant | Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| B.1.351 | Day 1, Pre- | n | | | | | | | |
| | Dose | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 15 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 29 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 43 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 57 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 119 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 209 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | <b>Day 394</b> | n | | | | | | | |

| Variant | Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| B.1.617.2 | Day 1, Pre- | n | | | | | | | |
| | Dose | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 15 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 29 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 43 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 57 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 119 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 209 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 394 | n | | | | | | | |

| Variant | Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| P.1 | Day 1, Pre- | n | | | | | | | |
| | Dose | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 15 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 29 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 43 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 57 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 119 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 209 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 394 | n | | | | | | | |

| Variant | Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| B.1.1.7 | Day 1, Pre- | n | | | | | | | |
| | Dose | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 15 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 29 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 43 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 57 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 119 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 209 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 394 | n | | | | | | | |

| Variant | Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| B.1.1.529 | Day 1, Pre- | n | | | | | | | |
| | Dose | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 15 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 29 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 43 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 57 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 119 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 209 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 394 | n | | | | | | | |

| Variant | Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |

Notes: N=Number of subjects in the mITT population.

n=Number of subjects with results available at time point.

GMR=Geometric Mean Ratio, NE=Not Estimable.

Geometric Mean Ratio was calculated by taking the ratio of the result for each variant divided by the result of the D614G variant for each subject and calculating the geometric mean.

Confidence interval calculated based on the Student's t-distribution

- Table 376: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 377: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 378: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Table 379: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population, Treatment Arms 2C-H (Two Vaccinations)

| Variant | Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| B.1.351 | Day 1, Pre- | n | | | | | | | |
| | Dose | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 15 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 29 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 43 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 57 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 119 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 209 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | <b>Day 394</b> | n | | | | | | | |

| Variant | Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| B.1.1.529 | Day 1, Pre- | n | | | | | | | |
| | Dose | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 15 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 29 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 43 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 57 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 119 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 209 | n | | | | | | | |
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 394 | n | | | | | | | |

| Variant | Planned<br>Time Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | GMR | | | | | | | |
| | | 95% CI | | | | | | | |

Notes: N=Number of subjects in the mITT population.

n=Number of subjects with results available at time point.

GMR=Geometric Mean Ratio, NE=Not Estimable.

Geometric Mean Ratio was calculated by taking the ratio of the result for each variant divided by the result of the D614G variant for each subject and calculating the geometric mean.

Confidence interval calculated based on the Student's t-distribution

- Table 380: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 381: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Table 382: Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Table 383: Summary of N-Antibody Expression and Self-Reported Infection Status by Time Point and Treatment Group – mITT Population, Treatment Arms 2A-B (Three Vaccinations)

| Planned Time Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|
| Day 1, Pre-Dose | n | | , , | |
| | % Positive | | | |
| | 95% CI | | | |
| | % Reported Infection | | | |
| | 95% CI | | | |
| Day 15 | n | | | |
| | % Positive | | | |
| | 95% CI | | | |
| | % Reported Infection | | | |
| | 95% CI | | | |
| Day 29 | n | | | |
| | % Positive | | | |
| | 95% CI | | | |
| | % Reported Infection | | | |
| | 95% CI | | | |
| Day 43 | n | | | |
| | % Positive | | | |
| | 95% CI | | | |
| | % Reported Infection | | | |
| | 95% CI | | | |
| Day 57 | n | | | |
| | % Positive | | | |

| Planned Time Point | Statistic | Arm 2A | Arm 2B | 23 May 2023<br>All Subjects |
|---|---|---|---|---|
| | | (N=X) | (N=X) | All Subjects<br>(N=X) |
| | 95% CI | (5.4.55) | (2.1.25) | |
| | % Reported Infection | | | |
| | 95% CI | | | |
| Day 71 | n | | | |
| | % Positive | | | |
| | 95% CI | | | |
| | % Reported Infection | | | |
| | 95% CI | | | |
| Day 85 | n | | | |
| | % Positive | | | |
| | 95% CI | | | |
| | % Reported Infection | | | |
| | 95% CI | | | |
| Day 147 | n | | | |
| | % Positive | | | |
| | 95% CI | | | |
| | % Reported Infection | | | |
| | 95% CI | | | |
| Day 237 | n | | | |
| | % Positive | | | |
| | 95% CI | | | |
| | % Reported Infection | | | |
| | 95% CI | | | |
| Day 422 | n | | | |

| Planned Time Point | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| | % Positive | , | | |
| | 95% CI | | | |
| | % Reported Infection | | | |
| | 95% CI | | | |
| Any Time Point | n | | | |
| | % Positive | | | |
| | 95% CI | | | |
| | % Reported Infection | | | |
| | 95% CI | | | |

Notes: n=number of subjects with results available at time point.

Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

### Table with Similar Format:

Table 384: Summary of N-Antibody Expression and Self-Reported Infection Status by Time Point and Treatment Group – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Table 385: Summary of N-Antibody Expression and Self-Reported Infection Status by Time Point and Treatment Group – mITT Population, Treatment Arms 2C-H (Two Vaccinations)

| Planned Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Day 1, Pre-Dose | n | | | | | | | |
| | % Positive | | | | | | | |
| | 95% CI | | | | | | | |
| | % Reported<br>Infection | | | | | | | |
| | 95% CI | | | | | | | |
| Day 15 | n | | | | | | | |
| | % Positive | | | | | | | |
| | 95% CI | | | | | | | |
| | % Reported<br>Infection<br>95% CI | | | | | | | |
| Day 20 | | | | | | | | |
| Day 29 | n | | | | | | | |
| | % Positive | | | | | | | |
| | 95% CI | | | | | | | |
| | % Reported<br>Infection | | | | | | | |
| | 95% CI | | | | | | | |
| Day 43 | n | | | | | | | |
| | % Positive | | | | | | | |
| | 95% CI | | | | | | | |
| | % Reported<br>Infection | | | | | | | |
| | 95% CI | | | | | | | |
| Day 57 | n | | | | | | | |

| Planned Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | 23 May 202 All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|
| | % Positive | , , | , | , | , , | , , | , , | |
| | 95% CI | | | | | | | |
| | % Reported<br>Infection<br>95% CI | | | | | | | |
| D 110 | | | | | | | | |
| Day 119 | n | | | | | | | |
| | % Positive | | | | | | | |
| | 95% CI | | | | | | | |
| | % Reported<br>Infection<br>95% CI | | | | | | | |
| Day 200 | | | | | | | | |
| Day 209 | n | | | | | | | |
| | % Positive | | | | | | | |
| | 95% CI | | | | | | | |
| | % Reported<br>Infection | | | | | | | |
| | 95% CI | | | | | | | |
| Day 394 | n | | | | | | | |
| | % Positive | | | | | | | |
| | 95% CI | | | | | | | |
| | % Reported<br>Infection | | | | | | | |
| | 95% CI | | | | | | | |
| <b>Any Time Point</b> | n | | | | | | | |
| | % Positive | | | | | | | |
| | 95% CI | | | | | | | |

| Planned Time<br>Point | Statistic | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| | % Reported<br>Infection | | | | | | | |
| | 95% CI | | | | | | | |

Notes: n=number of subjects with results available at time point.

Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

### Table with Similar Format:

Table 386: Summary of N-Antibody Expression and Self-Reported Infection Status by Time Point and Treatment Group – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

# 14.3 Safety Data

## 14.3.1 Displays of Adverse Events

 Table 387:
 Overall Summary of Adverse Events by Treatment Group - All Subjects

| Subjects <sup>a</sup> with | | | n 2A<br>=X) | Arm<br>(N= | | | n 2C<br>=X) | | n 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | n 2G<br>=X) | | n 2H<br>=X) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category 1 | Category 2 | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| At least one local solicited adverse event | NA | | | | | | | | | | | | | | | | | | |
| At least one systemic solicited adverse event | NA | | | | | | | | | | | | | | | | | | |
| At least one unsolicited adverse event | NA | | | | | | | | | | | | | | | | | | |
| At least one related unsolicited adverse event | Any Grade | | | | | | | | | | | | | | | | | | |
| | Mild (Grade 1) | | | | | | | | | | | | | | | | | | |
| | Moderate (Grade 2) | | | | | | | | | | | | | | | | | | |
| | Severe (Grade 3) | | | | | | | | | | | | | | | | | | |
| At least one<br>severe (Grade 3)<br>unsolicited<br>adverse event | Any relationship | | | | | | | | | | | | | | | | | | |
| | Related | | | | | | | | | | | | | | | | | | |
| | Unrelated | | | | | | | | | | | | | | | | | | |
| At least one<br>serious adverse<br>event <sup>b</sup> | Any relationship | | | | | | | | | | | | | | | | | | |

| Subjects <sup>a</sup> with | | | 1 2A<br>=X) | Arm<br>(N= | 1 2B<br>=X) | | n 2C<br>=X) | | n 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | n 2G<br>=X) | | 1 2H<br>=X) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category 1 | Category 2 | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Related | | | | | | | | | | | | | | | | | | |
| | Unrelated | | | | | | | | | | | | | | | | | | |
| At least one<br>adverse event<br>leading to early<br>termination <sup>c</sup> | N/A | | | | | | | | | | | | | | | | | | |
| Any Vital Signs<br>Adverse Event | N/A | | | | | | | | | | | | | | | | | | |
| At least one medically attended adverse event | N/A | | | | | | | | | | | | | | | | | | |
| At least one new onset chronic medical condition | N/A | | | | | | | | | | | | | | | | | | |

N = Number of subjects in the Safety Population

<sup>a</sup>Subjects are counted once for each category regardless of the number of events.

<sup>b</sup>A listing of Serious Adverse Events is included in Table 157.

<sup>c</sup>As reported on the Adverse Event eCRF.

Table 388: Serious Adverse Events and Non-Serious Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - All Subjects

| Preferred<br>Term | MedDRA<br>System<br>Organ<br>Class | | | n 2A<br>=X) | | | Arm 2B<br>(N=X) | | rm Z<br>(N=X | | | Arm 2<br>(N=X | | | rm 2<br>(N=X | | | Arm 2<br>(N=X | | | Arm Z<br>(N=X | | | Arm<br>(N=) | | A | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | Events | n | % | Events | n | % I | Events | n | % E | vents | n | % E | vents | n | % E | events | n | % ] | Events | n | % | Events | n | % | Events |
| Serious Adverse | Events | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| All | All | X | х | X | X | х | X | X | х | х | X | х | х | Х | х | х | Х | Х | х | х | х | х | Х | х | X | X | X | Х |
| PT1 | SOC1 | Х | х | Х | Х | х | X | X | х | х | Х | х | х | Х | Х | х | Х | Х | х | Х | х | х | Х | х | Х | Х | X | Х |
| Etc. | Etc. | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Other (Non-serio | us) Adverse I | Even | its | | | | | | | | | | | | | | | | | | | | | | | | | |
| All | All | х | X | X | X | х | X | X | х | х | х | х | x | Х | X | х | Х | X | х | Х | Х | х | х | х | х | Х | X | X |
| PT1 | SOC1 | х | х | х | х | х | X | X | х | х | х | Х | х | Х | х | х | Х | Х | Х | х | х | х | х | х | X | х | X | х |
| Etc | Etc | | | | | | | | | | | | | | | | | | | | | | | | | | | |

N = number of subjects in the Safety Population (number of subjects at risk).

n= number of subjects reporting event.

Events= total frequency of events reported.

## 14.3.1.1 Solicited Adverse Events

Table 389: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group

| | | Arm<br>(N= | 1 2A<br>=X) | | n 2B<br>=X) | | n 2C<br>=X) | | n 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | n 2G<br>=X) | | 1 2H<br>=X) | Sub | All<br>jects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any Symptom | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Any Systemic | None | | | | | | | | | | | | | | | | | | |
| Symptom | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Arthralgia | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Fatigue | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Fever <sup>a</sup> | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |

| | | | n 2A<br>=X) | | n 2B<br>=X) | | n 2C<br>=X) | | n 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | n 2G<br>=X) | Arn<br>(N= | | Sub | All<br>ojects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Feverishness | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Headache | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Myalgia | None | | | | | | | | | | | | | | | | | | |
| Myalgia | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Nausea | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Any Local Symptom | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Erythema/Redness | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |

| | | | n 2A<br>=X) | | n 2B<br>=X) | | n 2C<br>=X) | | n 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | 1 2G<br>=X) | | 1 2H<br>=X) | Sub | All<br>ojects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Erythema/Redness | None | | | | | | | | | | | | | | | | | | |
| Measurement (mm) | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | | | | | | | |
| Induration/Swelling | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | | | | | | | |
| Measurement (mm) | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Pain | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| _ | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |

Severity is the maximum severity reported over all solicited symptoms post dosing for each subject.

N=All subjects receiving vaccination with any solicited event data recorded in the database.
Table 390: Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2A (Three Vaccinations)

| | | | -Dose<br>(=X) | | -Dose<br>=X) | Da<br>(N | ay 1<br>=X) | | ny 2<br>=X) | Da<br>(N: | ıy 3<br>=X) | Da<br>(N | ay 4<br>(=X) | | ny 5<br>=X) | Da<br>(N | ıy 6<br>=X) | Da<br>(N | ay 7<br>=X) | Day<br>(N | 7 8+ 1<br>=X) | A<br>Post- | ny<br>-Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any | None | | | | | | | | | | | | | | | | | | | | | | |
| Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Any<br>Systemic | None | | | | | | | | | | | | | | | | | | | | | | |
| Systemic<br>Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Arthralgia | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Fatigue | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Fever | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Feverishness | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |

| | | Pre- | -Dose<br>(=X) | | -Dose<br>=X) | Da<br>(N | ay 1<br>=X) | Da<br>(Na | ny 2<br>=X) | Da<br>(N: | ny 3<br>=X) | Da<br>(N | ny 4<br>=X) | Da<br>(N: | ny 5<br>=X) | Da<br>(N: | y 6<br>=X) | Da<br>(N | ny 7<br>=X) | Day<br>(N: | 8+ 1<br>=X) | A<br>Post- | ny<br>-Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Headache | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Myalgia | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Nausea | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Any Local | None | | | | | | | | | | | | | | | | | | | | | | |
| Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Erythema/Redness | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | None | | | | | | | | | | | | | | | | | | | | | | |

| | | | Dose =X) | | -Dose<br>=X) | Da<br>(N: | ny 1<br>=X) | Da<br>(N | ay 2<br>=X) | | ny 3<br>=X) | | ay 4<br>=X) | Da<br>(N: | y 5<br>=X) | Da<br>(N | ny 6<br>=X) | Da<br>(N | ay 7<br>=X) | Day<br>(N: | 8+ 1<br>=X) | A<br>Post- | ny<br>-Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Erythema/Redness | Mild | | | | | | | | | | | | | | | | | | | | | | |
| Measurement (mm) | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | | | | | | | | | | | |
| Measurement (mm) | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Pain | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |

Notes: N=Number of subjects in the Safety Population.
Severity is the maximum severity reported post dosing for each subject for each day.

<sup>&</sup>lt;sup>1</sup> Day 8+ includes the maximum severity of each symptom reported on or after Day 8 (includes ongoing symptoms)
<sup>2</sup> Indicates how many subjects had "None", "Mild", "Moderate", or "Severe" as their maximum severity for any day. A subject may be counted in more than one of these categories.

#### Tables with Similar Format:

[Implementation note: For any symptoms or days with missing data, add a "Not Reported" row.]

**Table 391:** Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2A (Three Vaccinations) **Table 392:** Summary of Solicited Events by Days Post Dose 3, Symptom, and Treatment Group – Treatment Arm 2A (Three Vaccinations) **Table 393:** Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2B (Three Vaccinations) **Table 394:** Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2B (Three Vaccinations) **Table 395:** Summary of Solicited Events by Days Post Dose 3, Symptom, and Treatment Group – Treatment Arm 2B (Three Vaccinations) **Table 396:** Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2C (Two Vaccinations) **Table 397:** Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2C (Two Vaccinations) **Table 398:** Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2D (Two Vaccinations) **Table 399:** Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2D (Two Vaccinations) **Table 400:** Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2E (Two Vaccinations) **Table 401:** Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2E (Two Vaccinations) **Table 402:** Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2F (Two Vaccinations) **Table 403:** Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2F (Two Vaccinations) **Table 404:** Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2G (Two Vaccinations) **Table 405:** Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2G (Two Vaccinations) **Table 406:** Summary of Solicited Events by Days Post Dose 1, Symptom, and Treatment Group – Treatment Arm 2H (Two Vaccinations) **Table 407:** Summary of Solicited Events by Days Post Dose 2, Symptom, and Treatment Group – Treatment Arm 2H (Two Vaccinations)

 Table 408:
 Summary of Number of Days of Solicited Symptoms by Treatment Group - All Subjects

| Variable | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| Any Symptom | n | | | | | | | | | |
| | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| Any Systemic | n | | | | | | | | | |
| Symptom | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| Arthralgia | n | | | | | | | | | |
| | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| Fatigue | n | | | | | | | | | |
| | Mean | | | | | | | | | |

| Variable | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| | Standard<br>Deviation<br>Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| Fever | n | | | | | | | | | |
| | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| Feverishness | n | | | | | | | | | |
| | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| Headache | n | | | | | | | | | |
| | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |

| Variable | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| Myalgia | n | | | | | | | | | |
| | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| Nausea | n | | | | | | | | | |
| | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| Any Local | n | | | | | | | | | |
| Symptom | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| Erythema/redness | n | | | | | | | | | |
| | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |

| Variable | Statistic | Arm 2A<br>(N=X) | Arm 2B<br>(N=X) | Arm 2C<br>(N=X) | Arm 2D<br>(N=X) | Arm 2E<br>(N=X) | Arm 2F<br>(N=X) | Arm 2G<br>(N=X) | Arm 2H<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| Induration/swelling | n | | | | | | | | | |
| | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |
| Pain | n | | | | | | | | | |
| | Mean | | | | | | | | | |
| | Standard<br>Deviation | | | | | | | | | |
| | Median | | | | | | | | | |
| | Minimum | | | | | | | | | |
| | Maximum | | | | | | | | | |

Notes: N=Number of subjects in the Safety Population. n=Number of solicited adverse events.

#### 14.3.1.2 Unsolicited Adverse Events

Table 409: All Adverse Events Cross-Classified by MedDRA System Organ Class, Severity, Relationship to Study Treatment, and Treatment Group

| | | | Rela | ationship to | Vaccination |
|---|---|---|---|---|---|
| Treatment Group | MedDRA System Organ Class | Severity | Not Related (n) | Related (n) | Not Yet Determined (n) |
| Arm 2A | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| Arm 2B | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| Arm 2C | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| Arm 2D | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |

| | | | Rela | tionship to | Vaccination |
|---|---|---|---|---|---|
| Treatment Group | MedDRA System Organ Class | Severity | Not Related (n) | Related (n) | Not Yet Determined (n) |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| Arm 2E | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| Arm 2F | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| Arm 2G | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |

| | | | Rela | ationship to | Vaccination |
|---|---|---|---|---|---|
| Treatment Group | MedDRA System Organ Class | Severity | Not Related (n) | Related (n) | Not Yet Determined (n) |
| Arm 2H | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| All Subjects | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |

Notes: N=Number of subjects in the Safety Population. n=Number of events.

Table 410: Summary of All Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship, and Treatment Group

| | | | | | Severity | | Relatio | nship to Study | y Vaccination |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | System Organ Class<br>(SOC) | Preferred Term (PT) | Total<br>Events<br>(n) | Mild (n) | Moderate (n) | Severe (n) | Not<br>Related<br>(n) | Related (n) | Not Yet<br>Determined<br>(n) |
| Arm 2A | Any SOC | Any PT | | | | | | | |
| (N=X) | [SOC 1] | Any PT | | | | | | | |
| | | [PT 1] | | | | | | | |
| | | [Repeat for all reported PT] | | | | | | | |
| | [Repeat for all | Any PT | | | | | | | |
| | reported SOC] | [Repeat for all reported PT] | | | | | | | |
| Arm 2B | Any SOC | Any PT | | | | | | | |
| (N=X) | [Repeat for all | Any PT | | | | | | | |
| | reported SOC] | [Repeat for all reported PT] | | | | | | | |
| all Subjects | Any SOC | Any PT | | | | | | | |
| N=X) | [Repeat for all | Any PT | | | | | | | |
| | reported SOC] | [Repeat for all reported PT] | | | | | | | |

Notes: N=Number of subjects in the Safety Population.

n=Number of events.

Table 411: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Severity, Relationship, and Treatment Group

| | | | <u> </u> | | | | Sev | erity | | | Rel | ationsh<br>Vacci | ip to S<br>nation | tudy |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | ny<br>dence | M | lild | Mod | lerate | Se | vere | | ot<br>ated | Rel | ated |
| Treatment Group | MedDRA System<br>Organ Class | MedDRA Preferred Term | n | % | n | % | n | % | n | % | n | % | n | % |
| Arm 2A | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all | Any PT | | | | | | | | | | | | |
| | reported SOC] | [Repeat for all reported PT] | | | | | | | | | | | | |
| | [Repeat for all | Any PT | | | | | | | | | | | | |
| | reported SOC] | [Repeat for all reported PT] | | | | | | | | | | | | |
| Arm 2B | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all reported | Any PT | | | | | | | | | | | | |
| | SOC] | [Repeat for all reported PT] | | | | | | | | | | | | |
| Arm 2C | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all reported | Any PT | | | | | | | | | | | | |
| | SOC] | [Repeat for all reported PT] | | | | | | | | | | | | |
| Arm 2D | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all reported | Any PT | | | | | | | | | | | | |
| | SOC] | [Repeat for all reported PT] | | | | | | | | | | | | |
| Arm 2E | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all reported SOC] | Any PT | | | | | | | | | | | | |
| | 300] | [Repeat for all reported PT] | | | | | | | | | | | | |

| | | | | | | | Sev | erity | | | Rel | ationsh<br>Vacci | ip to S<br>nation | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | ny<br>dence | M | lild | Mod | erate | Sev | vere | I | lot<br>lated | Rel | ated |
| Treatment Group | MedDRA System<br>Organ Class | MedDRA Preferred Term | n | % | n | % | n | % | n | % | n | % | n | % |
| Arm 2F | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all reported | Any PT | | | | | | | | | | | | |
| | SOC] | [Repeat for all reported PT] | | | | | | | | | | | | |
| Arm 2G | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | - | Any PT | | | | | | | | | | | | |
| | SOC | [Repeat for all reported PT] | | | | | | | | | | | | |
| Arm 2H | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all reported | Any PT | | | | | | | | | | | | |
| | SOC] | [Repeat for all reported PT] | | | | | | | | | | | | |
| | [Repeat for all reported | Any PT | | | | | | | | | | | | |
| | SOC] | [Repeat for all reported PT] | | | | | | | | | | | | |
| All Subjects | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all | Any PT | | | | | | | | | | | | |
| | reported SOC] | [Repeat for all reported PT] | | | | | | | | | | | | |

Note: N=Number of subjects in the Safety Population. n=Number of subjects reporting event with the specified SOC.

This table presents number and percentage of subjects. A subject is only counted once per PT and is summarized according to their highest severity and closest relationship.

# 14.3.2 Listing of Deaths, Other Serious and Significant Adverse Events

## **Table 412:** Listing of Serious Adverse Events

| Adverse<br>Event | No. of Days Post Associated Dose (Duration) | No. of Days<br>Post Dose<br>the Event<br>Became<br>Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | :, Treatment | Group: , AE N | umber: | | | | | | | | |
| | | | | | | T | | | | | |
| Comments: | | | | | | | | | | | |
| Subject ID | :, Treatment | Group: , AE N | umber: | | | | | | | | |
| | T | | | | | | T | | | | |
| G . | | | | | | | | | | | |
| Comments: | | | | | | | | | | | |

## Table 413: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events

| Adverse<br>Event | No. of Days<br>Post<br>Vaccination<br>(Duration) | Severity | Relationship to Vaccination | If Not<br>Related,<br>Alternative<br>Etiology | Action Taken<br>with Study<br>Vaccination | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA®<br>Sytem Organ<br>Class | MedDRA®<br>Preferred<br>Term | Adverse<br>Event |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Grou | ip: , Dose #: :, Sub | oject ID, AE Num | ber: | | | | | | | |
| | | | T | | T | | T | | | |
| Comments: | | | l | | I | | I | | | |
| Treatment Grou | ip: , Dose #: :, Sub | oject ID, AE Num | ber: | | | | | | | |
| Comments: | | | | | | | | | | |

# Table 414: Listing of AESIs, MAAEs, and NOCMCs

| Subject ID | Treatment<br>Group | Event<br>Description | Date of Product Administration <sup>a</sup> | Duration of<br>Event | Date of Onset | MedDRA®<br>Sytem Organ Class | MAAEs | NOCMCs | Relationship <sup>b</sup> | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|

## 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

(not included in SAP, but this is a placeholder for the CSR)

#### 14.3.6 Displays of Vital Signs

Table 415: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Any Assessment – All Subjects, Treatment Arms 2A-B (Three Vaccinations)

| | | Arm<br>(N= | 1 2A<br>=X) | | n 2B<br>=X) | All So<br>(N | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|
| Time Point | Severity | n | % | n | % | n | % |
| Baseline | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Day 15 | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Day 29 | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Day 43 | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Day 57 | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |

| _ | | Arm<br>(N= | | | n 2B<br>=X) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|
| Time Point | Severity | n | % | n | % | n | % |
| <b>Day 71</b> | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Day 85 | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Day 147 | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Day 237 | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Day 422 | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Max Severity Post<br>Baseline | None | | | | | | |
| Baseline | Mild | | | | | | |
| | Moderate | | | | | | |

| | | | m 2A<br>=X) | Arm<br>(N= | | | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|
| Time Point | Severity | n | % | n | % | n | % |
| | Severe | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N = Number of subjects in the Safety Population.

#### Tables with Similar Format:

- Table 416: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Systolic Blood Pressure All Subjects, Treatment Arms 2A-B (Three Vaccinations)
- Table 417: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Diastolic Blood Pressure All Subjects, Treatment Arms 2A-B (Three Vaccinations)
- Table 418: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Pulse Rate All Subjects, Treatment Arms 2A-B (Three Vaccinations)
- Table 419: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Temperature All Subjects, Treatment Arms 2A-B (Three Vaccinations)

Table 420: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Any Assessment – All Subjects, Treatment Arms 2C-H (Two Vaccinations)

| | | Arm<br>(N= | | | n 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | n 2G<br>=X) | | m 2H<br>=X) | All Su<br>(N= | ibjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | None | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | |
| Day 15 | None | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | |
| Day 29 | None | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | |
| Day 43 | None | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | |
| Day 57 | None | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | |

| | | | n 2C<br>=X) | | m 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | n 2G<br>=X) | | n 2H<br>=X) | All Su<br>(N= | ibjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Severity | n | % | n | % | n | 0/0 | n | % | n | % | n | % | n | % |
| Day 119 | None | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | |
| Day 209 | None | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | |
| <b>Day 394</b> | None | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | |
| Max | None | | | | | | | | | | | | | | |
| Severity<br>Post | Mild | | | | | | | | | | | | | | |
| Baseline | Moderate | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N = Number of subjects in the Safety Population.

#### Tables with Similar Format:

- Table 421: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Systolic Blood Pressure All Subjects, Treatment Arms 2C-H (Two Vaccinations)
- Table 422: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Diastolic Blood Pressure All Subjects, Treatment Arms 2C-H (Two Vaccinations)
- Table 423: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Pulse Rate All Subjects, Treatment Arms 2C-H (Two Vaccinations)
- Table 424: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Temperature All Subjects, Treatment Arms 2C-H (Two Vaccinations)

#### 14.4 Summary of Concomitant Medications

Table 425: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group – All Subjects

[Implementation Note: Table below contains example medications.]

| | | | n 2A<br>=X) | | n 2B<br>=X) | | n 2C<br>=X) | | n 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | n 2G<br>=X) | | 1 2H<br>=X) | | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| WHO Drug Code<br>Level 1, Anatomic<br>Group | WHO Drug Code<br>Level 2,<br>Therapeutic Group | n | % | n | % | n | % | n | % | n | % | n | 0/0 | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |
| Alimentary Tract | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |
| And<br>Metabolism | Antidiarrheals,<br>Intestinal<br>Antiinflammatory<br>/Antiinfective<br>Agents | | | | | | | | | | | | | | | | | | |
| | Antiemetics And<br>Antinauseants | | | | | | | | | | | | | | | | | | |
| | Digestives, Incl.<br>Enzymes | | | | | | | | | | | | | | | | | | |
| | Drugs For Acid<br>Related<br>Disorders | | | | | | | | | | | | | | | | | | |
| | Drugs For<br>Constipation | | | | | | | | | | | | | | | | | | |
| | Drugs Used In<br>Diabetes | | | | | | | | | | | | | | | | | | |
| | Mineral<br>Supplements | | | | | | | | | | | | | | | | | | |

| | | | n 2A<br>=X) | | n 2B<br>=X) | | n 2C<br>=X) | | n 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | n 2G<br>=X) | | n 2H<br>=X) | | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| WHO Drug Code<br>Level 1, Anatomic<br>Group | WHO Drug Code<br>Level 2,<br>Therapeutic Group | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Other Alimentary<br>Tract And<br>Metabolism<br>Products | | | | | | | | | | | | | | | | | | |
| | Stomatological<br>Preparations | | | | | | | | | | | | | | | | | | |
| | Vitamins | | | | | | | | | | | | | | | | | | |
| <b>Antiinfectives For</b> | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |
| Systemic Use | Antibacterials For<br>Systemic Use | | | | | | | | | | | | | | | | | | |
| | Antimycotics For<br>Systemic Use | | | | | | | | | | | | | | | | | | |
| | Antivirals For<br>Systemic<br>Use | | | | | | | | | | | | | | | | | | |
| | Vaccines | | | | | | | | | | | | | | | | | | |
| Antineoplastic And | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |
| Immunomodulating Agents | Antineoplastic<br>Agents | | | | | | | | | | | | | | | | | | |
| | Endocrine<br>Therapy | | | | | | | | | | | | | | | | | | |
| Blood And Blood | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |
| Forming Organs | Antianemic<br>Preparations | | | | | | | | | | | | | | | | | | |
| | Antithrombotic<br>Agents | | | | | | | | | | | | | | | | | | |
| | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |

| | | | n 2A<br>=X) | | n 2B<br>=X) | | n 2C<br>=X) | | n 2D<br>=X) | | n 2E<br>=X) | Arn<br>(N= | n 2F<br>=X) | | 1 2G<br>=X) | | n 2H<br>=X) | All Su<br>(N= | bjects |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| WHO Drug Code<br>Level 1, Anatomic<br>Group | WHO Drug Code<br>Level 2,<br>Therapeutic Group | n | % | n | % | n | % | n | % | n | % | n | 0/0 | n | % | n | % | n | 0/0 |
| Cardiovascular<br>System | Agents Acting On<br>The<br>Renin-Angiotensin<br>System | | | | | | | | | | | | | | | | | | |
| | Beta Blocking<br>Agents | | | | | | | | | | | | | | | | | | |
| | Calcium Channel<br>Blockers | | | | | | | | | | | | | | | | | | |
| | Cardiac Therapy | | | | | | | | | | | | | | | | | | |
| | Diuretics | | | | | | | | | | | | | | | | | | |
| | Lipid Modifying<br>Agents | | | | | | | | | | | | | | | | | | |
| | Vasoprotectives | | | | | | | | | | | | | | | | | | |
| Dermatologicals | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |
| | Anti-Acne<br>Preparations | | | | | | | | | | | | | | | | | | |
| | Antibiotics And<br>Chemotherapeutics<br>For<br>Dermatological<br>Use | | | | | | | | | | | | | | | | | | |
| | Antifungals For<br>Dermatological<br>Use | | | | | | | | | | | | | | | | | | |
| | Antipruritics, Incl.<br>Antihistamines,<br>Anesthetics, Etc. | | | | | | | | | | | | | | | | | | |

| | | | n 2A<br>=X) | | m 2B<br>=X) | | n 2C<br>=X) | | n 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | 1 2G<br>=X) | | n 2H<br>=X) | | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| WHO Drug Code<br>Level 1, Anatomic<br>Group | WHO Drug Code<br>Level 2,<br>Therapeutic Group | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | 0/0 |
| | Antiseptics And<br>Disinfectants | | | | | | | | | | | | | | | | | | |
| | Corticosteroids,<br>Dermatological<br>Preparations | | | | | | | | | | | | | | | | | | |
| | Emollients And<br>Protectives | | | | | | | | | | | | | | | | | | |
| | Other<br>Dermatological<br>Preparations | | | | | | | | | | | | | | | | | | |
| | Preparations For<br>Treatment Of<br>Wounds<br>And Ulcers | | | | | | | | | | | | | | | | | | |
| Genito Urinary | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |
| System<br>And Sex Hormones | Gynecological<br>Antiinfectives And<br>Antiseptics | | | | | | | | | | | | | | | | | | |
| | Other<br>Gynecologicals | | | | | | | | | | | | | | | | | | |
| | Sex Hormones And<br>Modulators Of The<br>Genital System | | | | | | | | | | | | | | | | | | |
| | Urologicals | | | | | | | | | | | | | | | | | | |
| Musculo-Skeletal | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |
| System | Antiinflammatory<br>And<br>Antirheumatic<br>Products | | | | | | | | | | | | | | | | | | |

| | | | n 2A<br>=X) | | n 2B<br>=X) | | n 2C<br>=X) | | n 2D<br>=X) | | n 2E<br>=X) | | n 2F<br>=X) | | n 2G<br>=X) | | n 2H<br>=X) | All Su | y 2023<br>ibjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| WHO Drug Code<br>Level 1, Anatomic<br>Group | WHO Drug Code<br>Level 2,<br>Therapeutic Group | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Drugs For<br>Treatment<br>Of Bone Diseases | | | | | | | | | | | | | | | | | | |
| | Muscle Relaxants | | | | | | | | | | | | | | | | | | |
| | Other Drugs For<br>Disorders Of The<br>Musculo-Skeletal<br>System | | | | | | | | | | | | | | | | | | |
| Nervous System | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |
| | Analgesics | | | | | | | | | | | | | | | | | | |
| | Anesthetics | | | | | | | | | | | | | | | | | | |
| | Other Nervous<br>System<br>Drugs | | | | | | | | | | | | | | | | | | |
| | Psychoanaleptics | | | | | | | | | | | | | | | | | | |
| | Psycholeptics | | | | | | | | | | | | | | | | | | |
| Respiratory System | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |
| | Antihistamines For<br>Systemic Use | | | | | | | | | | | | | | | | | | |
| | Cough And Cold<br>Preparations | | | | | | | | | | | | | | | | | | |
| | Drugs For<br>Obstructive<br>Airway Diseases | | | | | | | | | | | | | | | | | | |
| | Nasal Preparations | | | | | | | | | | | | | | | | | | |
| Sensory Organs | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |

| | | Arm 2A Arm 2B (N=X) | | Arm 2C<br>(N=X) | | Arm 2D<br>(N=X) | | Arm 2E<br>(N=X) | | Arm 2F<br>(N=X) | | Arm 2G<br>(N=X) | | Arm 2H<br>(N=X) | | All Subjects<br>(N=X) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| WHO Drug Code<br>Level 1, Anatomic<br>Group | WHO Drug Code<br>Level 2,<br>Therapeutic Group | n | % | n | % | n. | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Ophthalmologicals | | | | | | | | | | | | | | | | | | |
| Systemic Hormonal | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |
| Preparations, Excl.<br>Sex<br>Hormones And<br>Insulins | Corticosteroids<br>For<br>Systemic Use | | | | | | | | | | | | | | | | | | |
| | Thyroid Therapy | | | | | | | | | | | | | | | | | | |
| Various | Any Level 2 Codes | | | | | | | | | | | | | | | | | | |
| | General Nutrients | | | | | | | | | | | | | | | | | | |
| | Unspecified Herbal<br>And Traditional<br>Medicine | | | | | | | | | | | | | | | | | | |

Notes: N=Number of subjects in the Safety Population. n=Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

# APPENDIX 2. FIGURE MOCK-UPS

# LIST OF FIGURES

| Figure 1: | CONSORT Flow Diagram | 331 |
|---|---|---|
| Figure 2: | Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group - S-2P-Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 332 |
| Figure 3: | Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 333 |
| Figure 4: | Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 333 |
| Figure 5: | Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 333 |
| Figure 6: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 333 |
| Figure 7: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 333 |
| Figure 8: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 333 |
| Figure 9: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 333 |
| Figure 10: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 333 |
| Figure 11: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 333 |
| Figure 12: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 333 |

| Figure 13: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 333 |
|---|---|---|
| Figure 14: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 333 |
| Figure 15: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 333 |
| Figure 16: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 334 |
| Figure 17: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 334 |
| Figure 18: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 334 |
| Figure 19: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 334 |
| Figure 20: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 334 |
| Figure 21: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 334 |
| Figure 22: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 334 |
| Figure 23: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 334 |
| Figure 24: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 334 |
| Figure 25: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 334 |

| Figure 26: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 334 |
|---|---|---|
| Figure 27: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 334 |
| Figure 28: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 334 |
| Figure 29: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 335 |
| Figure 30: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 335 |
| Figure 31: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 335 |
| Figure 32: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 335 |
| Figure 33: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 335 |
| Figure 34: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 35: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 36: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 335 |
| Figure 37: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 38: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 39: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 335 |
|---|---|---|
| Figure 40: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 335 |
| Figure 41: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 335 |
| Figure 42: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 336 |
| Figure 43: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 336 |
| Figure 44: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 336 |
| Figure 45: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 336 |
| Figure 46: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 47: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 48: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 49: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 50: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 51: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 52: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 336 |
|---|---|---|
| Figure 53: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 336 |
| Figure 54: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 336 |
| Figure 55: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 337 |
| Figure 56: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 337 |
| Figure 57: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 58: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 59: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 60: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 61: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 62: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 63: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 64: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 65: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 337 |
|---|---|---|
| Figure 66: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 337 |
| Figure 67: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 337 |
| Figure 68: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 338 |
| Figure 69: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 338 |
| Figure 70: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 338 |
| Figure 71: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 72: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 73: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 74: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 75: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 76: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 77: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 78: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 338 |
|---|---|---|
| Figure 79: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 338 |
| Figure 80: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 338 |
| Figure 81: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 339 |
| Figure 82: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 339 |
| Figure 83: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 339 |
| Figure 84: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 339 |
| Figure 85: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 339 |
| Figure 86: | Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group - S-2P—Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 340 |
| Figure 87: | Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 341 |
| Figure 88: | Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 341 |
| Figure 89: | Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 90: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 91: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 341 |
|---|---|---|
| Figure 92: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 341 |
| Figure 93: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 341 |
| Figure 94: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 341 |
| Figure 95: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 341 |
| Figure 96: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 341 |
| Figure 97: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 341 |
| Figure 98: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 341 |
| Figure 99: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 341 |
| Figure 100: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 342 |
| Figure 101: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 342 |
| Figure 102: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 103: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area<br>Under the Curve by Time Point and Treatment Group – S-2P–B.1.617.2, Per<br>Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 104: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 342 |
|---|---|---|
| Figure 105: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 342 |
| Figure 106: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 342 |
| Figure 107: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 342 |
| Figure 108: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 342 |
| Figure 109: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 342 |
| Figure 110: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 342 |
| Figure 111: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 342 |
| Figure 112: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 342 |
| Figure 113: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 343 |
| Figure 114: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 115: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 116: | Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 117: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 343 |
|---|---|
| Figure 118: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 343 |
| Figure 119: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 343 |
| Figure 120: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 343 |
| Figure 121: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 343 |
| Figure 122: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 343 |
| Figure 123: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 343 |
| Figure 124: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 343 |
| Figure 125: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 343 |
| Figure 126: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 344 |
| Figure 127: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 344 |
| Figure 128: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 344 |
| Figure 129: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 130: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
|---|---|
| Figure 131: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay I by Time Point and Treatment Group – B.1.1.529, Per Protocol Populati Treatment Arms 2C-H (Two Vaccinations) | on, |
| Figure 132: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 133: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay I by Time Point and Treatment Group – B.1.1.529, Per Protocol Populati Treatment Arms 2C-H (Two Vaccinations) | on, |
| Figure 134: Reverse Cumulative Distribution of Focus Reduction Neutralization As ID <sub>50</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | • |
| Figure 135: Reverse Cumulative Distribution of Focus Reduction Neutralization As ID <sub>50</sub> by Time Point and Treatment Group – D614G, Per Protocol Popul Treatment Arms 2C-H (Two Vaccinations) | ation, |
| Figure 136: Reverse Cumulative Distribution of Focus Reduction Neutralization As ID <sub>80</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | • |
| Figure 137: Reverse Cumulative Distribution of Focus Reduction Neutralization As ID <sub>80</sub> by Time Point and Treatment Group – D614G, Per Protocol Popul Treatment Arms 2C-H (Two Vaccinations) | ation, |
| Figure 138: Reverse Cumulative Distribution of Focus Reduction Neutralization As ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | • |
| Figure 139: Reverse Cumulative Distribution of Focus Reduction Neutralization As ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | say |
| Figure 140: Reverse Cumulative Distribution of Focus Reduction Neutralization As ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | say |
| Figure 141: Reverse Cumulative Distribution of Focus Reduction Neutralization As ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | say |
| Figure 142: Reverse Cumulative Distribution of Focus Reduction Neutralization As ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population Treatment Arms 2C-H (Two Vaccinations) | ssay<br>n, |

| _ | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 345 |
|---|---|---|
| Figure 144: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 345 |
| | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 345 |
| | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 345 |
| Figure 147: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 345 |
| | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 345 |
| | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 345 |
| Figure 150: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 345 |
| Figure 151: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 345 |
| Figure 152: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 346 |
| Figure 153: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 346 |
| Figure 154: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 156: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 346 |
|---|---|---|
| Figure 157: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 346 |
| Figure 158: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 346 |
| Figure 159: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 346 |
| Figure 160: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 346 |
| Figure 161: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 346 |
| Figure 162: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 346 |
| Figure 163: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 164: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 346 |
| Figure 165: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 166: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 347 |
| Figure 167: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 168: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 169: | Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 347 |
|---|---|---|
| Figure 170: | Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group — S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 348 |
| Figure 171: | Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 172: | Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group - RBD-Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 173: | Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group — RBD—Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 174 | Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 175 | Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 176: | Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 177 | Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 178 | Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 179 | Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 180: | Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 181: | Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 182: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
|---|---|---|
| Figure 183: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 184: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 185: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 186: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 187: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 349 |
| Figure 188: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 189: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 190: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 191: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 192: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 193: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 194: | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 195 | : Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three | |
|---|---|---|
| | Vaccinations) | 350 |
| Figure 196 | : Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 197 | : Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 198 | : Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 199 | : Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 200 | : Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 201 | : Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 202 | : Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 203 | : Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 204 | : Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 205 | : Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 350 |
| Figure 206 | : Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| Figure 207 | : Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| Figure 208 | : Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| Figure 209 | : Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| Figure 210 | : Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |

| | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
|---|---|---|
| Figure 212: | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| _ | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| _ | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| _ | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| _ | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 351 |
| _ | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 225: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
|---|---|
| Figure 226: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 227: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 228: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 229: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 230: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)352 |
| Figure 231: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 232: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)352 |
| Figure 233: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 234: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 235: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 236: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 237: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 238: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) |

| Figure 239: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 352 |
|---|---|---|
| Figure 240: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 352 |
| Figure 241: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 352 |
| Figure 242: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 352 |
| Figure 243: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 352 |
| Figure 244: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 353 |
| Figure 245: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 353 |
| Figure 246: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 353 |
| Figure 247: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 353 |
| Figure 248: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 249: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 250: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 251: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 252: | : Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 353 |
|---|---|---|
| Figure 253: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 353 |
| Figure 254: | : Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group - S-2P-Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 354 |
| Figure 255: | : Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group — S-2P—Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |
| Figure 256: | Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |
| Figure 257: | Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group — RBD—Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |
| Figure 258: | Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |
| Figure 259: | : Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and<br>Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms<br>2C-H (Two Vaccinations) | 355 |
| Figure 260: | : Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and<br>Treatment Group – S-2P– B.1.351, mITT Population, Treatment Arms 2C-H<br>(Two Vaccinations) | 355 |
| Figure 261: | : Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |
| Figure 262: | Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 263: | Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |
| Figure 264: | : Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |
| Figure 265: | : Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |

| | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |
|---|---|---|
| | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |
| | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |
| | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |
| | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |
| | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 355 |
| Figure 272: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 273: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 274: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 275: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 276: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 277: | Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 278: | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 279: | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
|---|---|---|
| Figure 280: | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 281: | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 282: | Pseudovirus Neutralization Assay $ID_{50}$ by Time Point and Treatment Group $-$ B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 283: | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 284: | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 285: | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 286: | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 287: | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 288: | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 289: | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 356 |
| Figure 290: | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 291: | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 292: | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| _ | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 294: | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |

| Figure 295: | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
|---|---|---|
| Figure 296: | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 297: | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 298: | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 299: | Pseudovirus Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 300: | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 301: | Pseudovirus Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 302: | : Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 303: | : Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 304: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 305: | : Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 306: | : Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 307: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 357 |
| Figure 308: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 309: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 8 |
|---|---|---|
| Figure 310: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 8 |
| Figure 311: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 8 |
| Figure 312: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 8 |
| Figure 313: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 8 |
| Figure 314: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)35 | 8 |
| Figure 315: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 8 |
| Figure 316: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)35 | 8 |
| Figure 317: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 8 |
| Figure 318: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 8 |
| Figure 319: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 8 |
| Figure 320: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 8 |
| Figure 321: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 8 |
| Figure 322: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 8 |

| Figure 323: | Focus Reduction Neutralization Assay ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 358 |
|---|---|---|
| Figure 324: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 358 |
| Figure 325: | Focus Reduction Neutralization Assay ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 358 |
| Figure 326: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 358 |
| Figure 327: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 358 |
| Figure 328: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 359 |
| Figure 329: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 359 |
| Figure 330: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 359 |
| Figure 331: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 359 |
| Figure 332: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 359 |
| Figure 333: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 359 |
| Figure 334: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 359 |
| Figure 335: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>50</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 336: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 359 |
|---|---|---|
| Figure 337: | Focus Reduction Neutralization Assay (TMPRS cells) ID <sub>80</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 359 |
| Figure 338: | Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 360 |
| Figure 339: | Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 361 |
| Figure 340: | Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 361 |
| Figure 341: | Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 361 |
| Figure 342: | Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 361 |
| Figure 343: | Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 361 |
| Figure 344: | Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 345: | Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 361 |
| Figure 346: | Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 361 |
| Figure 347: | Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 348: | Geometric Mean Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 349: Geometric Mean Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
|---|---|
| Figure 350: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 361 |
| Figure 351: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 361 |
| Figure 352: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 361 |
| Figure 353: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 362 |
| Figure 354: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 362 |
| Figure 355: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 362 |
| Figure 356: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 362 |
| Figure 357: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 358: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 359: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 360: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 361: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |

| | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 362 |
|---|---|---|
| | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 362 |
| | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 362 |
| | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 363 |
| | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 363 |
| | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 363 |
| | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 363 |
| Figure 369: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 363 |
| | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 363 |
| Figure 371: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 372: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 373: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 374: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 375: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 363 |
|---|---|---|
| Figure 376: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 363 |
| Figure 377: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 363 |
| Figure 378: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 363 |
| Figure 379: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 364 |
| Figure 380: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 364 |
| Figure 381: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 364 |
| Figure 382: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 364 |
| Figure 383: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 384: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 385: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 386: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 387: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 388: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 364 |
|---|---|---|
| Figure 389: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 364 |
| Figure 390: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 364 |
| Figure 391: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 364 |
| Figure 392: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 365 |
| Figure 393: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 365 |
| Figure 394: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 365 |
| Figure 395: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 396: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 365 |
| Figure 397: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 365 |
| Figure 398: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 365 |
| Figure 399: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 400: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 401: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 365 |
|---|---|---|
| Figure 402: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 365 |
| Figure 403: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 365 |
| Figure 404: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 365 |
| Figure 405: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 365 |
| Figure 406: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 366 |
| Figure 407: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 408: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 366 |
| Figure 409: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 366 |
| Figure 410: | Geometric Mean Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 366 |
| Figure 411: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 366 |
| Figure 412: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 413: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 414: Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 366 |
|---|---|
| Figure 415: Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 366 |
| Figure 416: Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 366 |
| Figure 417: Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 366 |
| Figure 418: Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 366 |
| Figure 419: Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 367 |
| Figure 420: Geometric Mean Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 421: Geometric Mean Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 367 |
| Figure 422: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 368 |
| Figure 423: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 369 |
| Figure 424: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 369 |
| Figure 425: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 426: Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Poir | ometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time nt and Treatment Group – S-2P–Wa-1, Per Protocol Population, atment Arms 2C-H (Two Vaccinations) | 369 |
|---|---|---|
| Poir | ometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time nt and Treatment Group – S-2P– B.1.351, mITT Population, Treatment ns 2C-H (Two Vaccinations) | 369 |
| Poir | ometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time nt and Treatment Group – S-2P– B.1.351, Per Protocol Population, atment Arms 2C-H (Two Vaccinations) | 369 |
| Poir | ometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time nt and Treatment Group – RBD– B.1.351, mITT Population, Treatment ns 2C-H (Two Vaccinations) | 369 |
| Poir | ometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time nt and Treatment Group – RBD– B.1.351, Per Protocol Population, atment Arms 2C-H (Two Vaccinations) | 369 |
| by T | ometric Mean Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL<br>Γime Point and Treatment Group – S-2P–Wa-1, mITT Population,<br>atment Arms 2C-H (Two Vaccinations) | 369 |
| by T | ometric Mean Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL<br>Γime Point and Treatment Group – S-2P–Wa-1, Per Protocol Population,<br>atment Arms 2C-H (Two Vaccinations) | 369 |
| Tim | ometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by the Point and Treatment Group – S-2P–Wa-1, mITT Population, atment Arms 2C-H (Two Vaccinations) | 369 |
| Figure 435: Geo | ometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by the Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, atment Arms 2C-H (Two Vaccinations) | 369 |
| Figure 436: Geo | ometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by the Point and Treatment Group – S-2P–B.1.351, mITT Population, | 369 |
| Figure 437: Geo | ometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by the Point and Treatment Group – S-2P–B.1.351, Per Protocol Population, | 370 |
| Figure 438: Geo | ometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by the Point and Treatment Group – S-2P–B.1.617.2, mITT Population, atment Arms 2C-H (Two Vaccinations) | |
| Figure 439: Geo | ometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by the Point and Treatment Group – S-2P–B.1.617.2, Per Protocol oulation, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 440: | Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 370 |
|---|---|---|
| Figure 441: | Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 370 |
| Figure 442: | Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 370 |
| Figure 443: | Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 370 |
| Figure 444: | Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 370 |
| Figure 445: | Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 370 |
| Figure 446: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 447: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 448: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 449: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 450: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 451: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 452: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 453: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 371 |
|---|---|---|
| Figure 454: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 371 |
| Figure 455: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 371 |
| Figure 456: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 371 |
| Figure 457: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 371 |
| Figure 458: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 371 |
| Figure 459: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 371 |
| Figure 460: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 461: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 462: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 463: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 464: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 465: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 466: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 372 |
|---|---|---|
| Figure 467: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 372 |
| Figure 468: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 372 |
| Figure 469: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 372 |
| Figure 470: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 372 |
| Figure 471: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 372 |
| Figure 472: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 473: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 474: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 475: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 476: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 477: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 478: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 373 |
|---|---|---|
| | Geometric Mean Focus Reduction Neutralization Test $ID_{80}$ Titers by Time Point and Treatment Group $-$ B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations). | 373 |
| | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 373 |
| | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 373 |
| | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 373 |
| | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 373 |
| Figure 485: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 373 |
| | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 373 |
| Figure 488: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| _ | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| _ | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| _ | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 492: Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 374 |
|---|---|
| Figure 493: Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 374 |
| Figure 494: Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 374 |
| Figure 495: Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 374 |
| Figure 496: Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 374 |
| Figure 497: Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 374 |
| Figure 498: Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 499: Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 500: Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 501: Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 502: Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 503: Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 504: Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 505: Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 375 |
|---|---|
| Figure 506: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 376 |
| Figure 507: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 377 |
| Figure 508: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 377 |
| Figure 509: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 377 |
| Figure 510: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 377 |
| Figure 511: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 377 |
| Figure 512: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 513: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 514: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 515: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 516: Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 517: Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 518: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 377 |
|---|---|
| Figure 519: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 520: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 378 |
| Figure 521: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 378 |
| Figure 522: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 378 |
| Figure 523: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 378 |
| Figure 524: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 378 |
| Figure 525: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 526: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 527: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 528: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 529: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 530: Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 531: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 378 |
|---|---|---|
| Figure 532: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 378 |
| Figure 533: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 379 |
| Figure 534: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 379 |
| Figure 535: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 379 |
| Figure 536: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 379 |
| Figure 537: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 379 |
| Figure 538: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 539: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 540: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 379 |
| Figure 541: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 542: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 543: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 544: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 379 |
|---|---|---|
| Figure 545: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 379 |
| Figure 546: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 379 |
| Figure 547: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 380 |
| Figure 548: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 380 |
| Figure 549: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 380 |
| Figure 550: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 380 |
| Figure 551: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 380 |
| Figure 552: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 380 |
| Figure 553: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 554: | Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 555: | Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 556: | Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 557: | : Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 380 |
|---|---|---|
| Figure 558: | : Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 380 |
| Figure 559: | : Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 380 |
| Figure 560: | : Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 381 |
| Figure 561: | : Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 381 |
| Figure 562: | : Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 381 |
| Figure 563: | : Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 381 |
| Figure 564: | : Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 381 |
| Figure 565: | : Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 381 |
| Figure 566: | : Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 381 |
| Figure 567: | : Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 568: | : Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 569: | : Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 570: Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 381 |
|---|---|
| Figure 571: Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 381 |
| Figure 572: Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 381 |
| Figure 573: Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 381 |
| Figure 574: Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 382 |
| Figure 575: Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 382 |
| Figure 576: Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 577: Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 578: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 579: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 580: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 581: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 582: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 583: Distribution of Focus Reduction Neutralization Test (TMPRS cells) II Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
|---|---|
| Figure 584: Distribution of Focus Reduction Neutralization Test (TMPRS cells) II Titers by Time Point and Treatment Group – B.1.351, mITT Populatio Treatment Arms 2A-B (Three Vaccinations) | n, |
| Figure 585: Distribution of Focus Reduction Neutralization Test (TMPRS cells) II Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 586: Distribution of Focus Reduction Neutralization Test (TMPRS cells) II Titers by Time Point and Treatment Group – B.1.1.529, mITT Populat Treatment Arms 2A-B (Three Vaccinations) | ion, |
| Figure 587: Distribution of Focus Reduction Neutralization Test (TMPRS cells) II Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 588: Distribution of Focus Reduction Neutralization Test (TMPRS cells) II Titers by Time Point and Treatment Group – B.1.1.529, mITT Populat Treatment Arms 2A-B (Three Vaccinations) | ion, |
| Figure 589: Distribution of Focus Reduction Neutralization Test (TMPRS cells) II Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 590: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 20 (Two Vaccinations) | and<br>C-H |
| Figure 591: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment A 2C-H (Two Vaccinations) | and<br>rms |
| Figure 592: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point Treatment Group – RBD–Wa-1, mITT Population, Treatment Arms 20 (Two Vaccinations) | and<br>C-H |
| Figure 593: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point Treatment Group – RBD–Wa-1, Per Protocol Population, Treatment A 2C-H (Two Vaccinations) | and<br>Arms |
| Figure 594: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by 7 Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | Γime<br>nt |
| Figure 595: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by 7 Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | Γime |

| _ | Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 385 |
|---|---|---|
| _ | Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – S-2P–B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 385 |
| _ | Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 385 |
| _ | Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 385 |
| Figure 600: | Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 385 |
| Figure 601: | Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 385 |
| Figure 602: | Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 385 |
| Figure 603: | Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 385 |
| Figure 604: | Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 386 |
| Figure 605: | Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 386 |
| Figure 606: | Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 607: | Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 608: | Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Time | ribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by e Point and Treatment Group – S-2P– P.1, Per Protocol Population, tment Arms 2C-H (Two Vaccinations) | .386 |
|---|---|---|
| Time | ribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by e Point and Treatment Group – S-2P– B.1.1.7, mITT Population, tment Arms 2C-H (Two Vaccinations) | .386 |
| Time | ribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by e Point and Treatment Group – S-2P– B.1.1.7, Per Protocol Population, tment Arms 2C-H (Two Vaccinations) | .386 |
| Time | ribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by e Point and Treatment Group – S-2P– B.1.1.529, mITT Population, tment Arms 2C-H (Two Vaccinations) | .386 |
| Time | ribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by e Point and Treatment Group – S-2P– B.1.1.529, Per Protocol lation, Treatment Arms 2C-H (Two Vaccinations) | .386 |
| and ' | ribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point Treatment Group – D614G, mITT Population, Treatment Arms 2C-H o Vaccinations) | .386 |
| and ' | ribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point Treatment Group – D614G, Per Protocol Population, Treatment Arms H (Two Vaccinations) | .386 |
| Figure 616: Distant | ribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point Treatment Group – D614G, mITT Population, Treatment Arms 2C-H | .386 |
| Figure 617: Distrand | ribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point Treatment Group – D614G, Per Protocol Population, Treatment Arms H (Two Vaccinations) | .387 |
| Figure 618: Distand | ribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H | .387 |
| Figure 619: Distand | ribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point Treatment Group – B.1.351, Per Protocol Population, Treatment Arms | .387 |
| Figure 620: Distant | ribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H | .387 |
| Figure 621: Distrand | ribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point Treatment Group – B.1.351, Per Protocol Population, Treatment Arms H (Two Vaccinations) | |

| Figure 622: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 387 |
|---|---|---|
| Figure 623: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 387 |
| Figure 624: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 387 |
| Figure 625: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 387 |
| Figure 626: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 387 |
| Figure 627: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 387 |
| Figure 628: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 387 |
| Figure 629: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 387 |
| Figure 630: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 387 |
| Figure 631: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 388 |
| Figure 632: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 388 |
| Figure 633: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 634: | Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 635: Distribution of Pseudovirus Neutralization Assay IDs and Treatment Group – B.1.1.529, Per Protocol Popu 2C-H (Two Vaccinations) | lation, Treatment Arms |
|---|---|
| Figure 636: Distribution of Pseudovirus Neutralization Assay IDs and Treatment Group – B.1.1.529, mITT Population, (Two Vaccinations) | Treatment Arms 2C-H |
| Figure 637: Distribution of Pseudovirus Neutralization Assay ID8 and Treatment Group – B.1.1.529, Per Protocol Popu 2C-H (Two Vaccinations) | lation, Treatment Arms |
| Figure 638: Distribution of Focus Reduction Neutralization Test Point and Treatment Group – D614G, mITT Populati 2C-H (Two Vaccinations) | on, Treatment Arms |
| Figure 639: Distribution of Focus Reduction Neutralization Test Point and Treatment Group – D614G, Per Protocol Po Arms 2C-H (Two Vaccinations) | opulation, Treatment |
| Figure 640: Distribution of Focus Reduction Neutralization Test Point and Treatment Group – D614G, mITT Populati 2C-H (Two Vaccinations) | ID <sub>80</sub> Titers by Time on, Treatment Arms |
| Figure 641: Distribution of Focus Reduction Neutralization Test Point and Treatment Group – D614G, Per Protocol Po Arms 2C-H (Two Vaccinations) | ID <sub>80</sub> Titers by Time opulation, Treatment |
| Figure 642: Distribution of Focus Reduction Neutralization Test Point and Treatment Group – B.1.351, mITT Population 2C-H (Two Vaccinations) | ID <sub>50</sub> Titers by Time ion, Treatment Arms |
| Figure 643: Distribution of Focus Reduction Neutralization Test Point and Treatment Group – B.1.351, Per Protocol P Arms 2C-H (Two Vaccinations) | ID <sub>50</sub> Titers by Time opulation, Treatment |
| Figure 644: Distribution of Focus Reduction Neutralization Test Point and Treatment Group – B.1.351, mITT Population 2C-H (Two Vaccinations) | ID <sub>80</sub> Titers by Time ion, Treatment Arms |
| Figure 645: Distribution of Focus Reduction Neutralization Test Point and Treatment Group – B.1.351, Per Protocol P Arms 2C-H (Two Vaccinations) | ID <sub>80</sub> Titers by Time opulation, Treatment |
| Figure 646: Distribution of Focus Reduction Neutralization Test Point and Treatment Group – B.1.617.2, mITT Popul 2C-H (Two Vaccinations) | ID <sub>50</sub> Titers by Time ation, Treatment Arms |
| Figure 647: Distribution of Focus Reduction Neutralization Test Point and Treatment Group – B.1.617.2, Per Protocol Arms 2C-H (Two Vaccinations) | ID <sub>50</sub> Titers by Time<br>Population, Treatment |

| | Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 389 |
|---|---|---|
| | Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 389 |
| | Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 389 |
| | Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 389 |
| | Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 389 |
| | Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 389 |
| | Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 389 |
| | Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 389 |
| Figure 656: | Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 657: | Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 658: | Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 659: | Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 660: | Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 661: Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
|---|---|
| Figure 662: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 390 |
| Figure 663: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 390 |
| Figure 664: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 390 |
| Figure 665: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 390 |
| Figure 666: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 390 |
| Figure 667: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 390 |
| Figure 668: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 390 |
| Figure 669: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 670: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 671: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 672: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 673: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 674: Correlation Heatmap, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 392 |
|---|---|
| Figure 675: Correlation Heatmap, D614G – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 393 |
| Figure 676: Correlation Heatmap, B.1.351 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 393 |
| Figure 677: Correlation Heatmap, B.1.351 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 393 |
| Figure 678: Correlation Heatmap, B.1.617.2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 393 |
| Figure 679: Correlation Heatmap, B.1.617.2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 393 |
| Figure 680: Correlation Heatmap, P.1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 393 |
| Figure 681: Correlation Heatmap, P.1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 393 |
| Figure 682: Correlation Heatmap, B.1.1.7 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 393 |
| Figure 683: Correlation Heatmap, B.1.1.7 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 393 |
| Figure 684: Correlation Heatmap, B.1.1.529 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 393 |
| Figure 685: Correlation Heatmap, B.1.1.529 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 393 |
| Figure 686: Correlation Heatmap, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 394 |
| Figure 687: Correlation Heatmap, D614G – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 395 |
| Figure 688: Correlation Heatmap, B.1.351 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 689: Correlation Heatmap, B.1.351 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 690: Correlation Heatmap, B.1.617.2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 691: Correlation Heatmap, B.1.617.2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 692: Correlation Heatmap, P.1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 693: | Correlation Heatmap, P.1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 395 |
|---|---|---|
| Figure 694: | Correlation Heatmap, B.1.1.7 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 395 |
| Figure 695: | Correlation Heatmap, B.1.1.7 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 395 |
| Figure 696: | Correlation Heatmap, B.1.1.529 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 395 |
| Figure 697: | Correlation Heatmap, B.1.1.529 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 395 |
| Figure 698: | Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 396 |
| Figure 699: | Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 397 |
| Figure 700: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 397 |
| Figure 701: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 397 |
| Figure 702: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 397 |
| Figure 703: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 397 |
| Figure 704: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 397 |
| Figure 705: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 397 |
| Figure 706: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 397 |
| Figure 707: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 397 |
| Figure 708: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta<br>Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 397 |
| Figure 709: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta<br>Mutations – Per Protocol Population, Treatment Arms 2A-B (Three<br>Vaccinations) | 397 |
| Figure 710: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 397 |

| Figure 711: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 397 |
|---|---|---|
| Figure 712: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 713: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 714: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 715: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 716: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 717: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 718: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 719: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 720: | Percentages of CD4 T Cells Expressing IFNγ, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 721: | Percentages of CD4 T Cells Expressing IFNγ, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| | Percentages of CD4 T Cells Expressing IL-17, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 723: | Percentages of CD4 T Cells Expressing IL-17, Beta Mutations – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 724: | Percentages of CD4 T Cells Expressing IL-2, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 725: | Percentages of CD4 T Cells Expressing IL-2, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 726: | Percentages of CD4 T Cells Expressing IL-4 and 154, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 398 |
| Figure 727: | Percentages of CD4 T Cells Expressing IL-4 and 154, Beta Mutations – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |

| Figure 728: | : Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |
|---|---|---|
| Figure 729: | : Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta<br>Mutations – Per Protocol Population, Treatment Arms 2A-B (Three<br>Vaccinations) | 399 |
| Figure 730: | : Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta<br>Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |
| Figure 731: | : Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta<br>Mutations – Per Protocol Population, Treatment Arms 2A-B (Three<br>Vaccinations) | 399 |
| Figure 732: | : Percentages of CD4 T Cells Expressing TNFα, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |
| Figure 733: | : Percentages of CD4 T Cells Expressing TNFα, Beta Mutations – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |
| Figure 734: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |
| Figure 735: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |
| Figure 736: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |
| Figure 737: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |
| Figure 738: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |
| Figure 739: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |
| Figure 740: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |
| Figure 741: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta S – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |
| Figure 742: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 399 |
| Figure 743: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta S – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
| Figure 744: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
| Figure 745: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 746: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
|---|---|---|
| Figure 747: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
| Figure 748: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
| Figure 749: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
| Figure 750: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
| Figure 751: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
| Figure 752: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
| Figure 753: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
| Figure 754: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
| Figure 755: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
| Figure 756: | Percentages of CD4 T Cells Expressing IFNγ, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
| Figure 757: | Percentages of CD4 T Cells Expressing IFNγ, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 400 |
| Figure 758: | Percentages of CD4 T Cells Expressing IL-17, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 401 |
| Figure 759: | Percentages of CD4 T Cells Expressing IL-17, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 401 |
| Figure 760: | Percentages of CD4 T Cells Expressing IL-2, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 401 |
| Figure 761: | Percentages of CD4 T Cells Expressing IL-2, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 401 |
| Figure 762: | Percentages of CD4 T Cells Expressing IL-4 and 154, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 401 |
| Figure 763: | Percentages of CD4 T Cells Expressing IL-4 and 154, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 764: | Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 765 | : Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)40 | 01 |
|---|---|---|
| Figure 766s | Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations)40 | 01 |
| Figure 767: | Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 01 |
| Figure 768: | Percentages of CD4 T Cells Expressing TNFα, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 01 |
| Figure 769: | Percentages of CD4 T Cells Expressing TNFα, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | <b>)</b> 1 |
| Figure 770 | Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)40 | 01 |
| Figure 771: | Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)40 | 01 |
| Figure 772: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)40 | 01 |
| Figure 773 | Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)40 | 01 |
| Figure 774 | Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)40 | 01 |
| Figure 775 | Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)40 | 02 |
| Figure 776 | Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)40 | 02 |
| Figure 777 | Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)40 | 02 |
| Figure 778 | Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)40 | 02 |
| Figure 779 | Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)40 | 02 |
| Figure 780 | Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)40 | 02 |
| Figure 781: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)40 | 02 |
| Figure 782: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)40 | 02 |
| Figure 783: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)40 | 02 |

| Figure 784: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 102 |
|---|---|---|
| Figure 785: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)4 | 102 |
| Figure 786: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 102 |
| Figure 787: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)4 | 102 |
| Figure 788: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 102 |
| Figure 789: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)4 | 103 |
| Figure 790: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 103 |
| Figure 791: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)4 | 103 |
| Figure 792: | Percentages of CD4 T Cells Expressing IFNγ, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)4 | 103 |
| Figure 793: | Percentages of CD4 T Cells Expressing IFNγ, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)4 | 103 |
| Figure 794: | Percentages of CD4 T Cells Expressing IL-17, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)4 | 103 |
| Figure 795: | Percentages of CD4 T Cells Expressing IL-17, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 103 |
| Figure 796: | Percentages of CD4 T Cells Expressing IL-2, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)4 | 103 |
| Figure 797: | : Percentages of CD4 T Cells Expressing IL-2, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)4 | 103 |
| Figure 798: | Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 103 |
| Figure 799: | : Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S1 – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 103 |
| Figure 800: | : Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 103 |
| Figure 801: | : Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 802: | Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 403 |
|---|---|---|
| Figure 803: | Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 403 |
| Figure 804: | Percentages of CD4 T Cells Expressing TNFα, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 805: | Percentages of CD4 T Cells Expressing TNFα, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 806: | Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 807: | Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 808: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 809: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 810: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 811: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 812: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 813: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 814: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 815: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 816: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 817: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 404 |
| Figure 818: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 405 |
| Figure 819: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 405 |
| Figure 820: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 405 |

| _ | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)405 |
|---|---|
| _ | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)405 |
| | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)405 |
| | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)405 |
| _ | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)405 |
| _ | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)405 |
| _ | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)405 |
| | Percentages of CD4 T Cells Expressing IFNγ, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| | Percentages of CD4 T Cells Expressing IFNγ, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| _ | Percentages of CD4 T Cells Expressing IL-17, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| _ | Percentages of CD4 T Cells Expressing IL-17, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| _ | Percentages of CD4 T Cells Expressing IL-2, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| _ | Percentages of CD4 T Cells Expressing IL-2, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| _ | Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| _ | Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| C | Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| C | Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| | Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |

| Figure 839: | Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)406 |
|---|---|
| Figure 840: | Percentages of CD4 T Cells Expressing TNFα, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations)406 |
| Figure 841: | Percentages of CD4 T Cells Expressing TNFα, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)406 |
| Figure 842: | Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations)406 |
| Figure 843: | Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)406 |
| Figure 844: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations)406 |
| Figure 845: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)406 |
| Figure 846: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations)406 |
| Figure 847: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)407 |
| Figure 848: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations)407 |
| Figure 849: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)407 |
| Figure 850: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations)407 |
| Figure 851: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)407 |
| Figure 852: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations)407 |
| Figure 853: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 854: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations)407 |
| Figure 855: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 856: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations)407 |

| Figure 857: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
|---|---|
| Figure 858: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations)407 |
| Figure 859: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 860: | Percentages of CD4 T Cells Expressing IFN $\gamma$ or IL-2 or 154/N, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations)407 |
| Figure 861: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 862: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations)408 |
| Figure 863: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 864: | Percentages of CD4 T Cells Expressing IFNγ, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 865: | Percentages of CD4 T Cells Expressing IFNγ, Original Matched – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations)408 |
| Figure 866: | Percentages of CD4 T Cells Expressing IL-17, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 867: | Percentages of CD4 T Cells Expressing IL-17, Original Matched – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| | Percentages of CD4 T Cells Expressing IL-2, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 869: | Percentages of CD4 T Cells Expressing IL-2, Original Matched – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 870: | Percentages of CD4 T Cells Expressing IL-4 and 154, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations)408 |
| Figure 871: | Percentages of CD4 T Cells Expressing IL-4 and 154, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)408 |
| Figure 872: | Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations)408 |
| Figure 873: | Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |

| Figure 874 | : Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 408 |
|---|---|---|
| Figure 875 | Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 408 |
| Figure 876 | Percentages of CD4 T Cells Expressing TNFα, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 877: | Percentages of CD4 T Cells Expressing TNFα, Original Matched – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 878: | Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 879 | Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original S – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 880 | Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 881: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 882: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 883 | Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 884 | Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 885 | Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 886 | Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 887 | Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 888 | Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 889 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 409 |
| Figure 890 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 891: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |

| Figure 892: | Percentages of CD4 T Cells Expressing IFN $\gamma$ or IL-2 or 154/C, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations)410 |
|---|---|
| Figure 893: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)410 |
| Figure 894: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations)410 |
| Figure 895: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)410 |
| Figure 896: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations)410 |
| Figure 897: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)410 |
| Figure 898: | Percentages of CD4 T Cells Expressing IFN $\gamma$ or IL-2 or 154/T, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations)410 |
| Figure 899: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)410 |
| Figure 900: | Percentages of CD4 T Cells Expressing IFNγ, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations)410 |
| Figure 901: | Percentages of CD4 T Cells Expressing IFNγ, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 902: | Percentages of CD4 T Cells Expressing IL-17, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 903: | Percentages of CD4 T Cells Expressing IL-17, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 904: | Percentages of CD4 T Cells Expressing IL-2, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 905: | Percentages of CD4 T Cells Expressing IL-2, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 906: | Percentages of CD4 T Cells Expressing IL-4 and 154, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) |
| Figure 907: | Percentages of CD4 T Cells Expressing IL-4 and 154, Original S – Per<br>Protocol Population, Treatment Arms 2A-B (Three Vaccinations)411 |
| Figure 908: | Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations)411 |
| Figure 909: | Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)411 |
| Figure 910: | Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations)411 |

| Figure 911: | : Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 411 |
|---|---|---|
| Figure 912: | : Percentages of CD4 T Cells Expressing TNFα, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 411 |
| Figure 913: | : Percentages of CD4 T Cells Expressing TNFα, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 411 |
| Figure 914: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 412 |
| Figure 915: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta Mutations – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 413 |
| Figure 916: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 413 |
| Figure 917: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 413 |
| Figure 918: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 413 |
| Figure 919: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 413 |
| Figure 920: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 413 |
| Figure 921: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta Mutations – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 413 |
| Figure 922: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 413 |
| Figure 923: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 413 |
| Figure 924: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta<br>Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 413 |
| Figure 925: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta<br>Mutations – Per Protocol Population, Treatment Arms 2C-H (Two<br>Vaccinations) | 413 |
| Figure 926: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 413 |
| Figure 927: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta Mutations – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 413 |
| Figure 928: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta<br>Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 414 |

| Figure 929: | Percentages of CD4 T Cells Expressing IFN $\gamma$ or IL-2 or 154/C, Beta Mutations – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
|---|---|
| Figure 930: | Percentages of CD4 T Cells Expressing IFN $\gamma$ or IL-2 or 154/E, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations)414 |
| Figure 931: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta<br>Mutations – Per Protocol Population, Treatment Arms 2C-H (Two<br>Vaccinations) |
| Figure 932: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations)414 |
| Figure 933: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta<br>Mutations – Per Protocol Population, Treatment Arms 2C-H (Two<br>Vaccinations) |
| Figure 934: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations)414 |
| Figure 935: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta Mutations – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 936: | Percentages of CD4 T Cells Expressing IFNγ, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations)414 |
| Figure 937: | Percentages of CD4 T Cells Expressing IFNγ, Beta Mutations – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)414 |
| Figure 938: | Percentages of CD4 T Cells Expressing IL-17, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations)414 |
| Figure 939: | Percentages of CD4 T Cells Expressing IL-17, Beta Mutations – Per<br>Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| | Percentages of CD4 T Cells Expressing IL-2, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations)414 |
| Figure 941: | Percentages of CD4 T Cells Expressing IL-2, Beta Mutations – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 942: | Percentages of CD4 T Cells Expressing IL-4 and 154, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 943: | Percentages of CD4 T Cells Expressing IL-4 and 154, Beta Mutations – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 944: | Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations)415 |
| Figure 945: | Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta Mutations – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |

| Figure 946 | : Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta<br>Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 415 |
|---|---|---|
| Figure 947 | : Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta<br>Mutations – Per Protocol Population, Treatment Arms 2C-H (Two<br>Vaccinations) | 415 |
| Figure 948 | Percentages of CD4 T Cells Expressing TNFα, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 415 |
| Figure 949 | : Percentages of CD4 T Cells Expressing TNFα, Beta Mutations – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 415 |
| Figure 950 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 415 |
| Figure 951 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 415 |
| Figure 952 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 415 |
| Figure 953 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 415 |
| Figure 954 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 415 |
| Figure 955 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta S – Per<br>Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 415 |
| Figure 956 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 415 |
| Figure 957 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta S – Per<br>Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 415 |
| Figure 958 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 415 |
| Figure 959 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta S – Per<br>Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 416 |
| Figure 960 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 416 |
| Figure 961 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 416 |
| Figure 962 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | |
| Figure 963 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 964: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations)416 |
|---|---|
| Figure 965: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 966: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 967: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 968: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations)416 |
| Figure 969: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)416 |
| Figure 970: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 971: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 972: | Percentages of CD4 T Cells Expressing IFNγ, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 973: | Percentages of CD4 T Cells Expressing IFNγ, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)416 |
| Figure 974: | Percentages of CD4 T Cells Expressing IL-17, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 975: | Percentages of CD4 T Cells Expressing IL-17, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)417 |
| Figure 976: | Percentages of CD4 T Cells Expressing IL-2, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 977: | Percentages of CD4 T Cells Expressing IL-2, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)417 |
| Figure 978: | Percentages of CD4 T Cells Expressing IL-4 and 154, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations)417 |
| Figure 979: | Percentages of CD4 T Cells Expressing IL-4 and 154, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 980: | Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations)417 |
| Figure 981: | Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)417 |
| _ | Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |

| Figure 983: | Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 417 |
|---|---|---|
| Figure 984: | Percentages of CD4 T Cells Expressing TNFα, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 417 |
| Figure 985: | Percentages of CD4 T Cells Expressing TNFα, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 417 |
| Figure 986: | Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 417 |
| Figure 987: | Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 417 |
| Figure 988: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 417 |
| Figure 989: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 417 |
| Figure 990: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 417 |
| Figure 991: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |
| Figure 992: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |
| Figure 993: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |
| Figure 994: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |
| Figure 995: | Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |
| Figure 996: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |
| Figure 997: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |
| Figure 998: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |
| Figure 999: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |
| Figure 1000 | 0: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |

| Figure 1001: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |
|---|---|
| Figure 1002: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |
| Figure 1003: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |
| Figure 1004: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 418 |
| Figure 1005: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1006: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1007: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1008: Percentages of CD4 T Cells Expressing IFNγ, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1009: Percentages of CD4 T Cells Expressing IFNγ, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1010: Percentages of CD4 T Cells Expressing IL-17, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1011: Percentages of CD4 T Cells Expressing IL-17, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1012: Percentages of CD4 T Cells Expressing IL-2, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1013: Percentages of CD4 T Cells Expressing IL-2, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1014: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1015: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |

| Figure 1016: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two | 410 |
|---|---|
| Vaccinations) | 419 |
| Figure 1017: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1018: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1019: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1020: Percentages of CD4 T Cells Expressing TNFα, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 419 |
| Figure 1021: Percentages of CD4 T Cells Expressing TNFα, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 420 |
| Figure 1022: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 420 |
| Figure 1023: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 420 |
| Figure 1024: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 - mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 420 |
| Figure 1025: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 420 |
| Figure 1026: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 420 |
| Figure 1027: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 420 |
| Figure 1028: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 420 |
| Figure 1029: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 420 |
| Figure 1030: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 - mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 420 |
| Figure 1031: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 420 |
| Figure 1032: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 420 |

| Figure 1033: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | .420 |
|---|---|
| Figure 1034: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | .420 |
| Figure 1035: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | .421 |
| Figure 1036: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | .421 |
| Figure 1037: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | .421 |
| Figure 1038: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | .421 |
| Figure 1039: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | .421 |
| Figure 1040: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | .421 |
| Figure 1041: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | .421 |
| Figure 1042: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | .421 |
| Figure 1043: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | .421 |
| Figure 1044: Percentages of CD4 T Cells Expressing IFNγ, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | .421 |
| Figure 1045: Percentages of CD4 T Cells Expressing IFNγ, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | .421 |
| Figure 1046: Percentages of CD4 T Cells Expressing IL-17, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | .421 |
| Figure 1047: Percentages of CD4 T Cells Expressing IL-17, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | .421 |

| Figure 1048: Percentages of CD4 T Cells Expressing IL-2, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 421 |
|---|---|
| Figure 1049: Percentages of CD4 T Cells Expressing IL-2, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 421 |
| Figure 1050: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 422 |
| Figure 1051: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 422 |
| Figure 1052: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 422 |
| Figure 1053: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 422 |
| Figure 1054: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154,<br>Conserved S2 – mITT Population, Treatment Arms 2C-H (Two<br>Vaccinations) | 422 |
| Figure 1055: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154,<br>Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two<br>Vaccinations) | 422 |
| Figure 1056: Percentages of CD4 T Cells Expressing TNFα, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 422 |
| Figure 1057: Percentages of CD4 T Cells Expressing TNFα, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 422 |
| Figure 1058: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 422 |
| Figure 1059: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 422 |
| Figure 1060: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 422 |
| Figure 1061: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 422 |
| Figure 1062: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 422 |
| Figure 1063: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 422 |

| Figure 1064: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
|---|---|
| Figure 1065: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
| Figure 1066: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
| Figure 1067: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
| Figure 1068: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
| Figure 1069: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
| Figure 1070: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
| Figure 1071: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
| Figure 1072: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
| Figure 1073: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
| Figure 1074: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
| Figure 1075: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
| Figure 1076: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
| Figure 1077: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 423 |
| Figure 1078: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |

| Figure 1079: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
|---|---|
| Figure 1080: Percentages of CD4 T Cells Expressing IFNγ, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
| Figure 1081: Percentages of CD4 T Cells Expressing IFNγ, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
| Figure 1082: Percentages of CD4 T Cells Expressing IL-17, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
| Figure 1083: Percentages of CD4 T Cells Expressing IL-17, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
| Figure 1084: Percentages of CD4 T Cells Expressing IL-2, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
| Figure 1085: Percentages of CD4 T Cells Expressing IL-2, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
| Figure 1086: Percentages of CD4 T Cells Expressing IL-4 and 154, Original Matched - mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
| Figure 1087: Percentages of CD4 T Cells Expressing IL-4 and 154, Original Matched - Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
| Figure 1088: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
| Figure 1089: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
| Figure 1090: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
| Figure 1091: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
| Figure 1092: Percentages of CD4 T Cells Expressing TNFα, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 424 |
| Figure 1093: Percentages of CD4 T Cells Expressing TNFα, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 425 |
| Figure 1094: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 425 |
| Figure 1095: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 425 |

| Figure 10 | 96: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 425 |
|---|---|---|
| Figure 10 | 97: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 425 |
| Figure 10 | 98: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 425 |
| Figure 10 | 99: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 425 |
| Figure 11 | 00: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 425 |
| Figure 11 | 01: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 425 |
| Figure 11 | 02: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 425 |
| Figure 11 | 03: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 425 |
| Figure 11 | 04: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 425 |
| Figure 11 | <ul> <li>O5: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original S</li> <li>Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)</li> </ul> | 425 |
| Figure 11 | 06: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 425 |
| Figure 11 | 07: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 426 |
| Figure 11 | 08: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 426 |
| Figure 11 | 09: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 426 |
| Figure 11 | <ul> <li>10: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original S</li> <li>– mITT Population, Treatment Arms 2C-H (Two Vaccinations)</li> </ul> | 426 |
| Figure 11 | <ul> <li>11: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original S</li> <li>Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)</li> </ul> | 426 |
| Figure 11 | 12: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 426 |
| Figure 11 | <ul> <li>13: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original</li> <li>S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)</li> </ul> | 426 |
| Figure 11 | <ul> <li>14: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original S</li> <li>– mITT Population, Treatment Arms 2C-H (Two Vaccinations)</li> </ul> | 426 |

| Figure 1115: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original S - Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 426 |
|---|---|
| Figure 1116: Percentages of CD4 T Cells Expressing IFNγ, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 426 |
| Figure 1117: Percentages of CD4 T Cells Expressing IFNγ, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 426 |
| Figure 1118: Percentages of CD4 T Cells Expressing IL-17, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 426 |
| Figure 1119: Percentages of CD4 T Cells Expressing IL-17, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 426 |
| Figure 1120: Percentages of CD4 T Cells Expressing IL-2, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 426 |
| Figure 1121: Percentages of CD4 T Cells Expressing IL-2, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 426 |
| Figure 1122: Percentages of CD4 T Cells Expressing IL-4 and 154, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 426 |
| Figure 1123: Percentages of CD4 T Cells Expressing IL-4 and 154, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 426 |
| Figure 1124: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 427 |
| Figure 1125: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 427 |
| Figure 1126: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original S - mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 427 |
| Figure 1127: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original S - Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 427 |
| Figure 1128: Percentages of CD4 T Cells Expressing TNFα, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 427 |
| Figure 1129: Percentages of CD4 T Cells Expressing TNFα, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 427 |
| Figure 1130: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 428 |
| Figure 1131: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 429 |
| Figure 1132: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 429 |

| Figure 1133: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 429 |
|---|---|
| Figure 1134: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 1135: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three | 429 |
| Figure 1136: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 429 |
| Figure 1137: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 429 |
| Figure 1138: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 429 |
| Figure 1139: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 429 |
| Figure 1140: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 429 |
| Figure 1141: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 429 |
| Figure 1142: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 429 |
| Figure 1143: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 429 |
| Figure 1144: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta S – mITT | 429 |
| Figure 1145: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 429 |
| Figure 1146: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 430 |
| Figure 1147: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 1148: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 1149: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 1150: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | |
| Figure 1151: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 430 |
|---|---|
| Figure 1152: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 430 |
| Figure 1153: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 430 |
| Figure 1154: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 430 |
| Figure 1155: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 430 |
| Figure 1156: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 430 |
| Figure 1157: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 430 |
| Figure 1158: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 430 |
| Figure 1159: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 431 |
| Figure 1160: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 431 |
| Figure 1161: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 431 |
| Figure 1162: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 - mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 431 |
| Figure 1163: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 431 |
| Figure 1164: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 431 |
| Figure 1165: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 431 |
| Figure 1166: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S2 – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 431 |
| Figure 1167: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 431 |
| Figure 1168: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 - mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 431 |
| Figure 1169: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 431 |

| Figure 1170: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 431 |
|---|---|
| Figure 1171: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 431 |
| Figure 1172: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1173: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1174: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1175: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1176: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1177: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1178: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original Matched – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1179: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original Matched – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1180: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1181: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1182: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1183: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1184: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1185: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original S – Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |
| Figure 1186: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original S – mITT Population, Treatment Arms 2A-B (Three Vaccinations) | 432 |

| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original S – Per rotocol Population, Treatment Arms 2A-B (Three Vaccinations) | 433 |
|---|---|---|---|
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original S – ITT Population, Treatment Arms 2A-B (Three Vaccinations) | 433 |
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original S– Per rotocol Population, Treatment Arms 2A-B (Three Vaccinations) | 433 |
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta Mutations – ITT PopulationTreatment Arms 2C-H (Two Vaccinations) | 434 |
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta Mutations – er Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 435 |
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta Iutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 435 |
| Figure | M | Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta Intations – Per Protocol Population, Treatment Arms 2C-H (Two accinations) | 435 |
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta Iutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 435 |
| Figure | M | Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta Iutations – Per Protocol Population, Treatment Arms 2C-H (Two accinations) | 435 |
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 435 |
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 435 |
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 435 |
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 435 |
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta S – mITT opulation, Treatment Arms 2C-H (Two Vaccinations) | 435 |
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta S – Per rotocol Population, Treatment Arms 2C-H (Two Vaccinations) | 435 |
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta S – mITT opulation, Treatment Arms 2C-H (Two Vaccinations) | 435 |
| Figure | | Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta S – Per rotocol Population, Treatment Arms 2C-H (Two Vaccinations) | 435 |
| Figure | 1204: | Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta S – mITT opulation, Treatment Arms 2C-H (Two Vaccinations) | |

| Figure 1205: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
|---|
| Figure 1206: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 1207: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)436 |
| Figure 1208: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 1209: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 1210: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 1211: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 1212: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations)436 |
| Figure 1213: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 - Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 1214: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 - mITT Population, Treatment Arms 2C-H (Two Vaccinations)436 |
| Figure 1215: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 - Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 1216: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 1217: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 1218: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 – mITT Population, Treatment Arms 2C-H (Two Vaccinations)436 |
| Figure 1219: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)437 |
| Figure 1220: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 1221: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 1222: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 - mITT Population, Treatment Arms 2C-H (Two Vaccinations)437 |
| Figure 1223: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)437 |

| Figure 1224: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 437 |
|---|---|
| Figure 1225: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 437 |
| Figure 1226: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S2 – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 437 |
| Figure 1227: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 437 |
| Figure 1228: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 - mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 437 |
| Figure 1229: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 437 |
| Figure 1230: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 437 |
| Figure 1231: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 437 |
| Figure 1232: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 438 |
| Figure 1233: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 438 |
| Figure 1234: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 438 |
| Figure 1235: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 438 |
| Figure 1236: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 438 |
| Figure 1237: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 438 |
| Figure 1238: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original Matched – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 438 |
| Figure 1239: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original Matched – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) | 438 |
| Figure 1240: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) | 438 |

| Figure 1241: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)438 |
|---|
| Figure 1242: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations) |
| Figure 1243: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)438 |
| Figure 1244: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations)438 |
| Figure 1245: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)438 |
| Figure 1246: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations)438 |
| Figure 1247: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original S – Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)439 |
| Figure 1248: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original S – mITT Population, Treatment Arms 2C-H (Two Vaccinations)439 |
| Figure 1249: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original S– Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)439 |
| Figure 1250: Maximum Severity of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group – Post Dose 1 |
| Figure 1251: Maximum Severity of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group – Post Dose 2 |
| Figure 1252: Maximum Severity of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group – Post Dose 3 |
| Figure 1253: Maximum Severity of Solicited Local Symptoms by Days Post Vaccination and Treatment Group – Post Dose 1 |
| Figure 1254: Maximum Severity of Solicited Local Symptoms by Days Post Vaccination and Treatment Group – Post Dose 2 |
| Figure 1255: Maximum Severity of Solicited Local Symptoms by Days Post<br>Vaccination and Treatment Group – Post Dose 3 |
| Figure 1256: Onset of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group – Post Dose 1 |
| Figure 1257: Onset of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group – Post Dose 2 |
| Figure 1258: Onset of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group – Post Dose 3 |
| Figure 1259: Onset of Solicited Local Symptoms by Days Post Vaccination and Treatment Group – Post Dose 1 |

| | Symptoms by Days Post Vaccination and se 2445 |
|---|---|
| | Symptoms by Days Post Vaccination and se 3 |
| | Days Post Vaccination and Treatment Group –446 |
| | Days Post Vaccination and Treatment Group –447 |
| Figure 1274: Frequency of Adverse Ex | vents by MedDRA System Organ Class and448 |
| e e e e e e e e e e e e e e e e e e e | ents by MedDRA® System Organ Class and |

## 10.1 Disposition of Subjects

## Figure 1: CONSORT Flow Diagram

[Implementation Note: Below is an example CONSORT diagram. The final CONSORT will include Arms 2A-H.]



## 14.2.2 Immunogenicity Response Figures by Measure, Treatment/Vaccination, and Time Point

Figure 2: Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group - S-2P-Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

[Implementation Note: Below is an example figure. Lines will only be shown for the two three-vaccination cohort 2 groups on Days 1, 15, 29, 43, 57, 71, 85, 147, 237, and 422. The x-axis label should read "Arbitrary Units/mL (S-2P-Wa-1) (log<sub>10</sub>)." Asterisks on the Study Day labels will denote vaccination days.]



- Figure 3: Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 4: Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 5: Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 6: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 7: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 8: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 9: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 10: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 11: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 12: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 13: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 14: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 15: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 16: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 17: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 18: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 19: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 20: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 21: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 22: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 23: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 24: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 25: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 26: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 27: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 28: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 29: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 30: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 31: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 32: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 33: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 34: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 35: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 36: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 37: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 38: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 39: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 40: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 41: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 42: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 43: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 44: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 45: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 46: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 47: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 48: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 49: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 50: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 51: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 52: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 53: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 54: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 55: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 56: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 57: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 58: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 59: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 60: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 61: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 62: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 63: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 64: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 65: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 66: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 67: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 68: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 69: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 70: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 71: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 72: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 73: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 74: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 75: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 76: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 77: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 78: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 79: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 80: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 81: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 82: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 83: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 84: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 85: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Figure 86: Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group - S-2P-Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

[Implementation Note: Below is an example figure. Lines will only be shown for the six two-vaccination cohort 2 groups on Days 1, 15, 29, 43, 57, 119, 209, and 394. The x-axis label should read "Arbitrary Units/mL (S-2P-Wa-1) (log<sub>10</sub>)." Asterisks on the Study Day labels will denote vaccination days.]



- Figure 87: Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 88: Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 89: Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 90: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 91: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 92: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 93: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 94: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 95: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 96: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 97: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 98: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 99: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 100: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 101: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 102: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 103: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 104: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 105: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 106: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 107: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 108: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 109: Reverse Cumulative Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 110: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 111: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 112: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 113: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 114: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 115: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 116: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 117: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 118: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 119: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 120: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 121: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 122: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 123: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 124: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 125: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 126: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 127: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 128: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 129: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 130: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 131: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 132: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 133: Reverse Cumulative Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 134: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 135: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 136: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 137: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 138: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 139: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 140: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 141: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 142: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID50 by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 143: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 144: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 145: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 146: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 147: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 148: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 149: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 150: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID50 by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 151: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 152: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 153: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 154: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 155: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 156: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 157: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 158: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 159: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 160: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 161: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 162: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 163: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 164: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 165: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 166: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 167: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 168: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 169: Reverse Cumulative Distribution of Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Figure 170: Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P-Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

[Implementation Note: Below is an example figure. Panels will only be shown for the two three-vaccination cohort 2 groups on Days 1, 15, 29, 43, 57, 71, 85, 147, 237, and 422. The y-axis label should read "Arbitrary Units/mL (S-2P-Wa-1) (log<sub>10</sub>)." Asterisks on the Study Day labels will denote vaccination days.]



- Figure 171: Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 172: Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 173: Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 174: Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P-Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 175: Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P-Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 176: Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 177: Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 178: Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 179: Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 180: Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P-Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 181: Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 182: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P-Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 183: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 184: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 185: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 186: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 187: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 188: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 189: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 190: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 191: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 192: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 193: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 194: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 195: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 196: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 197: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 198: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 199: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 200: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 201: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 202: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 203: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 204: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 205: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 206: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 207: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 208: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 209: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 210: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 211: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 212: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 213: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 214: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 215: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 216: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 217: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 218: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 219: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 220: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 221: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 222: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 223: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 224: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 225: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 226: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 227: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 228: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 229: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 230: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 231: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 232: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 233: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 234: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 235: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 236: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 237: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 238: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 239: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 240: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 241: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 242: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 243: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 244: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 245: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 246: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 247: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 248: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 249: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 250: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 251: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 252: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 253: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Figure 254: Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P-Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

[Implementation Note: Below is an example figure. Panels will only be shown for the two three-vaccination cohort 2 groups on Days 1, 15, 29, 43, 57, 119, 209, and 394. The y-axis label should read "Arbitrary Units/mL (S-2P-Wa-1) (log<sub>10</sub>)." Asterisks on the Study Day labels will denote vaccination days.]



- Figure 255: Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 256: Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 257: Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 258: Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P-Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 259: Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P-Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 260: Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 261: Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 262: Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 263: Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 264: Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P-Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 265: Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 266: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 267: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 268: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 269: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 270: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 271: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 272: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 273: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 274: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 275: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 276: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 277: Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 278: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 279: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 280: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 281: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 282: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 283: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 284: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 285: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 286: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 287: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 288: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 289: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 290: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 291: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 292: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 293: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 294: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 295: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 296: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 297: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 298: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 299: Pseudovirus Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 300: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 301: Pseudovirus Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 302: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 303: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 304: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 305: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 306: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 307: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 308: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 309: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 310: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 311: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 312: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 313: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 314: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 315: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 316: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 317: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 318: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 319: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 320: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 321: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 322: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 323: Focus Reduction Neutralization Assay ID<sub>50</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 324: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 325: Focus Reduction Neutralization Assay ID<sub>80</sub> by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 326: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 327: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Figure 337:

Focus Reduction Neutralization Assay (TMPRS cells) ID80 by Time Point and Treatment Figure 328: Group – D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations) Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Figure 329: **Group – D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)** Figure 330: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>50</sub> by Time Point and Treatment **Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)** Focus Reduction Neutralization Assay (TMPRS cells) ID50 by Time Point and Treatment Figure 331: **Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)** Figure 332: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group – B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations) Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Figure 333: Group – B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) Figure 334: Focus Reduction Neutralization Assay (TMPRS cells) ID50 by Time Point and Treatment **Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)** Focus Reduction Neutralization Assay (TMPRS cells) ID50 by Time Point and Treatment Figure 335: Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations) Figure 336: Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment **Group – B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)** 

Focus Reduction Neutralization Assay (TMPRS cells) ID<sub>80</sub> by Time Point and Treatment Group – B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
Figure 338: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P-Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

[Implementation Note: Below is an example figure. Lines will only be shown for the two three-vaccination cohort 2 groups on Days 1, 15, 29, 43, 57, 71, 85, 147, 237, and 422. The y-axis label should read "Arbitrary Units/mL (S-2P-Wa-1) (log<sub>10</sub>)." Asterisks on the Study Day labels will denote vaccination days.]]



- Figure 339: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group S-2P-Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 340: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 341: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 342: Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 343: Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 344: Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 345: Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 346: Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 347: Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 348: Geometric Mean Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 349: Geometric Mean Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 350: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 351: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 352: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point

- and Treatment Group S-2P– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 353: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 354: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 355: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 356: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 357: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 358: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 359: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 360: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 361: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 362: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 363: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 364: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 365: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 366: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 367: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 368: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 369: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 370: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 371: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 372: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 373: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 374: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 375: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 376: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 377: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 378: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 379: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 380: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 381: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 382: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 383: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 384: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 385: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 386: Geometric Mean Focus Reduction Neutralization Test ID50 Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 387: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 388: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 389: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 390: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 391: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 392: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 393: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 394: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 395: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 396: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 397: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 398: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 399: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 400: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 401: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 402: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 403: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 404: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 405: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 406: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 407: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 408: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 409: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 410: Geometric Mean Focus Reduction Neutralization Test (TMPRS cells) ID50 Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 411: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 412: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 413: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 414: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 415: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 416: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 417: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 418: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 419: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 420: Geometric Mean Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 421: Geometric Mean Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Figure 422: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P-Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

[Implementation Note: Below is an example figure. Lines will only be shown for the two three-vaccination cohort 2 groups on Days 1, 15, 29, 43, 57, 119, 209, and 394. The y-axis label should read "Arbitrary Units/mL (S-2P-Wa-1) (log<sub>10</sub>)." Asterisks on the Study Day labels will denote vaccination days.]]



- Figure 423: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 424: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 425: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 426: Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 427: Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 428: Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 429: Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 430: Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 431: Geometric Mean Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 432: Geometric Mean Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 433: Geometric Mean Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 434: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 435: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 436: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point

- and Treatment Group S-2P– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 437: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 438: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 439: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 440: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 441: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 442: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 443: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 444: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 445: Geometric Mean Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 446: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 447: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 448: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 449: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 450: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 451: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 452: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 453: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 454: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 455: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 456: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 457: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 458: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 459: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 460: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 461: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 462: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 463: Geometric Mean Pseudovirus Neutralization Assay ID50 Titers by Time Point and

- Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 464: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 465: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 466: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 467: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 468: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 469: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 470: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 471: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 472: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 473: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 474: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 475: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 476: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 477: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 478: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 479: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 480: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 481: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 482: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 483: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 484: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 485: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 486: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 487: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 488: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 489: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 490: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 491: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 492: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 493: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 494: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 495: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 496: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 497: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 498: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 499: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 500: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 501: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 502: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 503: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 504: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 505: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> (TMPRS cells) Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Figure 506: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P-Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

[Implementation note: Below is an example figure. Plots will only be shown for the two three-vaccination cohort 2 groups on Days 1, 15, 29, 43, 57, 71, 85, 147, 237, and 422 The y-axis label should read "Arbitrary Units/mL (S-2P-Wa-1) (log<sub>10</sub>)." Asterisks on the Study Day labels will denote vaccination days.].]



- Figure 507: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 508: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 509: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 510: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 511: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 512: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 513: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 514: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 515: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 516: Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 517: Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 518: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 519: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 520: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 521: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 522: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 523: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 524: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 525: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 526: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 527: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 528: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 529: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 530: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 531: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 532: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 533: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 534: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 535: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 536: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 537: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 538: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 539: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 540: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 541: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 542: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 543: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 544: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 545: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 546: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 547: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 548: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 549: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 550: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 551: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 552: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 553: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 554: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 555: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 556: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 557: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 558: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 559: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 560: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 561: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 562: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 563: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 564: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 565: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 566: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 567: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 568: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 569: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 570: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 571: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 572: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 573: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 574: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 575: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 576: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 577: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 578: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID50 Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 579: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 580: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 581: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 582: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID50 Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 583: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID50 Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 584: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 585: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 586: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 587: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 588: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 589: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Figure 590: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P-Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

[Implementation note: Below is an example figure. Plots will only be shown for the six two-vaccination cohort 2 groups on Days 1, 15, 29, 43, 57, 119, 209, and 394. The y-axis label should read "Arbitrary Units/mL (S-2P-Wa-1) (log<sub>10</sub>)." Asterisks on the Study Day labels will denote vaccination days.]]



- Figure 591: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 592: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 593: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 594: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 595: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 596: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 597: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group S-2P–B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 598: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 599: Distribution of Serum IgG ECLIAv2 (4-plex) Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 600: Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 601: Distribution of Serum IgG ECLIAv2 (4-plex) Binding Antibody Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 602: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 603: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 604: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 605: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 606: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 607: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 608: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 609: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 610: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 611: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 612: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 613: Distribution of Serum IgG ECLIAv2 (10-plex) Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 614: Distribution of Pseudovirus Neutralization Assay ID50 Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 615: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 616: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 617: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 618: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 619: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 620: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 621: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 622: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 623: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 624: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 625: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 626: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 627: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 628: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 629: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 630: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 631: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 632: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 633: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 634: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 635: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 636: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 637: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 638: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 639: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 640: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 641: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 642: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 643: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 644: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 645: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 646: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 647: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 648: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 649: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 650: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 651: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 652: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 653: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 654: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 655: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 656: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 657: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 658: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 659: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 660: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 661: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 662: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID50 Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 663: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID50 Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 664: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 665: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 666: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID50 Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 667: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 668: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 669: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 670: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 671: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 672: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 673: Distribution of Focus Reduction Neutralization Test (TMPRS cells) ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.529, Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

[Implementation note: Below is a sample figure. The figure will include all immunoassays which measured D614G.]

Figure 674: Correlation Heatmap, D614G – mITT Population, Treatment Arms 2A-B (Three Vaccinations)



- Figure 675: Correlation Heatmap, D614G Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 676: Correlation Heatmap, B.1.351 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 677: Correlation Heatmap, B.1.351 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 678: Correlation Heatmap, B.1.617.2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 679: Correlation Heatmap, B.1.617.2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 680: Correlation Heatmap, P.1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 681: Correlation Heatmap, P.1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 682: Correlation Heatmap, B.1.1.7 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 683: Correlation Heatmap, B.1.1.7 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 684: Correlation Heatmap, B.1.1.529 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 685: Correlation Heatmap, B.1.1.529 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Figure 686: Correlation Heatmap, D614G – mITT Population, Treatment Arms 2C-H (Two Vaccinations)

| ELISA AUC<br>RBD | N=707<br>0.962<br>(0.956, 0.967) | N=707<br>0.975<br>(0.971, 0.978) | N=706<br>0.921<br>(0.909, 0.931) | N=245<br>0.930<br>(0.910, 0.945) | N=665<br>0.900<br>(0.884, 0.913) | N=80<br>0.656<br>(0.509, 0.765) |
|---|---|---|---|---|---|---|
| | ELISA AUC<br>S-2P | N=707<br>0.936<br>(0.926, 0.944) | N=706<br>0.968<br>(0.963, 0.972) | N=245<br>0.895<br>(0.867, 0.917) | N=665<br>0.871<br>(0.852, 0.889) | N=80<br>0.584<br>(0.418, 0.713) |
| | | Endpoint Titer<br>RBD | N=706<br>0.903<br>(0.889, 0.916) | N=245<br>0.879<br>(0.847, 0.905) | N=665<br>0.867<br>(0.847, 0.885) | N=80<br>0.568<br>(0.398, 0.701) |
| | | | Endpoint Titer<br>S-2P | N=245<br>0.846<br>(0.806, 0.878) | N=664<br>0.842<br>(0.819, 0.863) | N=80<br>0.529<br>(0.350, 0.671) |
| | | | | FRNT-mNG<br>ID <sub>50</sub> | N=245<br>0.930<br>(0.910, 0.945) | N=80<br>0.781<br>(0.678, 0.854) |
| | | | | | PsVNA (614D)<br>ID <sub>50</sub> | N=80<br>0.611<br>(0.452, 0.733) |
| | | | | | | Live-Virus Neut<br>PRNT <sub>80</sub> |

- Figure 687: Correlation Heatmap, D614G Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 688: Correlation Heatmap, B.1.351 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 689: Correlation Heatmap, B.1.351 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 690: Correlation Heatmap, B.1.617.2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 691: Correlation Heatmap, B.1.617.2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 692: Correlation Heatmap, P.1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 693: Correlation Heatmap, P.1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 694: Correlation Heatmap, B.1.1.7 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 695: Correlation Heatmap, B.1.1.7 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 696: Correlation Heatmap, B.1.1.529 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 697: Correlation Heatmap, B.1.1.529 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
Figure 698: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations)

[Implementation note: Below is a sample figure. There will be two panels (2 rows, 1 column) for the two three-vaccination cohort 2 groups on Days 1, 15, 29, 43, 57, 71, 85, 147, 237, and 422.]



Note: Open symbols represent Non-responders and closed symbols represent responders. Plots are annotated with Responder Rate.

## Figures with Similar Format:

- Figure 699: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 700: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 701: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 702: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 703: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 704: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 705: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 706: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 707: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 708: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 709: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 710: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 711: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 712: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 713: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 714: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 715: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 716: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 717: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 718: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 719: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 720: Percentages of CD4 T Cells Expressing IFNy, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 721: Percentages of CD4 T Cells Expressing IFNγ, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 722: Percentages of CD4 T Cells Expressing IL-17, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 723: Percentages of CD4 T Cells Expressing IL-17, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 724: Percentages of CD4 T Cells Expressing IL-2, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 725: Percentages of CD4 T Cells Expressing IL-2, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 726: Percentages of CD4 T Cells Expressing IL-4 and 154, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 727: Percentages of CD4 T Cells Expressing IL-4 and 154, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 728: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 729: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 730: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 731: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 732: Percentages of CD4 T Cells Expressing TNFα, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 733: Percentages of CD4 T Cells Expressing TNFα, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 734: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 735: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 736: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 737: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 738: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 739: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 740: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 741: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 742: Percentages of CD4 T Cells Expressing IFNy or IL-2/TD, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 743: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 744: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 745: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 746: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 747: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 748: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 749: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 750: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 751: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 752: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 753: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 754: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 755: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 756: Percentages of CD4 T Cells Expressing IFNγ, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 757: Percentages of CD4 T Cells Expressing IFNγ, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 758: Percentages of CD4 T Cells Expressing IL-17, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 759: Percentages of CD4 T Cells Expressing IL-17, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 760: Percentages of CD4 T Cells Expressing IL-2, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 761: Percentages of CD4 T Cells Expressing IL-2, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 762: Percentages of CD4 T Cells Expressing IL-4 and 154, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 763: Percentages of CD4 T Cells Expressing IL-4 and 154, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 764: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 765: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 766: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 767: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 768: Percentages of CD4 T Cells Expressing TNFα, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 769: Percentages of CD4 T Cells Expressing TNFα, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 770: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 771: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 772: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 773: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 774: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 775: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 776: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 777: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 778: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 779: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 780: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 781: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 782: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 783: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 784: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 785: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 786: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 787: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 788: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 789: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 790: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 791: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 792: Percentages of CD4 T Cells Expressing IFNγ, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 793: Percentages of CD4 T Cells Expressing IFNγ, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 794: Percentages of CD4 T Cells Expressing IL-17, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 795: Percentages of CD4 T Cells Expressing IL-17, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 796: Percentages of CD4 T Cells Expressing IL-2, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 797: Percentages of CD4 T Cells Expressing IL-2, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 798: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 799: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 800: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 801: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 802: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 803: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 804: Percentages of CD4 T Cells Expressing TNFα, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 805: Percentages of CD4 T Cells Expressing TNFα, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 806: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 807: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 808: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 809: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 810: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 811: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 812: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 813: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 814: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 815: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 816: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 817: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 818: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 819: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 820: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 821: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 822: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 823: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 824: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 825: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 826: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 827: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 828: Percentages of CD4 T Cells Expressing IFNγ, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 829: Percentages of CD4 T Cells Expressing IFNγ, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 830: Percentages of CD4 T Cells Expressing IL-17, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 831: Percentages of CD4 T Cells Expressing IL-17, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 832: Percentages of CD4 T Cells Expressing IL-2, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 833: Percentages of CD4 T Cells Expressing IL-2, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 834: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 835: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 836: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 837: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 838: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 839: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 840: Percentages of CD4 T Cells Expressing TNFα, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 841: Percentages of CD4 T Cells Expressing TNFα, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 842: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 843: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 844: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 845: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 846: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 847: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 848: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 849: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 850: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 851: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 852: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 853: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 854: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 855: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 856: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 857: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 858: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 859: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 860: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 861: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 862: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 863: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 864: Percentages of CD4 T Cells Expressing IFNγ, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 865: Percentages of CD4 T Cells Expressing IFNγ, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 866: Percentages of CD4 T Cells Expressing IL-17, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 867: Percentages of CD4 T Cells Expressing IL-17, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 868: Percentages of CD4 T Cells Expressing IL-2, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 869: Percentages of CD4 T Cells Expressing IL-2, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 870: Percentages of CD4 T Cells Expressing IL-4 and 154, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 871: Percentages of CD4 T Cells Expressing IL-4 and 154, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 872: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 873: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 874: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 875: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 876: Percentages of CD4 T Cells Expressing TNFα, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 877: Percentages of CD4 T Cells Expressing TNFα, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 878: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 879: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 880: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 881: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 882: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 883: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 884: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 885: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 886: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 887: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 888: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 889: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 890: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 891: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 892: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 893: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 894: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 895: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 896: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 897: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 898: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 899: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 900: Percentages of CD4 T Cells Expressing IFNγ, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 901: Percentages of CD4 T Cells Expressing IFNγ, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 902: Percentages of CD4 T Cells Expressing IL-17, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 903: Percentages of CD4 T Cells Expressing IL-17, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 904: Percentages of CD4 T Cells Expressing IL-2, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 905: Percentages of CD4 T Cells Expressing IL-2, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 906: Percentages of CD4 T Cells Expressing IL-4 and 154, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 907: Percentages of CD4 T Cells Expressing IL-4 and 154, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 908: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 909: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 910: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 911: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 912: Percentages of CD4 T Cells Expressing TNFα, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 913: Percentages of CD4 T Cells Expressing TNFα, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Figure 914: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta Mutations – mITT Population, Treatment Arms 2C-H (Two Vaccinations)

[Implementation note: Below is a sample figure. There will be six panels (2 rows, 3 columns) for the six two-vaccination cohort 2 groups on Days 1, 15, 29, 43, 57, 91, 209, and 394.]



Note: Open symbols represent Non-responders and closed symbols represent responders. Plots are annotated with Responder Rate.

## Figures with Similar Format:

- Figure 915: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 916: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 917: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 918: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 919: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 920: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 921: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 922: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 923: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 924: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 925: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 926: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 927: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 928: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 929: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 930: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 931: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 932: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 933: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 934: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 935: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 936: Percentages of CD4 T Cells Expressing IFNy, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 937: Percentages of CD4 T Cells Expressing IFNγ, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 938: Percentages of CD4 T Cells Expressing IL-17, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 939: Percentages of CD4 T Cells Expressing IL-17, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 940: Percentages of CD4 T Cells Expressing IL-2, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 941: Percentages of CD4 T Cells Expressing IL-2, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 942: Percentages of CD4 T Cells Expressing IL-4 and 154, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 943: Percentages of CD4 T Cells Expressing IL-4 and 154, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 944: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 945: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 946: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 947: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 948: Percentages of CD4 T Cells Expressing TNFα, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 949: Percentages of CD4 T Cells Expressing TNFα, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 950: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 951: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 952: Percentages of CD4 T Cells Expressing IFNy or IL-2/CM, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 953: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 954: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 955: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 956: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 957: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 958: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 959: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 960: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 961: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 962: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 963: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 964: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 965: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 966: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 967: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 968: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 969: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 970: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 971: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 972: Percentages of CD4 T Cells Expressing IFNγ, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 973: Percentages of CD4 T Cells Expressing IFNγ, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 974: Percentages of CD4 T Cells Expressing IL-17, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 975: Percentages of CD4 T Cells Expressing IL-17, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 976: Percentages of CD4 T Cells Expressing IL-2, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 977: Percentages of CD4 T Cells Expressing IL-2, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 978: Percentages of CD4 T Cells Expressing IL-4 and 154, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 979: Percentages of CD4 T Cells Expressing IL-4 and 154, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 980: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 981: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 982: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 983: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 984: Percentages of CD4 T Cells Expressing TNFa, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 985: Percentages of CD4 T Cells Expressing TNFα, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 986: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 987: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 988: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 989: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 990: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 991: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 992: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 993: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 994: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 995: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 996: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 997: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 998: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 999: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1000: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1001: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1002: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1003: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1004: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 1005: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1006: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1007: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1008: Percentages of CD4 T Cells Expressing IFNγ, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1009: Percentages of CD4 T Cells Expressing IFNγ, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1010: Percentages of CD4 T Cells Expressing IL-17, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1011: Percentages of CD4 T Cells Expressing IL-17, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1012: Percentages of CD4 T Cells Expressing IL-2, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1013: Percentages of CD4 T Cells Expressing IL-2, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1014: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1015: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1016: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1017: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1018: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1019: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1020: Percentages of CD4 T Cells Expressing TNFα, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 1021: Percentages of CD4 T Cells Expressing TNFα, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1022: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1023: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1024: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1025: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1026: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1027: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1028: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1029: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1030: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1031: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1032: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1033: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1034: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 1035: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1036: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1037: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1038: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1039: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1040: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1041: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1042: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1043: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1044: Percentages of CD4 T Cells Expressing IFNγ, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1045: Percentages of CD4 T Cells Expressing IFNγ, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1046: Percentages of CD4 T Cells Expressing IL-17, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1047: Percentages of CD4 T Cells Expressing IL-17, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1048: Percentages of CD4 T Cells Expressing IL-2, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1049: Percentages of CD4 T Cells Expressing IL-2, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 1050: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1051: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1052: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1053: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1054: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1055: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1056: Percentages of CD4 T Cells Expressing TNFα, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1057: Percentages of CD4 T Cells Expressing TNFα, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1058: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1059: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1060: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1061: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1062: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1063: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 1064: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1065: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1066: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1067: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1068: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1069: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1070: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1071: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1072: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1073: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1074: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1075: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1076: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1077: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 1078: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1079: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1080: Percentages of CD4 T Cells Expressing IFNγ, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1081: Percentages of CD4 T Cells Expressing IFNγ, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1082: Percentages of CD4 T Cells Expressing IL-17, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1083: Percentages of CD4 T Cells Expressing IL-17, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1084: Percentages of CD4 T Cells Expressing IL-2, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1085: Percentages of CD4 T Cells Expressing IL-2, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1086: Percentages of CD4 T Cells Expressing IL-4 and 154, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1087: Percentages of CD4 T Cells Expressing IL-4 and 154, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1088: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1089: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1090: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1091: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1092: Percentages of CD4 T Cells Expressing TNFα, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 1093: Percentages of CD4 T Cells Expressing TNFα, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1094: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1095: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1096: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1097: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1098: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1099: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1100: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1101: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1102: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1103: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1104: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1105: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1106: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 1107: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1108: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1109: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1110: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1111: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1112: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1113: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1114: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1115: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1116: Percentages of CD4 T Cells Expressing IFNy, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1117: Percentages of CD4 T Cells Expressing IFNγ, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1118: Percentages of CD4 T Cells Expressing IL-17, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1119: Percentages of CD4 T Cells Expressing IL-17, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1120: Percentages of CD4 T Cells Expressing IL-2, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1121: Percentages of CD4 T Cells Expressing IL-2, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1122: Percentages of CD4 T Cells Expressing IL-4 and 154, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1123: Percentages of CD4 T Cells Expressing IL-4 and 154, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 1124: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1125: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1126: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1127: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1128: Percentages of CD4 T Cells Expressing TNFα, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1129: Percentages of CD4 T Cells Expressing TNFα, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

Figure 1130: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta Mutations – mITT Population, Treatment Arms 2A-B (Three Vaccinations)

[Implementation note: Below is a sample figure. There will be two panels (2 rows, 1 column) for the two three-vaccination cohort 2 groups on Days 1, 15, 29, 43, 57, 71, 85, 147, 237, and 422.]



Figures with Similar Format:

- Figure 1131: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1132: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1133: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1134: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1135: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1136: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1137: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1138: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1139: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1140: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1141: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1142: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1143: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1144: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1145: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 1146: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1147: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1148: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1149: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1150: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1151: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1152: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1153: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1154: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1155: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1156: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1157: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1158: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 mITT Population, Treatment Arms 2A-B (Three Vaccinations)

- Figure 1159: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1160: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1161: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1162: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1163: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1164: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1165: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1166: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1167: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1168: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1169: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1170: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1171: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1172: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1173: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1174: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1175: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1176: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1177: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1178: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original Matched mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1179: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original Matched Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1180: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1181: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1182: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1183: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1184: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1185: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1186: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original S mITT Population, Treatment Arms 2A-B

(Three Vaccinations)

- Figure 1187: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original S Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1188: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original S mITT Population, Treatment Arms 2A-B (Three Vaccinations)
- Figure 1189: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original S– Per Protocol Population, Treatment Arms 2A-B (Three Vaccinations)

Figure 1190: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta Mutations – mITT Population Treatment Arms 2C-H (Two Vaccinations)

[Implementation note: Below is a sample figure. There will be six panels (2 rows, 3 columns) for the six two-vaccination cohort 2 groups on Days 1, 15, 29, 43, 57, 91, 209, and 394.]



#### Figures with Similar Format:

- Figure 1191: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1192: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1193: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1194: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1195: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1196: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1197: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1198: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1199: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1200: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1201: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1202: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1203: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1204: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1205: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta S Per Protocol Population, Treatment Arms 2C-H

- (Two Vaccinations)
- Figure 1206: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1207: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1208: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1209: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1210: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1211: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1212: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1213: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1214: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1215: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1216: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1217: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1218: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 mITT Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 1219: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1220: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1221: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1222: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1223: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1224: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1225: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1226: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1227: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1228: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1229: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1230: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1231: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

- Figure 1232: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1233: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1234: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1235: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1236: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1237: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1238: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original Matched mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1239: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original Matched Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1240: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1241: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1242: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1243: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1244: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1245: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1246: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original S mITT Population, Treatment Arms 2C-H

(Two Vaccinations)

- Figure 1247: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original S Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1248: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original S mITT Population, Treatment Arms 2C-H (Two Vaccinations)
- Figure 1249: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original S– Per Protocol Population, Treatment Arms 2C-H (Two Vaccinations)

#### 14.3.1.1 Solicited Adverse Events

Figure 1250: Maximum Severity of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group – Post Dose 1

[Implementation Note: Panels will only be shown for the eight Cohort 2 groups.]



Figures with Similar Format:

Figure 1251: Maximum Severity of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group – Post Dose 2

Figure 1252: Maximum Severity of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group – Post Dose 3

[Implementation note: This figure will only have two panels for Arms 2A-B.]

Figure 1253: Maximum Severity of Solicited Local Symptoms by Days Post Vaccination and Treatment Group – Post Dose 1

[Implementation Note: Panels will only be shown for the eight Cohort 2 groups.]



Figures with Similar Format:

Figure 1254: Maximum Severity of Solicited Local Symptoms by Days Post Vaccination and Treatment Group – Post Dose 2

Figure 1255: Maximum Severity of Solicited Local Symptoms by Days Post Vaccination and Treatment Group – Post Dose 3

[Implementation note: This figure will only have two panels for Arms 2A-B.]

Figure 1256: Onset of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group –
Post Dose 1

[Implementation Note: Panels will only be shown for the eight Cohort 2 groups.]



Figures with Similar Format:

- Figure 1257: Onset of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group Post Dose 2
- Figure 1258: Onset of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group Post Dose 3

[Implementation note: This figure will only have two panels for Arms 2A-B.]

- Figure 1259: Onset of Solicited Local Symptoms by Days Post Vaccination and Treatment Group Post Dose 1
- Figure 1260: Onset of Solicited Local Symptoms by Days Post Vaccination and Treatment Group Post Dose 2
- Figure 1261: Onset of Solicited Local Symptoms by Days Post Vaccination and Treatment Group Post Dose 3

[Implementation note: This figure will only have two panels for Arms 2A-B.]

Figure 1262: Solicited Symptoms by Days Post Vaccination and Treatment Group - Arthralgia

[Implementation note: Figure should be three columns with plots for each treatment arm. The third column (for Dose 3) will have plots for arms A and B only.]



#### Figures with Similar Format:

- Figure 1263: Solicited Symptoms by Days Post Vaccination and Treatment Group Feverishness
- Figure 1264: Solicited Symptoms by Days Post Vaccination and Treatment Group Erythema
- Figure 1265: Solicited Symptoms by Days Post Vaccination and Treatment Group Erythema (mm)
- Figure 1266: Solicited Symptoms by Days Post Vaccination and Treatment Group Fatigue
- Figure 1267: Solicited Symptoms by Days Post Vaccination and Treatment Group Fever
- Figure 1268: Solicited Symptoms by Days Post Vaccination and Treatment Group Headache
- Figure 1269: Solicited Symptoms by Days Post Vaccination and Treatment Group Induration
- Figure 1270: Solicited Symptoms by Days Post Vaccination and Treatment Group Induration (mm)
- Figure 1271: Solicited Symptoms by Days Post Vaccination and Treatment Group Myalgia
- Figure 1272: Solicited Symptoms by Days Post Vaccination and Treatment Group Nausea
- Figure 1273: Solicited Symptoms by Days Post Vaccination and Treatment Group Pain

#### 14.3.1.2 Unsolicited Adverse Events

Figure 1274: Frequency of Adverse Events by MedDRA System Organ Class and Severity

[Implementation Note: Figure should have columns for all eight treatment arms.]



Figure 1275: Incidence of Adverse Events by MedDRA® System Organ Class and Maximum Severity [Implementation Note: Figure should have columns for all eight treatment arms.]



# 14.3.5 Displays of Laboratory Results

Not Applicable.

# APPENDIX 3. LISTINGS MOCK-UPS

## **LISTINGS**

| Listing 1: | 16.1.6: Listing of Subjects Receiving Investigational Product | 452 |
|---|---|---|
| Listing 2: | 16.2.1: Early Terminations or Discontinued Subjects | 453 |
| Listing 3: | 16.2.2.1: Subject-Specific Protocol Deviations | 454 |
| Listing 4: | 16.2.2.2: Non-Subject-Specific Protocol Deviations | 455 |
| Listing 5: | 16.2.3: Subjects Excluded from Analysis Populations | 456 |
| Listing 6: | 16.2.4.1: Demographic Data | 457 |
| Listing 7: | 16.2.4.2: Pre-Existing and Concurrent Medical Conditions | 458 |
| Listing 8: | 16.2.6: Individual Immunogenicity Response Data | 460 |
| Listing 9: | 16.2.6: Individual T-cell Response Data | 460 |
| Listing 10: | 16.2.7.1: Solicited Events – Systemic Symptoms | 461 |
| Listing 11: | 16.2.7.2: Solicited Events – Local Symptoms | 462 |
| Listing 12: | 16.2.7.3: Unsolicited Adverse Events | 463 |
| Listing 13: | 16.2.9.1: Vital Signs | 465 |
| Listing 14: | 16.2.9.2: Physical Exam Findings | 466 |
| Listing 15: | 16.2.10: Concomitant Medications | 467 |
| Listing 16: | 16.2.11.1: Pregnancy Reports – Maternal Information | 468 |
| Listing 17: | 16.2.11.2: Pregnancy Reports – Gravida and Para | 468 |
| Listing 18: | 16.2.11.3: Pregnancy Reports – Live Birth Outcomes | 469 |
| Listing 19: | 16.2.11.4: Pregnancy Reports – Still Birth Outcomes | 469 |
| Listing 20: | 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes | 469 |

## Listing 1: 16.1.6: Listing of Subjects Receiving Investigational Product

(not included in SAP, but this is a placeholder for the CSR)

## 16.2 Database Listings by Subject

### **16.2.1 Discontinued Subjects**

## **Listing 2:** 16.2.1: Early Terminations or Discontinued Subjects

| Treatment Group | Subject ID | Category | Reason for Early Termination or Treatment Discontinuation | Study Day |
|---|---|---|---|---|

### **16.2.2 Protocol Deviations**

### **Listing 3:** 16.2.2.1: Subject-Specific Protocol Deviations

| Treatment<br>Group | Subject<br>ID | DV<br>Number | Deviation | Deviation<br>Category | Deviation<br>Severity | Study<br>Day | Reason<br>for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation Resulted in Subject Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

## Listing 4: 16.2.2.2: Non-Subject-Specific Protocol Deviations

| S | Site | Deviation<br>Number | Deviation | Deviation Severity | Reason for<br>Deviation | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|

### 16.2.3 Subjects Excluded from the Efficacy Analysis

### **Listing 5:** 16.2.3: Subjects Excluded from Analysis Populations

| Treatment Group | Subject ID | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason Subject Excluded |
|---|---|---|---|---|---|
| | | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Day x] | | |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

## 16.2.4 Demographic Data

# Listing 6: 16.2.4.1: Demographic Data

| Treatment<br>Group | Subject ID | Sex | Age at Enrollment (years) | Ethnicity | Race | BMI |
|---|---|---|---|---|---|---|

# Listing 7: 16.2.4.2: Pre-Existing and Concurrent Medical Conditions

| Treatment<br>Group | Subject ID | MH Number | Medical History Term | Condition Start Day | Condition End Day | MedDRA System Organ Class | MedDRA Preferred Term |
|---|---|---|---|---|---|---|---|

## 16.2.5 Compliance and/or Drug Concentration Data (if available)

Not Applicable.

### 16.2.6 Individual Immunogenicity Response Data

Listing 8: 16.2.6: Individual Immunogenicity Response Data

| Treatment<br>Group | Subject ID | Planned Time Point | Actual Study Day | Assay | Units | Results |
|---|---|---|---|---|---|---|

## **Listing 9:** 16.2.6: Individual T-cell Response Data

| Treatment<br>Group | Subject ID | Planned Time Point | Actual Study Day | T-Cell | Peptide Pool | Cytokine | Adjusted Percent | Responder (Y/N) |
|---|---|---|---|---|---|---|---|---|

#### 16.2.7 Adverse Events

### **Listing 10:** 16.2.7.1: Solicited Events – Systemic Symptoms

| Treatment<br>Group | Subject ID | Post Dose Day | Assessmenta | Symptom | Severity | Attributed to<br>Alternate<br>Etiology? <sup>b</sup> | Alternate Etiology |
|---|---|---|---|---|---|---|---|
| | | | MA | | | | |
| | | | Clinic | | | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

<sup>&</sup>lt;sup>b</sup> Grade 3 events only.

**Listing 11:** 16.2.7.2: Solicited Events – Local Symptoms

| Treatment<br>Group | Subject ID | Post Dose Day | Assessment <sup>a</sup> | Symptom | Severity |
|---|---|---|---|---|---|
| | | | MA | | |
| | | | Clinic | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

## Listing 12: 16.2.7.3: Unsolicited Adverse Events

| Adverse<br>Event | Associated with Dose No. | No. of Days Post Associated Dose (Duration) | Severity | SAE? | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment ( | Group: , Subject | ID: , AE Numbe | er: | | | | | | | | |
| Comments: | <u> </u> | | | l | l | | | | | | |
| Treatment ( | Group: , Subject | ID: , AE Numbe | er: | | | | | | | | |
| Comments: | 1 | | l | 1 | l | | | | | | |
| Note: For a | dditional details | s about SAEs, se | ee Table: xx. | | | | | | | | |

## 16.2.8 Individual Laboratory Measurements

Not Applicable.

### 16.2.9 Vital Signs and Physical Exam Findings

Listing 13: 16.2.9.1: Vital Signs

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual Study<br>Day | Temperature<br>(°C) | Systolic Blood<br>Pressure<br>(mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Heart Rate<br>(beats/min) | Weight (kg) | Height (cm) |
|---|---|---|---|---|---|---|---|---|---|

Listing 14: 16.2.9.2: Physical Exam Findings

| Treatment<br>Group | Subject ID | Visit<br>Number | Body System | Interpretation | If Abnormal,<br>Findings | If Abnormal,<br>Reported as an AE? |
|---|---|---|---|---|---|---|

### **16.2.10** Concomitant Medications

### **Listing 15:** 16.2.10: Concomitant Medications

| Treatment<br>Group | Subject<br>ID | CM<br>Number | Medication | Medication Start<br>Day | Medication End<br>Day | Indication | Taken for an AE? (AE Description; Number) | Taken for a condition<br>on Medical History?<br>(MH Description;<br>Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|---|---|

#### 16.2.11 Pregnancy Reports

### **Listing 16:** 16.2.11.1: Pregnancy Reports – Maternal Information

| Treatment<br>Group | Subject<br>ID | Pregnancy<br>Number | Study Day<br>Corresponding<br>to Estimated<br>Date of<br>Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco,<br>Alcohol, or<br>Drug Use<br>During<br>Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or<br>Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| _ | | | | | | | | | | | |

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

### Listing 17: 16.2.11.2: Pregnancy Reports – Gravida and Para

| | | | | Live Births | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Pregnancy<br>Number | Gravida | Extremely<br>PB <sup>a</sup> | Very<br>Early<br>PB <sup>a</sup> | Early<br>PB <sup>a</sup> | Late<br>PB <sup>a</sup> | Early<br>TB <sup>b</sup> | Full<br>TB <sup>b</sup> | Late<br>TB <sup>b</sup> | Post<br>TB <sup>b</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly<br>with<br>Previous<br>Pregnancy? |

Note: Gravida includes the current pregnancy, para events do not.

<sup>&</sup>lt;sup>a</sup> Preterm Birth

<sup>&</sup>lt;sup>b</sup> Term Birth

### **Listing 18:** 16.2.11.3: Pregnancy Reports – Live Birth Outcomes

| Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal<br>Distress<br>During<br>Labor and<br>Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month of<br>Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Congenital Anomalies are included in the Adverse Event listing.

### **Listing 19:** 16.2.11.4: Pregnancy Reports – Still Birth Outcomes

| ibject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress<br>During<br>Labor and<br>Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital<br>Anomalies? | Autopsy<br>Performed? | If Autopsy, Etiology<br>for Still Birth<br>Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

### **Listing 20:** 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy Outcome<br>(for this Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|